

### Werewolf Therapeutics, Inc.

### STATISTICAL ANALYSIS PLAN

Protocol Title : A Phase 1 (First-In-Human [FIH]), Multi-Site, Dose Escalation and

Expansion Study of WTX-330 in Adult Patients with Advanced or

Metastatic Solid Tumors or Lymphoma

**Protocol Number** : WTX-330x2101

Compound Number : WTX-330

Version : V2.0

Effective Date : [26Feb2025]

### **Description:**

- The purpose of this Statistical Analysis Plan (SAP) is to describe the planned final analyses and output to be included in the Clinical Study Report (CSR) for Protocol WTX-330x2101.
- Any post-hoc, or unplanned analyses performed to provide results for inclusion in the CSR but not specified in this SAP will be clearly specified in the CSR.

### Author's Name, Institution, and Job Title:

Author: Shuangli Guo

Senior Manager Biostatistics

Caidya

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |





# **Approval and Signature Page**

# Approved by:

| Name, Institution, and Job Title | Signature | Date |
|---|---|---|
| Shuangli Guo<br>Senior Manager Biostatistics<br>Caidya | Signed by: Signer Name: Shuangli Guo Signing Reason: I am the author of this document Signing Time: 26-Feb-2025 7:28:35 PM GMT 3F1277AD321D4048BF564AE5BED08E47 | 26-Feb-2025 |
| Oliver Schonborn-Kellenberger<br>Biostatistician<br>Werewolf Therapeutics, Inc. | Signiert von: Oliver Schönborn-Kullenberger Name des Unterzeichners: Oliver Schönborn-Kellenb Signiergrund: Ich habe dieses Dokument geprüft Signierzeit: 26-Feb-2025 8:00:33 PM GMT 988B94B1FDA24A35AEB8361DCA46EBF3 | 26-Feb-2025<br>erger |

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |





# **Version History**

This Statistical Analysis Plan (SAP) for study WTX-330x2101 is based on the protocol 02 dated 06 April 2023.

| SAP Version | Effective Date | Author | Summary of Changes |
|---|---|---|---|
| 0.1 | [19Dec2023] | Shuangli Guo | Original version based on the protocol Version<br>Number 02, Dated on 06 April 2023 |
| 0.2 | [12June2024] | Shuangli Guo | Add summary for Deauville Score |
| 0.3 | [21June2024] | Shuangli Guo | Add ASTCT Grade for Cytokine Release Syndrome |
| 1.0 | [21June2024] | Shuangli Guo | Accept changes in version 0.3 |
| 1.1 | [25Feb2025] | Shuangli Guo | Add Free IL-12 PK analysis |
| 2.0 | [26Feb2025] | Shuangli Guo | Accept changes in draft 1.1 |

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



## **Table of Contents**

| Summary of Key Protocol Information | |
|---|---|
| • | |
| 1.0 | |
| • | |
| V 1 | |
| • | |
| <b>A</b> | |
| · · | |
| · | |
| Programming Environment | |
| Analysis Groups | |
| List of Data Display and Handling Appendices | 11 |
| Study Conduct and Study Population | |
| Overview of Planned Analyses of Study Conduct and Study Population. | |
| Study Conduct | |
| Summary of Analysis Sets | 12 |
| Subject Disposition | |
| Protocol Deviations | |
| Demographics and Baseline Disease Characteristics | 14 |
| Demographics and General Baseline Characteristics | |
| Cancer History | |
| Prior Cancer Therapy | |
| General Medical History | |
| Prior Non-cancer Therapies & Concomitant Therapies | |
| Prior and Concomitant Medications | |
| Prior and Concurrent Procedures | |
| Exposure and Compliance | 17 |
| Efficacy Analyses | |
| v | |
| • | |
| * | |
| - | |
| · · | |
| • | |
| • | |
| ment Name: Statistical Analysis Plan Template(EN) | |
| Hent Name. Statistical Analysis Plan Template(EN) | Page 4 01 41 |
| | Analysis Groups List of Data Display and Handling Appendices Study Conduct and Study Population Overview of Planned Analyses of Study Conduct and Study Population. Study Conduct Summary of Analysis Sets Subject Disposition Protocol Deviations Demographics and Baseline Disease Characteristics Demographics and General Baseline Characteristics Cancer History Prior Cancer Therapy General Medical History Prior Non-cancer Therapies & Concomitant Therapies Prior and Concomitant Medications Prior and Concurrent Procedures Exposure and Compliance |



| Protoco | ol Number: WTX-330x2101 | SAP v2.0 [26Feb2025] |
|---|---|---|
| 8.3.4. | Analysis of CBR and iCBR | 22 |
| 8.3.5. | Analysis of Time to Events | |
| 8.4. | Subgroup Analyses | |
| 9. | Safety Analyses | 22 |
| 9.1. | Overview of Planned Safety Analyses | |
| 9.2. | MTD and DLT Events | 23 |
| 9.2.1. | Dose Escalation and Determination of MTD | 23 |
| 9.2.2. | DLT Events | |
| 9.3. | Adverse Events (AEs) | 24 |
| 9.3.1. | AE-related Definitions and Derivations | 24 |
| 9.3.2. | Planned Analysis of Adverse Events | 24 |
| 9.4. | Deaths | 25 |
| 9.5. | Clinical Safety Laboratory Tests | 25 |
| 9.6. | Electrocardiograms (ECG) | 26 |
| 9.7. | Vital Signs and Body Measurements | 26 |
| 9.8. | Physical Examination | 27 |
| 9.9. | ECOG Performance Status | 27 |
| 9.10. | Pregnancies | 27 |
| 10. | Pharmacokinetics | 27 |
| 10.1. | Schedule for PK Sampling | 27 |
| 10.2. | Pharmacokinetic Parameters | 27 |
| 10.3. | Analysis of Pharmacokinetic Parameters | 28 |
| 11. | Anti-Drug Antibody (ADA) | 28 |
| 12. | Pharmacodynamics | 28 |
| 12.1. | Overview of Pharmacodynamic Analyses | |
| 12.2. | Immune Cells | |
| 12.3. | Circulating Cytokines and Soluble Factors | 31 |
| 13. | Multiplicity | |
| 14. | References | |
| <b>15.</b> | Appendices | |
| 15.1. | Appendix 1: Referenced Study Documents, Software and Standards | |
| 15.2. | Appendix 2: Descriptive Statistical Summaries | |
| 15.3. | Appendix 3: Data Display Conventions | |
| 15.4. | Appendix 4: Study Day, Duration, Period, Visit and Analysis Windows | |
| 15.5. | Appendix 5: Derived Data And Definitions | |
| 15.6. | Appendix 6: Premature Withdrawals & Handling of Missing Data | |
| 15.7. | Appendix 7: List of Abbreviations | 39 |

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



#### **Summary of Key Protocol Information** 1.

Study documents, software, and/or standards on which this version of SAP is based are given in Subsection 15.1. Up-versioning of these documents do not necessarily require an update of this SAP, unless the changes affect the planned analyses or the interpretation of analysis results.

#### 1.1. Changes to the Protocol Defined Statistical Analysis Plan

There is no major changes from the originally planned statistical analysis specified in the protocol v02 dated 06 April 2023, except for the addition of Efficacy Evaluable Analysis Set, Pharmacodynamics Analysis Set, and ADA analysis set.

#### 1.2. **Study Objectives and Endpoints**

| Objectives | Outcome Variables |
|---|---|
| Primary Objectives and Endpoints for Dose Escalation | |
| To determine the MTD and/or<br>recommended dose for expansion<br>(RDE). | Frequency, severity, and relatedness of treatment-<br>emergent adverse events (TEAEs) and serious adverse<br>events (SAEs), changes in safety laboratory<br>parameters, and DLTs (if observed) for WTX- 330. |
| Dose Escalation and Expansion (Parts 1 a | and 2) |
| To further characterize the safety of<br>WTX- 330 | Frequency, severity, and relatedness of TEAEs and SAEs, changes in safety laboratory parameters, and DLTs (if observed) for WTX-330 |
| To evaluate the anti-tumor activity of<br>WTX-330 | Overall response rate (ORR) (complete response [CR] + partial response [PR]), duration of response (DOR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and immune-overall response rate (iORR) (immune-complete response [iCR] + immune-partial response [iPR]) by immune-RECIST (iRECIST), or response by Lugano criteria (for lymphoma only) |
| Secondary Objectives and Endpoints (Pa | rts 1 and 2) |
| To evaluate the immunogenicity of<br>WTX330 | Incidence and titers of ADAs towards WTX-330 |

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



# **Objectives Outcome Variables** Secondary Objectives and Endpoints (Parts 2) To evaluate the antitumor activity of ORR (CR + PR) based on best overall response (BOR) WTX-330 patients in DOR relapsed/refractory (r/r) advanced or metastatic malignancies who have Disease control rate at month 3, 6 and 9 progressed on CPIs or who have tumor Progression free survival (PFS) per RECIST v1.1 indications for which CPIs are not (solid tumor) and iRECIST or Lugano classification approved (lymphoma; Cheson et al., 2014) assessed by Investigator. Overall survival (OS) Exploratory Objectives and Endpoints (Parts 1 and 2)

### 1.3. Study Design

This study is a Phase 1, FIH, multi-site study to determine the safety profile and MTD and/or RDE of WTX-330 in patients with advanced or metastatic solid tumors or lymphomas.

The study consists of a dose escalation part and a dose expansion part. The study design is illustrated in the Figure below.

### 1.3.1. Dose Escalation – Monotherapy

The dose escalation part of the study will be conducted in patients with relapsed/refractory advanced and/or metastatic solid tumors. Patients with primary CNS malignancies are ineligible. WTX-330 will be administered as a single agent at a dose based on body weight on Days 1 and 15 via IV over 15 minutes (Q2W) of the 28-day treatment cycle (in the absence of infusion-related reactions) at the first and all subsequent infusions. The dose escalation cohorts have been planned as 0.016 mg/kg, 0.032 mg/kg, 0.056 mg/kg, 0.084 mg/kg, 0.126 mg/kg, 0.190 mg/kg, 0.290 mg/kg, and potentially higher than 0.440 mg/kg.

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



An adaptive 2-parameter BLRM incorporating EWOC will be used during the Dose Escalation (Part 1) to select dose levels and to estimate the MTD (See Protocol Appendix F). Determination of the MTD during dose escalation will be based upon an estimation of the probability of a DLT in Cycle 1 in the dosedetermining set (DDS). If the MTD is not reached during dose escalation, the recommended dose for expansion (RDE) will be determined based on review of DLTs, AEs and SAEs, laboratory, PK and PD data by the DEC as the dose with the optimal therapeutic window for WTX-330.



CPI = checkpoint inhibitor; MTD = maximum tolerated dose; Q2W = every 2 weeks; r/r = relapsed/refractory; SOC = standard of care.

#### 1.3.2. **Dose Expansion**

Once the MTD/RDE is identified from Dose Escalation (Part 1), the Dose Expansion part (Part 2) will open and begin enrollment. Patients will have a confirmed diagnosis of a r/r locally advanced or metastatic solid tumor or lymphoma for which the patient has progressed on or is intolerant of standard therapy, or for whom no standard therapy with proven benefit exists. Dose Expansion will be conducted in 2 arms that will enroll patients based on the following criteria:

- Arm A: Patients with indications for which a CPI is indicated/approved (e.g., cutaneous malignant melanoma, RCC, non-small cell lung cancer [NSCLC], head and neck squamous cell carcinoma [HNSCC], urothelial carcinoma, etc.) who have received a CPI regimen and who demonstrate primary or secondary resistance to CPI therapy.
- Arm B: Patients with tumor types for which CPI therapy is not indicated/approved (e.g., pancreatic cancer, microsatellite-stable [MSS] colorectal carcinoma, castrate-resistant prostate cancer (CRPC), non-Hodgkin lymphoma) and who are CPI naïve. Patients with NHL should have either follicular lymphoma or diffuse large B-cell lymphoma (DLBCL), though other subtypes of NHL such as T-cell lymphomas may be considered after discussion with the Sponsor. All patients with NHL must have received at least 2 prior systemic therapies.

#### 2. **Statistical Hypotheses**

Hypothesis testing is not preplanned in this study for efficacy endpoints. Confidence intervals may be provided for information purposes only.

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



### 3. Sample Size Considerations

The overall sample size for this study is approximately 75 patients between the dose escalation and dose expansion parts of the study and will depend on the observed DLT profiles of WTX-330.

### 3.1. Dose Escalation Phase

Approximately 30 to 35 patients will be enrolled into the dose escalation part including all dosing groups (0.008 mg/kg (Dose Level -1), 0.016 mg/kg, 0.032 mg/kg, 0.056 mg/kg, 0.084 mg/kg, 0.126 mg/kg, 0.190 mg/kg, 0.290 mg/kg, and potentially higher than 0.440 mg/kg). For the first dose level of WTX-330, at least 1 patient needs to be evaluable. Dose groups will be included in the dose escalation part with 3 to 6 patients in each group.

During dose escalation, additional patients may be enrolled into cohorts at dose levels that have previously been determined to be safe to better understand the safety, tolerability, and PK of WTX-330 before or while proceeding with further dose escalation. Up to 10 patients may be enrolled into an enrichment group. Enrichment groups will enter the DDS and be accounted for in the BLRM for the assessment of DLTs.

The exact sample size cannot be prespecified in advance because it is a dynamic feature of the design. The actual sample size of the dose escalation part of the study will depend upon the underlying dose toxicity profile and variability in actual data realization.

## 3.2. Dose Expansion Phase

Once the MTD and/or RDE is determined for WTX-330 as a monotherapy in the dose escalation (Part 1), the dose expansion (Part 2) with WTX-330 as a monotherapy will initiate in each of the 2 dose expansion cohorts (Arms A and B; Section 1.3.2). Cohorts of up to 20 patients each are planned for each of the dose expansion arms.

These sample sizes were selected based on practical consideration to confirm safety of WTX-330 for each indication and without formal power calculation.

To show that these sample sizes will also give early evidence on clinical benefit, Table below provides probabilities of declaring success for varying true response rate based on independent Bayesian Betabinomial models assuming Beta (0.5, 0.5) priors for each expansion arm and declaring success if the posterior probability that the true response rate exceeds 10% is large (at least 90%). This translates to declaring success for an expansion arm if at least 4/20 are observed.

| True response rate (%) | 10 | 15 | 20 | 25 | 30 | 40 | 50 | 60 |
|---|---|---|---|---|---|---|---|---|
| Probability of declaring success (%) | 13.3 | 35.2 | 58.9 | 77.5 | 89.3 | 98.4 | 99.9 | 100 |

# 4. Planned Analyses

# 4.1. Interim Analyses

Each dose escalation step is considered an interim analysis. The BLRM will be updated with the respective number of subjects treated and the number of DLTs observed in the last cohort. The updated model will then give a statistical recommendation for the next escalation step. In addition, a risk-benefit assessment that includes a comprehensive analysis of safety and available clinical information will be done to decide on the next escalation steps.

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



After the dose escalation an interim analysis to review the safety data may be performed for this trial. The analyses will be based on a data snapshot. As this trial is of exploratory nature and no inferential statistics are planned, no adjustment for multiple testing will be done.

### 4.2. Final Analyses

One final planned primary analysis will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed, and final database release and database freeze has been declared by Data Management.

### 5. Analysis Sets

| Analysis Set | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened Subjects | All subjects who provided informed consent. | <ul> <li>Disposition</li> </ul> |
| Enrolled Subjects | All subjects who provided informed consent and met all study eligibility criteria as recorded in the eCRF. | Disposition |
| Safety Analysis Set | This will include all patients who received at least 1 dose of WTX-330 and had at least 1 post-baseline safety assessment. Safety analyses will in general be descriptive and will be presented in tabular format with the appropriate summary statistics for the Safety Analysis Set. The safety set will be the primary population for all safety related endpoints except determination of the dose-DLT relationship. | <ul> <li>Demographics</li> <li>Cancer history</li> <li>Exposure and compliance</li> <li>Previous and concomitant therapies</li> <li>Safety evaluations except for DLT</li> </ul> |
| Dose-determining (DDS) Analysis Set | This will include all patients in the safety set who have either (a) experienced a DLT at any time during Cycle 1, or (b) completed Cycle 1 without experiencing a DLT. The DDS, which is the analysis set used for determination of the MTD, will consist of patients who have met the minimum treatment and safety evaluation requirements of the study, and/or who experience a DLT during Cycle 1. The minimum treatment and safety evaluation requirements will have been met if, in Cycle 1, the patient received 75% of assigned study treatment dose, completed the required safety evaluations for Cycle 1, and did not experience a DLT. Patients who do not meet these minimum treatment and safety evaluation requirements will be regarded as ineligible for inclusion in the DDS and will be replaced, if | • DLT events |

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



| Protocol Number: WTX-330x2101 | SAP v2.0 [26Feb2025] |
|-------------------------------|----------------------|
|-------------------------------|----------------------|

| Analysis Set | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | needed, until the minimum number of patients required for evaluation is reached. | |
| Efficacy Evaluable Analysis<br>Set | All subjects who receive at least one dose of study drug and with both baseline and post-baseline disease assessment, or all subjects who receive at least one dose of study drug with baseline disease assessment and without post-baseline disease assessment due to death or progression. | Efficacy: ORR, iORR, DCR, iDCR, PFS, iPFS, DoR, iDoR, OS |
| Pharmacokinetics (PK)<br>Analysis Set | This will consist of all patients who have received at least 1 dose of study drug and have at least 1 post-dose PK measurement. | • PK |
| Anti-Drug Antibody (ADA)<br>Analysis Set | All subjects who received at least 1 dose of WTX-330 and have at least 1 baseline WTX-330 IG sample or at least 1 post-baseline WTX- | • ADA |

Note: Data after withdrawn of ICF will be excluded in analysis.

#### 6. **General Considerations and Data Handling Conventions**

330 IG sample.

#### **Programming Environment** 6.1.

Unless otherwise specified, all analyses will be conducted using SAS® version 9.4 or later.

#### **6.2. Analysis Groups**

Unless otherwise specified, the statistical analyses will be presented by dose level in dose escalation phase and by arm in the dose expansion phase for the different analysis sets as defined in Section 5.

#### 6.3. List of Data Display and Handling Appendices

Table 2 Overview of Data Display and Handling Appendices

| Component |
|---------------------------------------------------------------------|
| Appendix 2: Descriptive Statistical Summaries |
| Appendix 3: Data Display Conventions |
| Appendix 4: Study Day, Duration, Period, Visit and Analysis Windows |
| Appendix 5: Derived Data And Definitions |
| Appendix 6: Premature Withdrawals & Handling of Missing Data |

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



# 7. Study Conduct and Study Population

# 7.1. Overview of Planned Analyses of Study Conduct and Study Population

Table 3 Overview of Planned Analyses of Study Conduct & Study Population

| | Data Displays Generated | | rated |
|---|---|---|---|
| | Table | Figure | Listing |
| Study Conduct | | | |
| Subject Disposition | Y | | Y |
| Analysis Sets | Y | | Y |
| Protocol Deviations | Y | | Y |
| Demographics and Baseline Disease Characteristics | | | |
| Demographics and General Baseline Characteristics | Y | | Y |
| (Vital Signs, Body Measurements, Performance Status) | 1 | | 1 |
| Cancer History & Characteristics | Y | | Y |
| Prior Cancer Therapy | Y | | Y |
| General Medical History by SOC and PT | Y | | Y |
| Prior Non-cancer Therapies and Concomitant Therapie | es | | |
| Prior Medications by ATC level II and PN | Y | | Y |
| Concomitant Medications ATC level II and PN | Y | | ĭ |
| Prior and Concomitant Procedures | | | Y |
| Exposure and Compliance | | | |
| Study Drug Exposure & Compliance | Y | | Y |
| Infusion Interruptions & Dose Modifications | Y | | Y |

### 7.2. Study Conduct

### 7.2.1. Summary of Analysis Sets

The number and relative frequency of subjects in each analysis set as defined in Section 5 will be descriptively summarized.

- Number of screened subjects (percentage not to be calculated)
- Number of screen failures (percentage not to be calculated)
- Reason for screen failure (percentage not to be calculated, include non 0 categories only)
  - Adverse event
  - o Death
  - o Failure to meet continuation criteria
  - o Logistical problem
  - Met eligibility criteria but not needed
  - Never dosed
  - o Other
  - Physician decision
  - Pregnancy
  - o Protocol-specified withdrawal criterion met
  - Screen failure
  - Screening not completed

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |





- Technical problems
- Withdrawal by parent/guardian
- Withdrawal by subject
- Withdrawal of consent
- o COVID-19 Related
- Number of Enrolled Subjects (percentage not to be calculated)
- Safety Analysis Set (percentage not to be calculated)
- Dose-determining (DDS) Analysis Set
- Efficacy Evaluable Analysis Set
- Pharmacokinetics Analysis Set

ADA Analysis Set

Percentages will be calculated with based on the number of subjects in the Safety Analysis Set. Listing will be provided for all Screened Subjects.

### 7.2.2. Subject Disposition

The number and relative frequency of subjects of the following will be descriptively summarized using Safety Analysis Set:

- Subjects with ongoing or discontinued WTX-330 treatment
- Subjects who ongoing or discontinued the study
- Reasons for WTX-330 discontinuation
  - Adverse Event
  - o Death
  - Physician Decision
  - Pregnancy
  - o Progressive Disease
    - Radiographic
    - Clinical
  - o Study Terminated by Sponsor
  - Withdrawal of ICF
  - o Other
- Reasons for end of study
  - Completed study
  - Withdrawal of Consent by Patient
  - Lost to Follow-Up
  - o Death
  - Sponsor Terminated by Sponsor
  - o COVID-19 Related
  - o Other

Percentages will be calculated with based on the number of subjects in the Safety Analysis Set. Disposition of subjects will be provided in a data listing for the Safety Analysis Set.

### 7.2.3. Protocol Deviations

Protocol Deviation Management Plan (PDMP) version: 1.0 dated on 23Sep22 defined the study specific procedures and responsibilities for managing Protocol Deviations. The document listed the definition of

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |





Bioclinica Deviation Description and Deviation Area, as well the Deviation Category (major vs minor). Subject level protocol deviations will be documented in the Clinical Trial Management System (CTMS).

Deviations from the clinical protocol may include, but are not limited to:

- ICF/Subject Information
- Ineligible Subject Enrolled
- IMP Dose Error
- IMP Other Error
- **Prohibited Medication**
- Procedure/ Test Not Done
- Procedure/ Test Out of Window
- Procedure/ Test Not Performed per Protocol
- Visit Out of Window
- SAE or AESI Reporting Failure
- Other

The number and percentage of subjects with any protocol deviation, major protocol deviation, or minor protocol deviation will be summarized using the Safety Analysis Set separately.

#### 7.3. **Demographics and Baseline Disease Characteristics**

Demographic and baseline disease characteristics as specified in detail below will be presented descriptively using the Safety Analysis Set.

#### 7.3.1. **Demographics and General Baseline Characteristics**

The following baseline characteristics will be descriptively (n, mean, Mean, Standard Deviation, Median, Min, Max) summarized using the Safety Analysis Set:

- Age at informed consent (years)
- Weight (kg) at baseline
- Height (cm) at baseline

The number and percentage of subjects under each of the following baseline characteristics will be summarized using the Safety Analysis Set:

- Sex (Female [with childbearing potential, without childbearing potential], Male)
- Age group (<45, 45 through 65, and  $\ge$ 65)
- Race (American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, White, Other, and Unknown)
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino, and Unknown)
- Eastern Cooperative Oncology Group (ECOG) performance status (0, 1)

#### 7.3.2. **Cancer History**

The following cancer history characteristics of solid tumor will be summarized descriptively (n, mean, Mean, Standard Deviation, Median, Min, Max) using the Safety Analysis Set:

- Time since date of initial histopathological diagnosis (months) = (date of first dose date of initial histopathological diagnosis)/30.4375
- Time since date of most recent disease recurrence/progression (months) = (date of first dose date of most recent disease recurrence/progression)/30.4375

The number and percentage of subjects with the following primary and metastatic cancer history for solid tumor will be summarized using the Safety Analysis Set:

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |





- Time since date of initial histopathological diagnosis (<12 months, >=12 months < 24 months,  $\geq$  24 months - < 36 months,  $\geq$  36 months)
- Cancer type as recorded in eCRF
- Primary site of solid tumor as recorded in eCRF
- Any pathologic sub-type (Yes, No)
- Stage of solid tumor at initial diagnosis (0, I, II, III, IV)
- Stage of solid tumor at baseline (0, I, II, III, IV)
- Characterization of disease at study entry (locally advanced, metastatic)
- Metastatic site as recorded in eCRF
- Any known genetic mutations (Yes [BRAF, EGFR, HER2, KRAS, KIT, PDGFRA, PIK3CA, NRAS, VHL, Other], No)
- MSI status (Known [MSI-H, MSI-L, MSS dMMR, pMMR] Unknown, Not Applicable)
- TMB Status Known? (No, Not Applicable, Yes [High, Intermediate, Other])
- Tumoral genetic characterization (Yes. No. Not Applicable)

The following cancer history characteristics of lymphoma will be summarized descriptively (n, mean, Mean, Standard Deviation, Median, Min, Max) using the Safety Analysis Set:

- Time since date of diagnosis (months) = (date of first dose date of initial diagnosis)/30.4375
- Time since date of transformation (months) = (date of first dose date of transformation)/30.4375

The number and percentage of subjects with the following cancer history for lymphoma will be summarized using the Safety Analysis Set:

- Time since date of diagnosis (<12 months, >=12 months < 24 months, >=24 months < 36 months,  $\geq 36$  months)
- Disease at screening as recorded in eCRF
- Current disease stage (I, IE, II, IIE, II BULKY, III, IV)
- Current Ann Arbor Staging (Stage I, Stage IE, Stage II, Stage IIE, Stage III, Stage IIIE, Stage IIIS, Stage IIIE/S, Stage IV, Not Applicable)
- Bone Marrow Involvement? (Yes, No)

Cancer history characteristics will also be provided in a data listing using the Safety Analysis Set.

#### **Prior Cancer Therapy** 7.3.3.

Prior cancer therapy information will be summarized using descriptive statistics. Denominators for calculating percentages will be based on the number of subjects in the Safety Analysis Set. Summaries will include the following:

- Any prior anti-cancer therapy
- Type of prior anti-cancer therapy (Surgery, Radiation therapy, Systemic therapy)
- Type of Systemic Therapy (Chemotherapy, Immunotherapy, Hormonal therapy, Targeted therapy, Other)
- Systemic therapy setting (Advance/metastatic, Palliative, Other)
- Best overall response across all prior systemic therapies (CR, PR, SD, PD, NE, NA, Unknown)
- Best overall response from the latest prior systemic therapy (CR, PR, SD, PD, NE, NA, Unknown)
- Reason for stopping treatment in the latest prior systemic therapy (Treatment completed, Progressive disease, Toxicity, Adverse event, Other)
- Number of line of therapies  $(0, 1, 2, 3, \ge 4)$

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |





Time since the last prior systemic therapy started (months, date of first dose – start date of the last prior systemic therapy)/30.4375) will be descriptively (n, mean, Mean, Standard Deviation, Median, Min, Max) summarized using the Safety Analysis Set:

Prior systemic anti-cancer medications will be coded according to the latest version of World Health Organization drug dictionary (WHODRUG Global B3 March 2023) and stored with ATC categories and preferred names (PN). A primary ATC category will be selected before DBL based on considerations such as indication, route of administration, and dosage.

The number and percentage of subjects with medication use coded to each primary ATC level 2 category and preferred name (PN) combination will be summarized descriptively using the Safety Analysis Set. If a subject has received more than 1 drug within an ATC class or PN, the subject will be counted only once for this ATC class or PN.

Prior cancer therapy will be reported in data listings using the Safety Analysis Set.

### **General Medical History**

The medical conditions will be coded according to Medical Dictionary for Regulatory Activities (MedDRA 26.0) according to the Data Management Plan.

The number and percentage of subjects with conditions coded to each primary system organ class (SOCs) and preferred terms (PTs) will be summarized descriptively using the Safety Analysis Set. If a subject has more than 1 medical condition within an SOC or PT, the subject will be counted only once for the respective SOC or PT.

Data listings of all medical history records will be provided using the Safety Analysis Set.

#### 7.4. **Prior Non-cancer Therapies & Concomitant Therapies**

#### 7.4.1. **Prior and Concomitant Medications**

Prior and concomitant medications will be coded according to the latest version of World Health Organization drug dictionary (WHODRUG Global B3 March 2023) according to the Data Management Plan and stored with ATC categories and preferred names (PN). A primary ATC category will be selected before DBL based on considerations such as indication, route of administration, and dosage. For classification of prior and concomitant use and the imputation of (partial) missing dates, refer to Subsections 15.5 and 15.6. Prior medication is the medication that stopped before the first dose of WTX-330. Concomitant medication is the medication that are used on/after the first dose of WTX-330.

The number and percentage of subjects with medication use coded to each primary ATC level 2 category and preferred name (PN) combination will be summarized descriptively using the Safety Analysis Set as described. If a subject has received more than 1 drug within an ATC class or PN, the subject will be counted only once for this ATC class or PN. For medications with a common PN but being used in different scenarios with different primary ATC level 2 categories, the PN needs to be summarized under all these ATC level categories.

Prior and concomitant medications information will also be provided in a data listing using the Safety Analysis Set.

#### 7.4.2. **Prior and Concurrent Procedures**

Prior and concomitant procedure information will also be provided in a data listing using the Safety Analysis Set.

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



#### 7.5. **Exposure and Compliance**

The following exposure and compliance summaries will be derived for each subject for WTX-330:

- Duration of exposure (weeks) is (the date of last administration of WTX-330 the date of first administration of WTX-330 + 14)/7.
- Total Planned Dose (mg/kg) is calculated by sum of the individual Planned Dose Level being reported in eCRFs.
- Cumulative Dose (mg/kg) is calculated by sum of the individual Total Dose Administered being reported in eCRFs.
- Treatment compliance (%) is 100\*(Cumulative Dose/Total Planned Dose).
- Average Dose Intensity (mg/kg) /cycle) is calculated by Cumulative Dose / number of treatment cycles started (any amount of the study drug was administered)

The duration of exposure (weeks), number of treatment cycle started, and number of study drug infusions, cumulative Dose, Treatment Compliance and Average Dose Intensity will be summarized using descriptive statistics as numerical variables; percent compliance will also be summarized as a categorical variable ( <80%, 80-120%, ≥120%); duration of exposure will also be summarized as a categorical variable (<4 weeks, 4 to <12 weeks,  $\ge$ 12 weeks).

Additionally, the number and percentage of subjects with 0, 1, 2, or  $\geq 3$  WTX-330 infusion interruption events and reason for infusion interruption (Infusion Reaction, Adverse Event other than Infusion Reaction, Other) will be summarized; the number and percentage of subjects with WTX-330 dose adjustment (Dose Missed, Dose Reduced, Dose Discontinued, Dose Interrupted) and reason for WTX-330 dose adjustment (Adverse Event, PI/Sponsor Decision, Other)) will be summarized.

Exposure, dosage, and compliance data will be presented in a data listing.

#### 8. **Efficacy Analyses**

#### 8.1. **Overview of Planned Efficacy Analyses**

All analyses of efficacy outcomes will be primarily based on the Efficacy-Evaluable Set.

Table 1 Overview of Planned Efficacy Analyses

| | <b>Data Displays Generated</b> | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Target Lesion Size and Individual Assessment | | | |
| Spider (line) plot of percent CFB of sum of target lesion diameters (Solid tumors) | | Y | |
| Spider (line) plot of percent CFB of sum of the product of the diameters (Lymphomas) | | | |
| Waterfall plot of best percent CFB of sum of target lesion diameters (Solid tumors) | | Y | Y |
| Waterfall plot of best percent CFB of sum of the product of the diameters (Lymphomas) | | | |
| Swimming lane plot of individual time point response assessment and time on treatment | | Y | |
| ORR and iORR | | | |
| Number and percentages of subjects in each BOR (iBOR) category ORR (iORR) and 95% Clopper-Pearson interval | Y | | Y |

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



| | | Data Displays Generated | |
|---|---|---|---|
| | Table | Figure | Listing |
| CBR and iCBR | | | |
| CBR (iCBR) at 3, 6, and 9 months | Y | | Y |
| DOR and iDOR | | | |
| Number of responders | | | |
| Number of events | | | |
| Number of censored observations | | | |
| Kaplan-Meier estimates of survivor function at landmark time points and | Y | | Y |
| associated asymptotic 95% CI | | | |
| Estimated quartiles of DOR (iDOR) and associated asymptotic 95% CI | | | |
| PFS and iPFS | | | |
| Number of events | | | |
| Number of censored observations | | | |
| Kaplan-Meier estimates of survivor function at landmark time points and | Y | | Y |
| associated asymptotic 95% CI | 1 | Y | 1 |
| Estimated quartiles of PFS (iPFS) and associated asymptotic 95% CI | | | |
| OS | | | |
| Number of deaths | | | |
| Number of censored observations | | | |
| Kaplan-Meier estimates of survivor function at landmark time points and | Y | | Y |
| associated asymptotic 95% CI | | Y | |
| Estimated quartiles of OS and associated asymptotic 95% CI | | | |

#### 8.2. **Definitions of Efficacy Outcome Variables**

#### Solid tumors

Assessment of solid tumors will be based on RECIST 1.1 and iRECIST during Screening within 28 days of Cycle 1 Day 1. On-study scans should be performed every 8 weeks (±7 days) from Cycle 1 Day 1 for the first 6 cycles and every 12 weeks (±7 days) thereafter. Disease assessments will include radiographic measurements of tumors using computed tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET)/CT. The modality for screening/baseline imaging will be used until progressive disease (PD) per RECIST 1.1 and confirmed progressive disease iRECIST (iCPD) for solid tumor, withdrawal of consent, or initiation of a new anticancer therapy.

### Lymphomas

Assessment of lymphomas (NHL) in Dose Expansion Part B will be based on Lugano classification during Screening within 28 days of Cycle 1 Day 1. On-study scans should be performed every 8 weeks (±7 days) from Cycle 1 Day 1 for the first 6 cycles and every 12 weeks (±7 days) thereafter. At Screening, lymphoma patients with FDG-avid disease will undergo fluorodeoxyglucose (FDG) PET/CT imaging. All subsequent disease assessments should also be performed with FDG PET/CT, using the Deauville 5-point scale. The avidity of up to six of the largest dominant nodes, nodal masses and/or extranodal lesions, selected to be clearly measurable in two diameters, should be assessed. Nodes should preferably be from disparate regions of the body and should include, where applicable, mediastinal and retroperitoneal areas. Non-nodal lesions include those in solid organs, the GI tract, cutaneous lesions, or those noted on palpation. Non-measured lesions are any disease not selected as dominant or measurable. For patients with non-FDG-avid or variably FDG-avid tumors, a CT scan of the chest/abdomen/pelvis and any additional known sites of disease will be

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |





performed with IV contrast. The modality for screening/baseline imaging will be used until progressive disease (PD) per Lugano, withdrawal of consent, or initiation of a new anticancer therapy.

### **Individual Time Point Response**

According to RECIST 1.1, the time point response will be evaluated as Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD), Not Evaluable (NE). According to iRECIST, the time point response will be evaluated as Immune unconfirmed progressive disease (iUPD), Immune confirmed progressive disease (iCPD), Immune complete response (iCR), Immune partial response (iPR), Immune stable disease (iSD), Not Evaluable (NE). According to Lugano classification, the Lugano (Metabolic/PET-CT Based) time point response will be evaluated as Complete Response (CR), Partial Remission/Response (PR), Stable Disease (SD), and Progressive Disease (PD).

The following RECIST 1.1, iRECIST 1.1, and Lugano time point response(s) will be excluded from derivation of Best Overall Response (BOR), Clinical Benefit Rate (CBR), Duration of Response (DOR), Progression free Survival (PFS), Immuno Best Overall Response (iBOR), Immuno Clinical Benefit Rate (iCBR); Immuno Duration of Response (iDOR), Immuno Progression free Survival (iPFS):

- All RECIST 1.1, iRECIST 1.1 and Lugano time point response(s) after Antineoplastic therapy (including radiotherapy, surgery and medication) will be excluded
- For RECIST 1.1 and Lugano, any time point response(s) after the first PD will be excluded
- For iRECIST, any time point response(s) after the first iCPD will be excluded

#### 8.2.2. **Best Overall Response**

Best Overall Response (BOR) of each subject per RECIST 1.1 is based on the tumor response among all visits. CR or PR needs to be confirmed in a subsequent assessment at least 28 days apart. Unconfirmed PR or CR will be categorized as SD. See the derivation rules below:

- If a subject has at least 2 CRs at least 28 days apart, and there are no other assessments in between being PR, SD or PD, then the BOR is defined as confirmed CR;
- If a subject has a PR, another CR/PR at least 28 days later, and there are no other assessments in between being SD or PD, then the BOR is defined as confirmed PR;
- For those subjects who do not meet confirmed CR or PR conditions above, if the subject had at least 1 tumor assessment record of CR/PR/SD which is at least 49 days after date of first dose of any study drug, and if the assessment is not preceded by any prior PD, then the BOR is defined as SD;
- For those subjects who do not meet confirmed CR, confirmed PR or SD conditions defined as above, but they have any tumor assessment as PD, their BOR is PD:
- Otherwise, BOR is defined as NE for subjects without any post-baseline tumor assessment data.

Immune Best Overall Response (iBOR) of each subject per iRECIST 1.1 is deleted from all visit responses according to the following sequence: iCR, iPR, iSD, iCPD, iUPD, NE.

Best Overall Response (BOR) of each subject with lymphomas (NHL) per Lugano is seleted from all visit responses according to the following sequence: CR, PR, SD, PD.

The subjects without postbaseline assessment will be categories as NE.

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



#### 8.2.3. **Overall Response Rate**

Overall response rate (ORR) per RECIST 1.1 and per Lugano is defined as the proportion of subjects achiving CR or PR of BOR.

Immune Overall response rate (iORR) per iRECIST 1.1 is defined as the proportion of subjects achiving iCR or iPR of iBOR.

#### 8.2.4. **Clinical Benefit and Clinical Benefit Rate**

Clinical benefit for 3, 6, and 9 months based on RECIST 1.1 and Lugano is defined as the subject achiving CR, PR, or SD with duration  $\geq 3$ , 6, and 9 months after the date of first dose, respectively. Duration will be calculated as (the date of last CP/PR/SD, whichever occurs late) – date of first WTX-330 dose + 1)/30.4375.

Immuno Clinical benefit for 3, 6, and 9 months based on iRECIST 1.1 is defined as the subject achiving iCR, iPR, or iSD with duration  $\geq 3$ , 6, and 9 months, respectively. Duration will be calculated as (the date of last iCP/iPR/iSD – date of first WTX-330 dose + 1)/30.4375.

Clinical Benifit Rate (CBR) or Immuno Clinical Benifit Rate (iCBR) is defined as the propotion of subjects achieving clinical benefit, which will be summarized for 3, 6, and 9 months: CBR3, CBR6, CBR9, iCBR3, iCBR6, and iCBR9.

#### 8.2.5. **Duration of Response**

Duration of response (DOR), reported the subjects achieving confirmed PR or CR per RECIST 1.1, is calculated from the date of first observation of CR or PR to the date of disease progression using RECIST 1.1 criteria or death, whichever occurs first. The subjects without disease progression or death will be censored on the date of last disease assessment. See below for event/censoring rules.

| Situation | Date of Event or Censoring | Event or Censoring |
|---|---|---|
| ** using the derived dataset as descripted in section 8.2.1 | | |
| Progression after one or none missing assessment | Date of progression | Event |
| Death after one or none missing assessment | Date of death | Event |
| No progression (or death) | Date of last assessment | Censored |
| Progression or death after two or more missing | Date of last assessment prior to | Censored |
| assessment | missed assessments | Celisoreu |

Duration of response (DOR), reported the subjects achieving CR or PR of BOR per Lugano, is calculated from the date of first observation of CR or PR to the date of disease progression using RECIST 1.1 criteria or death, whichever occurs first. The subjects without disease progression or death will be censored on the date of last disease assessment. See above for event/censoring rules.

Immuno Duration of response (iDOR), reported the subjects achieving iCR or iPR per iRECIST, is calculated from the date of first observation of iCR or iPR to the date of first iUPD that is confirmed in subsequent assessments (iCPD), the date of first iUPD that is not followed any of iSD/iPR/iCR in subsequent assessments, or death, whichever occurs first. The subjects without iUPD/death, or with iUPD being annulled by subsequent assessments (iSD, iPR, iCR) will be censored at the date of last assessment.

#### 8.2.6. **Progression-free Survival**

Progression-free Survival (PFS) per RECIST1.1 and Lugano is calculated from the date of first WTX-330 dose to the date of disease progression or death, whichever occurs first. The subjects without disease progression or death will be censored on the date of last disease assessment. See event/censoring rules in section 8.2.5.

Immuno Progression-free Survival (iPFS) per iRECIST, is calculated from the date of first WTX-330 dose to the date of first iUPD that is confirmed in subsequent assessments (iCPD), the date of first iUPD that is

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |





not followed any of iSD/iPR/iCR in subsequent assessments, or death, whichever occurs first. The subjects without iUPD/death, or with iUPD being annulled by subsequent assessments (iSD, iPR, iCR) will be censored at the date of last assessment.

Alive subjects without postbaseline assessment will be censored at the date of first WTX-330 dose (day 1).

#### 8.2.7. **Overall Survival (OS)**

Overall survival (OS) is is calculated from the date of first WTX-330 dose to the date of death. The subjects without death during study will be censored at the date of last known alive.

#### 8.3. **Analysis of Efficacy Outcome Variables**

#### 8.3.1. **Analysis of Target Lesion Sizes and Individual Assessments**

For sum of target lesion in solid tumor, longest diameters for non-nodal lesions and short axis for nodal lesions will be added by subject and assessment visit. Assessments after the start of subsequent anticancer therapy will not be included when deriving the change from baseline (CFB) and best (i.e., the minimum of) percent CFB.

For sum of the product of the diameters in Lymphomas, the product of the diameters of each measurable lesion will be added by subject and assessment visit. Assessments after the start of subsequent anticancer therapy will not be included when deriving the change from baseline (CFB) and best (i.e., the minimum of) percent CFB.

A line (spider) plot for the percent CFB of sum of target lesion diameters over time in solid tumor and the percent CFB of sum of the product of the diameters over time in Lymphomas will be made for each subject in escalation part and expansion part.

A waterfall plot for best percent CFB of sum of target lesion diameters in solid tumor best percent CFB of sum of the product of the diameters over time in Lymphomas will be made for each subject in escalation part and expansion part. The plot is restricted to subjects with measurable disease at baseline and at least one valid post-baseline assessment.

Swimming lane plots will be presented for time (month) on treatment, iRECIST response assessments in solid tumor or Lugano response assessments in Lymphomas at all visits, as well as reasons for WTX-330 discontinuation for each subject in escalation part and expansion part.

#### 8.3.2. **Analysis of Deuville Scale**

Deauville 5-point scale in FDG PET/CT include: score 1 - no uptake; score 2 - uptake < to mediastinum; score 3 - uptake > mediastinum but < liver; score 4 - moderately increased uptake > liver; score 5 - markedly increased uptake and or new lesions (s) likely to be lymphoma; score x - new areas of FDG uptake unlikely to be related to lymphoma. The shift of 5-point scale from baseline to post-baseline at each scheduled visit will be summarized.

#### 8.3.3. Analysis of ORR and iORR

The number and percentage of subjects with BOR per RECIST 1.1, with iBOR per iRECIST, and with BOR per Lugano in each of the response categories will be summarized descriptively. ORR, iORR, and their 2-sided 95% confidence intervals being estimated with Clopper-Pearson method will be presented.

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



### 8.3.4. Analysis of CBR and iCBR

The number and percentage of subjects with CBR3, CBR6, CBR9, iCBR3, iCBR6, iCBR9, and their 95% confidence intervals will be estimated with Clopper-Pearson method.

### 8.3.5. Analysis of Time to Events

Time to event parameters (DoR, iDoR, PFS, iPFS, OS) will be estimated using the Kaplan-Meier method (Kaplan & Meier, 1958). The number and percentage of subjects with events/censored, the 1<sup>st</sup> quantile (25%), median, 3<sup>rd</sup> quantile (75%), and their 2-sided 95% confidence interval, event-free rate at 3/6/9/12/15 months and their 2-sided 95% confidence interval will be presented.

Event or censor category of each subject in the summary for DoR, iDoR, PFS, iPFS will be presented. Event categories include progression and death. Censor categories include No progression and death, Progression or death after antineoplastic therapy, Progression or death after two or more missing assessment.

Kaplan-Meier curves for PFS, iPFS and OS of expansion cohorts will be plotted.

### 8.4. Subgroup Analyses

No subgroup analysis is planned.

### 9. Safety Analyses

### 9.1. Overview of Planned Safety Analyses

The Safety Analysis Set will be used to evaluate all safety endpoints unless otherwise specified. In particular, the DLT-Evaluable Analysis Set will be used to evaluate DLT endpoint and to estimate MTD.

Table 2 Overview of Planned Safety Analyses

| | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Maximum Tolerated Dose (MTD) and Dose Limiting T | oxicity (DLT) | Events | |
| Number and percentage of subjects having experienced | Y | | Y |
| DLT events | 1 | | 1 |
| Adverse Events | | | |
| Overview of TEAEs | Y | | |
| All TEAEs | Y | | |
| TEAEs related to each study drug | Y | | |
| All Serious TEAEs | Y | | |
| Serious TEAEs related to each study drug | Y | | 1 |
| Grade 3 or higher TEAEs | Y | | Y |
| Grade 3 or higher TEAEs related to each study drug | Y | | |
| TEAEs leading to any study drug modification | Y | | |
| TEAEs leading to deaths | Y | | |
| TEAEs of Special Interest | Y | | |
| Immune Related Adverse Event (irAE) | Y | | Y |
| Infusion Related Reaction (IRR) | Y | | Y |
| Cytokine Release Syndrome (CRS) | Y | | Y |
| TEAEs leading to any study drug discontinuation | Y | | Y |
| All Serious TEAEs during screening period(s) | | | Y |

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



| | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Primary Cause of Deaths | | | |
| On study Deaths | | | |
| Deaths within 28 days of last administration | Y | | Y |
| Deaths after 28 days since last administration | | | |
| Clinical Safety Laboratory Tests | | | |
| Hematology | Y | | Y |
| Clinical Chemistry | Y | | Y |
| Coagulation | Y | | Y |
| Dipstick Urinalysis | Y | | Y |
| ECGs | | | |
| Heart Rate (beats/min) | | | |
| PR Interval (msec) | | | |
| QRS Interval (msec) | | | |
| QT Interval (msec) | | | |
| QTcF Interval (msec) | | | Y |
| <ul> <li>Highest post-baseline QTcF &gt;450 msec</li> </ul> | Y | | 1 |
| <ul> <li>Highest post-baseline QTcF &gt;480 msec</li> </ul> | | | |
| <ul> <li>Highest post-baseline QTcF &gt;500 msec</li> </ul> | | | |
| <ul> <li>Maximum CFB of QTcF &gt; 30 msec</li> </ul> | | | |
| <ul> <li>Maximum CFB of QTcF &gt; 60 msec</li> </ul> | | | |
| Overall interpretation & Clinical Significance | | | Y |
| Vital Signs & Body Measurements | • | • | |
| Heart Rate (beats/min) | | | |
| Systolic Blood Pressure (mmHg) | 7, 7, | | 37 |
| Diastolic Blood Pressure (mmHg) | Y | | Y |
| Temperature (°C) | | | |
| Other Safety Data Listings | | | |
| Physical Examination | | | Y |
| ECOG Performance Status | | | Y |
| Pregnancies | | | Y |

#### 9.2. MTD and DLT Events

#### Dose Escalation and Determination of MTD 9.2.1.

The dose escalation and determination of the MTD and/or recommended dose will be guided by a BLRM with overdose control (EWOC) (see protocol section 4.1.1, and appendix F). The starting dose and some of the provisional dose levels that could be evaluated during this study are described in protocol Table 1. The doses to be investigated are not limited to the provisional dose level listed in the table. The proposed dose escalation scheme for WTX-330 includes a dose level -1 with a 50% lower dose than the first dose level, in the event that the first dose level is not tolerated. Doses are selected based on patient safety data and are subject to satisfying the EWOC criteria under BLRM. The RDE will be determined by the Dose Escalation Committee (DEC) considering all available data and is not stipulated in this SAP.

#### 9.2.2. **DLT Events**

The DLT will be listed using the DLT-evaluable set.

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



#### 9.3. Adverse Events (AEs)

Unless otherwise specified, adverse events will be summarized using frequency tables by System Organ Class (SOC) and Preferred Term (PT).

#### 9.3.1. **AE-related Definitions and Derivations**

#### 9.3.1.1. **Coding and Grading**

All adverse events (AEs) will be coded using MedDRA® 26.0 and will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 (see Subsection 15.1), except for Cytokine Release Syndrome which will be graded with American Society for Transplantation and Cellular Therapy (ASTCT) Grade.

If severity grading is missing, the event will be graded as severe (Grade 3) unless the event being recorded is leading to life-threatening or death and will be graded accordingly as Grade 4 (life-threatening) or 5 (death).

#### 9.3.1.2. Relatedness Assessment

The investigator will category the relatedness of AE to study drugs as 'Definite,' 'Probable,' 'Probable,' 'Unlikely,' and 'Unrelated.' In safety analyses, 'Definite,' 'Probable,' 'Possible' or missing relationship will be summarized as 'Related,' and other relationship will be treated as 'Unrelated."

#### 9.3.1.3. **Treatment Emergent Adverse Events (TEAEs)**

A TEAE is defined as an AEs that emerges or worsens (ie increase in CTCAE grade/ASTCT grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

#### 9.3.1.4. **TEAEs of Special Interest (AESIs)**

TEAEs of special interest (AESIs) include

- >=Grade 2 CRS
- >= Grade 3 Oral Mucositis
- Hy's Law or >= Grade 3 increased ALT or AST

### **Planned Analysis of Adverse Events**

Using the Safety Analysis Set, TEAE summaries will be presented by primary SOC and PT. Summaries will be presented by analysis groups described in Subsection 6.2. Although a PT or SOC may be reported more than once for a subject, each subject will only be counted once within the SOC or PT.

Number and percentage of subjects with the following TEAE categories will be presented in overview TEAE tables. Number and percentage of subjects with the following TEAE categories will be summarized by primary SOC and PT.

- All TEAEs
- TEAEs related to WTX-330
- All Serious TEAEs
- Serious TEAEs related to WTX-330
- Grade 3 or higher TEAEs
- Grade 3 or higher TEAEs related to WTX-330
- TEAEs leading to WTX-330 withdrawn
- WTX-330-related TEAEs leading to WTX-330 withdrawn

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |





- TEAEs leading to WTX-330 modification (including Dose Delayed, Dose Interrupted, Dose Reduced, Infusion Rate Reduced)
- WTX-330-related TEAEs leading to any study drug modification
- TEAEs leading to deaths
- **TEAEs of Special Interest**
- Immune Related TEAEs
- Infusion Related Reaction
- Cytokine Release Syndrome (CRS)
- DLT

The number and percentage of subjects with TEAEs, TEAEs related to each study drug, Serious TEAEs, Serious TEAEs related to each study drug will also be summarized by PT and/or SOC/PT/Maximum CTCAE/ASTCT Grade.

Subject listing(s) will be provided for subjects with all TEAEs, serious TEAEs, AESIs, Immune Related TEAEs, Infusion Related Reaction, Cytokine Release Syndrome, TEAE leading to death, TEAE leading to drug withdrawn, and TEAE leading to drug modification will be listed. All AEs will also be listed.

#### 9.4. **Deaths**

The number and percentage of subjects who died on study, within 30 days after the last study drug administration day, and beyond 30 days after the last study drug administration, as well the number and percentage of subjects who died due to each primary cause will be summarized using the Safety Analysis Set.

Death details as collected in the eCRF will be listed.

#### 9.5. **Clinical Safety Laboratory Tests**

For laboratory values in the form of  $\langle x, \leq x \rangle$ , below lower quantification limit, etc., the value will be imputed as x/2 or half of the lower quantification limit for the purpose of numerical descriptive summary. For laboratory values in the form of >x,  $\ge x$ , above upper quantification limit, etc., the value will be imputed as x or upper quantification limit for the purpose of numerical descriptive summary. When such imputation occurs, footnotes will be presented to clarify the imputation rule. The original laboratory values will be presented in data listings.

Hematology tests include Red blood cell (RBC) count, hemoglobin (Hb), hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH); white blood cell (WBC) count and differential count including, absolute lymphocyte count (ALC), and absolute neutrophil count (ANC), leukocytes with differential (manual microscopic review is performed only if WBC count and/or differential values are out of reference range); platelet count.

Clinical chemistry tests include Calcium, magnesium, potassium, sodium, bicarbonate, chloride phosphate, albumin, total blood urea nitrogen (BUN), C-reactive protein (CRP), creatinine, urate, estimated glomerular filtration rate, glucose, Alanine transaminase (ALT), aspartate transaminase (AST), bilirubin, alkaline phosphatase (ALP), lactic acid dehydrogenase (LDH), gamma-glutamyl transferase (GGT), Triiodothyronine (T3), thyroid-stimulating hormone (TSH), thyroxine (T4).

Coagulation laboratory tests Prothrombin time (PT) or International normalized ratio (INR), and Partial thromboplastin time (PTT) or Activated partial thromboplastin time (APTT).

Urinalysis tests include Dipstick (bilirubin, glucose, ketones, leukocytes, nitrite, occult blood, pH, protein, specific gravity, turbidity and colour, and urobilinogen) or microscopy.

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |





The value of hematology tests, coagulation tests, and chemistry tests will be graded with CTCAE 5.0. If a parameter includes both hypo- and hyper- CTCAE grade derivation, hypo- and hyper- will be derived separately. If the baseline is not CTCAE gradable (e.g., AST increase), the baseline measurement will be categorized as low/normal/high according to reference ranges.

- Quantitative laboratory data will be summarized using descriptive statistics (Subsection 15.2) of actual values and changes from baseline to each visit over time.
- Shift of the worst post-baseline CTCAE grade from baseline will be summarized as well.

Some tests (including red blood cells (RBC) count, hematocrit, Chloride, lactic acid dehydrogenase, prothrombin time, etc) with normal range and are not CTCAE gradable. The shift of these tests from baseline low/normal/high to lowest/highest post-baseline will be prepared.

The number and percentage of patients with elevated AST, ALT, total bilirubin, and alkaline phosphatase will be summarized for safety analysis set. Elevations will be summarized as a function of the ULN.

- 3 × ULN, 5 × ULN, 10 × ULN, and 20 × ULN elevations of AST, ALT, and either ALT or AST.
- $>1.5 \times ULN$  and  $>2 \times ULN$  elevations of Total bilirubin.
- Any elevations of ALP  $> 1.5 \times ULN$ .
- Elevation of ALT/AST ( $>3 \times$  ULN) accompanied by Total bilirubin ( $>1.5 \times$  ULN,  $>2 \times$  ULN).

A separate listing will also be provided for all hematology, coagulation, clinical chemistry (including thyroid function tests) and urinalysis. Laboratory values that are outside the normal range will also be flagged in the data listings, along with corresponding normal ranges. Any out-of-range values that are identified by the investigator as being clinically significant will also be shown in the data listing.

For all NCI-CTCAE programmatically gradable laboratory tests, separate listings will be provided for all Grade 3 or higher abnormal lab results (in either direction) together with corresponding baseline results.

#### 9.6. **Electrocardiograms (ECG)**

For triplicate ECG measurements, the mean of all assessments at each scheduled time point will be used for descriptive summarization purpose; however, all ECG measurements will be provided in data listings.

Local-read ECG data will be listed overall and a separate listing for any clinically significant finding in ECG values will be provided.

Absolute and CFB values for PR Interval, OT Interval, OTcF, ORS Duration and HR will be summarized descriptively by visit and by dose level in escalation phase and by arm in expansion phase. QTcF will be calculated with QT/(RR)<sup>1/3</sup>.

The frequency and percentage of subjects will be tabulated descriptively for the following:

- Highest post-baseline QTcF >450 msec
- Highest post-baseline QTcF >480 msec
- Highest post-baseline QTcF >500 msec
- Maximum CFB of OTcF > 30 msec
- Maximum CFB of QTcF > 60 msec

#### 9.7. Vital Signs and Body Measurements

The absolute values of vital sign and body measurements (including weight, systolic blood pressure, diastolic blood pressure, HR, and temperature) and the CFB measurements will be summarized descriptively for each analysis group over scheduled time points (visits) as defined in Subsection 6.2.

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



The number and percentage of patients with the following notably abnormal vital signs and body measurements will be presented by visit:

- Clinically notable elevated values:
  - o Systolic BP: ≥ 180 mmHg and an increase ≥ 20 mmHg from baseline
  - O Diastolic BP:  $\geq 105$  mmHg and an increase  $\geq 15$  mmHg from baseline
  - Weight: Increase of  $\ge 10\%$  from baseline
  - Heart rate:  $\geq 120$  bpm with an increase of  $\geq 15$  bpm from baseline
  - $\circ$  Temperature:  $> 38^{\circ}$  C
- Clinically notable decrease values:
  - o Systolic BP: ≤90 mmHg and a decrease ≥ 20 mmHg from baseline
  - o Diastolic BP: ≤ 50 mmHg and a decrease ≥ 15 mmHg from baseline
  - $\circ$  Weight: decrease of  $\geq 10\%$  from baseline
  - Heart rate:  $\leq$  50 bpm and a decrease  $\geq$  15 bpm from baseline
  - Temperature: < 35° C

Vital signs will be provided in a data listing by subject using the Safety Analysis Set.

### 9.8. Physical Examination

Any clinically significant findings at Screening should be reported on the Medical History; otherwise, new/worsened clinically significant findings should be reported as Adverse Events.

All physical examination data will be listed.

### 9.9. ECOG Performance Status

ECOG performance status will be provided in a data listing.

### 9.10. Pregnancies

Pregnancy test results will be provided in a data listing using the Safety Analysis Set.

### 10. Pharmacokinetics

# 10.1. Schedule for PK Sampling

On Cycle 1 Day  $1\sim$  Day 8 and Cycle 2 Day  $1\sim$  Day 8 of Dose Escalation, the samples will be collected at Pre-dose, Immediately after ( $\pm 5$  minutes) WTX-330 infusion, 4 hours ( $\pm 30$  minutes) post start of WTX-330 infusion, 8 hours ( $\pm 30$  minutes) post start of WTX-330 infusion, 24 hours ( $\pm 2$  hours) post start of WTX-330 infusion, 168 hours ( $\pm 4$  hours) post start of WTX-330 Infusion. On other visits, the samples will be collected at Pre-dose, Immediately after ( $\pm 5$  minutes) WTX-330 infusion. On Dose Expansion, the samples will be collected at Pre-dose, Immediately after ( $\pm 5$  minutes) WTX-330 infusion.

### 10.2. Pharmacokinetic Parameters

Plasma concentrations of WTX-330 and free IL-12 will be determined with a validated bioanalytical assay. PK parameters for WTX-330 and free IL-12 at Cycle 1 and Cycle 2 of Dose Escalation will be calculated from plasma concentrations using noncompartmental analyses:  $C_{max}$ ,  $T_{max}$ ,  $t\frac{1}{2}$ ,  $AUC_{0-14d}$ .

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |





# 10.3. Analysis of Pharmacokinetic Parameters

The PK Analysis Set will be used for summaries of all PK data.

WTX-330 and free IL-12 plasma concentrations will be summarized by visit and dose cohort (n, mean, geometric mean, standard deviation, coefficient of variation, median, Min and Max).

 $C_{max}$ ,  $T_{max}$ ,  $t\frac{1}{2}$ ,  $AUC_{0-14d}$  at Cycle 1 and Cycle 2 will be summarized with descriptive sctatistics (n, mean, geometric mean, standard deviation, coefficient of variation, median, Min and Max).  $T_{max}$  will be summarized with descriptive statistics (n, mean, standard deviation, median, Min and Max).

Plots of mean WTX-330 and free IL-12 plasma concentrations versus time will be generated by dose group and phase in linear and semi-logarithmic form. Individual plasma concentrations versus time graphs will also be provided.

### 11. Anti-Drug Antibody (ADA)

ADA Samples will be collected at pre-dose on each schedule and unscheduled visit.

Anti-drug antibody (ADA) data of WTX-330 will be provided in listing. ADA will be summarized in tabular by visit under the following categories:

- N (%) of patients with ADA at baseline (i.e. ADA detectable in the Cycle 1 Day 1 pre-dose sample)
- N (%) of patients with post-dose ADA (i.e. ADA detectable in any pre-dose sample from Cycle 1 Day 15 and later)
- N (%) of patients with treatment-induced ADA, defined as those patients with no ADA at baseline and one or more post-treatment (Cycle 1 Day 15 and later) ADA-positive sample.
- N (%) of patients with treatment-boosted ADA, defined as patients with a positive baseline ADA result who had one or more post-treatment (Cycle 1 Day 15 and later) ADA result with a higher titer than that of the baseline ADA sample.
- N (%) of patients with treatment-unaffected ADA, defined as patients with a positive baseline ADA result who had post-treatment (Cycle 1 Day 15 and later) ADA result with a lower titer than that of the baseline ADA sample.



| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |





| Protocol Number: WTX-330x2101 | SAP v2.0 [26Feb2025] |
|---|---|
| QMS Document Name: Statistical Analysis Plan Template(EN) | |

|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |
| QMS Document Name: Statistical Analysis Plan Template(EN) | |



| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |
|---------------------------------------------|--------------------------|





# 13. Multiplicity

No formal hypothesis testing will be performed on efficacy and safety endpoints.

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



### 14. References

- Cheson BD, Fisher RI, Barrington SF, et al. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol 2014;32(27):3059–68.
- Clopper, C. J., & Pearson, E. S. (1934). The Use of Confidence or Fiducial Limits Illustrated in the Case of the Binomial. *Biometrika*, 26, 404-413.
- Crowley, J., & Brookmeyer, R. (1982). A Confidence Interval for the Median Survival Time. *Biometrics*, 38, 29-41.
- Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, et al. New response evaluation criteria in solid tumors: revised RECIST guideline (version 1.1). Eur J Cancer 2009;45:228-47.
- Kaplan, E. L., & Meier, P. (1958). Nonparametric Estimation from Incomplete Observations. *Journal of the American Statistical Association*, 53, 457-481.
- Miller, R., & Siegmund, D. (1982). Maximumally Selected Chi Square Statistics. *Biometrics*, 38, 1011-1016.
- Seymour, L., Bogaerts, J., Perrone, A., Ford, R., Schwartz, L. H., Mandrekar, S., . . . RECIST working group. (2017). iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. *The Lancet Oncology, 18*, e143--e152.

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



### 15. Appendices

# 15.1. Appendix 1: Referenced Study Documents, Software and Standards

| Document, Software, or Standard | Version / Date |
|---|---|
| Protocol | Amendment V02 / 06 April 2023 |
| Electronic Case Report Form (eCRF) | V3.0 30JUN2023 |
| SAS® Software | 9.4 |
| National Cancer Institute-Common Terminology Criteria for | 5.0 / 27NOV2017 |
| Adverse Events (NCI-CTCAE) | |
| Medical Dictionary for Regulatory Activities (MedDRA®) | 26 or higher / latest version at database |
| | lock (DBL) |
| World Health Organization Drug Dictionary (WHODrug) | B3 Global / latest version at DBL |
| | (March 2023 or later) |
| Response Evaluation Criteria in Solid Tumours (RECIST) | 1.1 / 2009 |
| Immune-Response Evaluation Criteria in Solid Tumors | 2017 |
| (iRECIST) | |
| Lugano classification | 2014 |

15.2. Appendix 2: Descriptive Statistical Summaries

### **Descriptive Statistical Summaries**

### **Numerical Data**

Numerical variables will be summarized using descriptive statistics, displaying

- the number of subjects in the analysis group,
- the number of subjects with data,
- sample mean,
- sample standard deviation (calculated as the square root of an unbiased variance estimate),
- sample median,
- minimum (min) and
- maximum (max).

### Categorical Data

- Categorical variables will be summarized by using frequency counts and percentages.
- The number of subjects with missing values will be displayed.
- Unless otherwise specified, the denominators used for calculating sample proportions will be the number of subjects in the analysis group (Subsection 6.2) of the specified statistical analysis set (or a subset of the statistical analysis set under use).
- For select ordinal categorical variables, cumulative counts and cumulative percentages may be presented, if appropriate.

# 15.3. Appendix 3: Data Display Conventions

| Data Display Conventions | |
|---|---|
| Precision | |
| QMS Document Name: Statistical Analysis Plan Template(EN) | |
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



### **Data Display Conventions**

- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non-eCRF sources will follow the same principles as described below but may be adjusted to a clinically interpretable number of decimal places (dp).
- Means and medians will be presented by 1 additional decimal place, and standard deviation will be
  presented by 2 additional decimal places than the standard presentation level of the respective data.
  Minimum and maximum values will be presented using the same number of decimal places as the
  original data. Standard errors and CI limits will be presented by 1 additional decimal place than
  corresponding point estimates.
- If not otherwise stated, percentages will be presented to 1 decimal place. However, if the percentage (or estimated proportion) is 100% exactly, no decimal place will be shown, whereas presented as 100.0% implies that the percentage is in the half-open interval [99.95%, 100.0%).
- Reasonable number of dps will be adjusted for proper presentation and interpretation. The maximum number of decimal places reported shall be 4 for any summary statistic, unless otherwise stated.

| Default Presentation Precision | | |
|---|---|---|
| Name | Description | Decimal Place (dp) |
| N | Number of Subjects in the Treatment Group | Always 0 decimal. |
| n | Number of Subjects with Non-Missing Values | Always 0 decimal. |
| % | Percentage | 1 decimal for categorical data |
| Mean | Arithmetical Mean | 1 more decimal than original data |
| StdDev | Standard Deviation | 2 more decimal than original data |
| Median | Median | 1 more decimal than original data |
| Min. | Minimum | Same as original data |
| Max. | Maximum | Same as original data |
| SE | Standard Error | 1 more decimal than the corresponding |
| | | point estimate |
| CI | Confidence Interval | 1 more decimal Than the corresponding |
| | | point estimate |
| P value | P value | 3 significant digits |

### **Rounding Rules**

- In general, explicit rounding will only occur when presenting data but not when analyzing data. Thus, data in recorded in the Analysis Data Sets (e.g., ADaM data sets) will not be rounded.
- By default, presented data will be rounded to the nearest required presentation precision, with a "round ties to even" tie-breaking rule according to IEEE 754-2019.
- When presenting CIs, the lower interval limit will always be rounded down and the upper interval limit will always be rounded up in order preserve the claimed (exact or asymptotic) confidence level. When either limit is outside of the parameter space (e.g., below 0 or above 1 for proportions), the interval will be truncated at the boundary of the parameter space.

### **Zero Count Presentation**

- For descriptive summaries, if the number of subjects in a category is 0, then percentage will not be displayed, and only a count of 0 will be shown.
- However, structural zeros (e.g., when the count is deemed to be 0 before obtaining actual data), missing data or inapplicable/unevaluable summaries will be presented as –, NA or NE (not applicable or not evaluable, respectively).

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |



### **Data Display Conventions**

### **Sorting in Displays**

- In data listings, data records will be sorted by study phase (escalation vs expansion), therapy (monotherapy vs combination therapy), dose level / arm, site, and subject, and when appropriate by visit, scheduled time point or other identifiers for sequence or type of observation.
- In descriptive summaries involving categorical variables only, e.g., summaries of
  - medical history by SOC and PT,
  - · medications by ATC category and PN, and
  - adverse events by SOC and PT,

the categories and sub-categories will be presented by decreasing frequency using sorting variables in the following preference order:

- 1. Total count (irrespective of whether the total column is shown or not)
- Count from higher dose level for escalation part or from higher arm code for expansion part (D > C > B > A)
- 3. Alphabetical order of the category label

Sorting variables with lower preference will only be used if ties remain using sorting variables with higher preference.

# 15.4. Appendix 4: Study Day, Duration, Period, Visit and Analysis Windows

### Study Day, Duration, Period, Visit and Analysis Windows

#### Study Day

For each study subject, Day 1 is defined as the date corresponding to the first administration of any study drug.

Study days after Day 1 are calculated as the number of days from Day 1:

- Study Day = Date of interest Date of Day 1 + 1, if the date of interest is on or after date of Day 1;
- Study Day = Assessment date Date of Day 1, if the assessment date is prior to Day 1.
- Study Day is set to missing if the date of interest is missing.

### **Time Unit and Duration**

- Unless otherwise specified, day is the primary time unit for derived time and duration.
- Derived time units include
  - 1. Week = 7 days
  - **2.** Month = 30.4375 days,
  - 3. (Gregorian) Year = 365.25 days = 12 months.

Thus, 1 month and 4 weeks are considered different.

 Unless otherwise specified, duration of time is defined from the starting day through the ending day, inclusive of both boundary days.

### Study Periods

Screening period: beginning on the day of informed consent, or Study Day −28, whichever is latest, and ending on Day −1

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |


Protocol Number: WTX-330x2101

### Study Day, Duration, Period, Visit and Analysis Windows

- Treatment period: beginning on Study Day 1 and ending on the last day of the End of Treatment (EoT) visit. In case that the EoT visit is missed for any reason, the treatment period will end on the 28th day since the last dose of any study drug.
- Safety follow-up period: 30-day safety follow-up period since the first day after the treatment period and or study discontinuation date, whichever occurs first.
- Unless otherwise specified, events in the screening period are considered as pre-treatment, events
  in the treatment period and safety follow-up period are considered as on-treatment.

### **Time Points and Assessment Windows**

- Subject visits will be presented according to the nominal visit and/or time points as obtained on the eCRF.
- Unscheduled visits will be included in subject data listing but will not be presented in descriptive summary tables, except for deriving time to event (TTE) variables or otherwise specified.

### 15.5. Appendix 5: Derived Data And Definitions

#### **Derived Data And Definitions**

### **Baseline & Change From Baseline**

- The baseline is defined to be the last non-missing value prior to the first WTX-330 dose.
  - For assessments performed on Day 1, if the time of the day is missing but scheduled time
    point is recorded as pre-dose, the assessment may be considered the baseline assessment for
    the respective study procedures.
- Change from Baseline (CFB) = Post-baseline Assessment Baseline Assessment.
  - CFB will be set to missing if corresponding post-baseline assessment or the baseline assessment is missing
- Percent CFB =  $100 \times (CFB / Baseline Assessment)$  %, with the following exceptions:
  - o If both CFB and baseline assessment are 0, the corresponding percent CFB will be set to 0.
  - If baseline assessment is 0 or missing but the CFB is non-zero, the percent CFB will be set to missing.

### Age

Age at informed consent will be calculated from the date of birth to the date of informed consent.

### Prior and Concomitant Medications, Procedures, and Medical Conditions

- Prior medications all medications that ended before Day 1.
- Concomitant medications all non-study drug medications used on/after day 1.
- Prior and concomitant procedures are defined analogously.

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |
| CONFIDE | CONFIDENTIAL |



Protocol Number: WTX-330x2101 SAP v2.0 [26Feb2025]

#### **Derived Data And Definitions**

If the start and/or end dates are partially recorded or missing completely, refer to Subsection 15.6 for the determination of prior vs concomitant status.

#### 15.6. Appendix 6: Premature Withdrawals & Handling of Missing Data

### Premature Withdrawals & Handling of Missing Data

#### Premature Withdrawals

During the dose escalation phase, if a subject in Cycle 1 discontinues, holds, or modifies WTX-330 dose for a reason other than a DLT as reviewed by DEC and is not followed for safety for a minimum of 28 days, the subject may be replaced.

For the Dose Expansion Phase, subjects will be replaced if they do not have at least one post-baseline efficacy assessment and did not discontinue due to clinical progression.

### Handling of Missing or Partial Dates

In the presence of missing or partial dates, the determination of "prior" and "concomitant" status for nonstudy drug medications, and TEAE will follow the rules below:

### Partial start date for Adverse Event, partial start date for Medications, and partial date of diagnosis

- if month and day are missing, and the year is the same as the year of first WTX-330 dose, then assign the date of first WTX-330 dose as start date; else assign Jan 1st of the year.
- if only the day is missing, and the month and year are same as the month and year of first WTX-330 dose, then assign the date of first WTX-330 dose as AE start date; else assign 1st day of the month.
- Compare the imputed date with the date of last known alive/contact; if the imputed date is later than the date of last known alive/contact, then assign the date of last known alive/contact as AE start date.

Partial end date for Adverse Event, and partial end date for Medications:

- Assign DEC 31st of the year if both Month and Day are missing.
- Assign last day of the month if only Day is missing.
- Assign 'ongoing' if Year, Month and Day are missing.
- Compare the imputed date with the date of last known alive/contact; if the imputed date is later than the date of last known alive/contact, then assign the date of last known alive/contact as AE end date.

The data listings will report original data instead of the imputed date. The imputed date will be used to categorized TEAE, Prior/Concomitant Medication.

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |
| CONFIDE | NTIAL |



## 15.7. Appendix 7: List of Abbreviations

| Abbreviation | Description |
|--------------|-----------------------------------------|
| ADA | Anti-drug antibody |
| ADaM | Analysis Data Model |
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| ALP | Alkaline phosphatase |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BOR | Best overall response |
| CD | Cluster of differentiation |
| CFB | Change from baseline |
| CI | Confidence interval |
| COVID-19 | Coronavirus Disease 2019 |
| CR | Complete response |
| CRP | C-reactive protein |
| CRS | Cytokine release syndrome |
| CSR | Clinical Study Report |
| DLT | Dose-limiting toxicity |
| dMMR | Deficient mismatch repair |
| DoR | Duration of response |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Report Form |
| eGFR | Estimated glomerular filtration rate |
| EoT | End of Treatment |
| iBOR | Immune-best overall response |
| iCBR | Immune-clinical benefit rate |
| ICH | International Council for Harmonisation |
| IL | Interleukin |
| iCPD | Immune-confirmed progressive disease |

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |
| CONFIDE | NTIAL |



Protocol Number: WTX-330x2101

| Abbreviation | Description |
|---|---|
| iCR | Immune-complete response |
| iDoR | Immune-duration of response |
| IFN | Interferon |
| IL | Interleukin |
| IL-2R | Interleukin-2 receptor |
| iORR | Immune-overall response rate |
| iPFS | Immune-progression-free survival |
| iPR | Immune-partial response |
| iRECIST | Immune-Response Evaluation Criteria in Solid Tumors |
| iSD | Immune-stable disease |
| iUPD | Immune-unconfirmed progressive disease |
| LDH | Lactic acid dehydrogenase |
| Max. | Maximum |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Min. | Minimum |
| MMR | Mismatch repair |
| mRCC | Metastatic renal cell carcinoma |
| MSI | Microsatellite instability |
| MSI-H | MSI-High |
| MSI-L | MSI-Low |
| MSS | Microsatellite stable |
| MTD | Maximum tolerated dose |
| NCI-CTCAE | National Cancer Institute Common Terminology Criteria for Adverse Events |
| NE | Not evaluable |
| NK (cells) | Natural killer (cells) |
| ORR | Overall response rate |
| OS | Overall survival |
| PD | Progressive disease |
| PFS | Progression-free survival |
| PK | Pharmacokinetic(s) |
| pMMR | Proficient mismatch repair |

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |
| CONFIDE | NTIAL |





Protocol Number: WTX-330x2101

| Abbreviation | Description |
|---|---|
| PN | Preferred name |
| PR (except for PR interval) | Partial response |
| PT | Preferred term |
| PTT | Partial thromboplastin time |
| QTc | QT interval corrected for heart rate |
| QTcF | QT interval corrected for heart rate using Fridericia's formula |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| SAE | Serious adverse events |
| SAP | Statistical Analysis Plan |
| SD | Stable disease |
| SOC | System organ class |
| StdDev | Standard deviation |
| TEAE | Treatment-emergent adverse event |
| TNF | Tumor necrosis factor |
| TTE | Time to event |
| ULN | Upper limit of normal |
| WHODrug | World Health Organization Drug Dictionary |

| QMS Document Name: Statistical Analysis Plan Template(EN) | |
|---|---|
| QMS No (include version ref): STF-015-GL.03 | Document date: 14JUL2022 |
| CONFIDE | NTIAL |

Protocol: WTX-330x2101 Date: 26Feb2025



### Werewolf Therapeutics, Inc.

## A Phase 1 (First-In-Human [FIH]), Multi-Site, Dose Escalation and Expansion Study of WTX-330 in Adult Patients with Advanced or Metastatic Solid Tumors or Lymphoma

### **TFL Shells**

Author: Shuangli Guo

SAP Version: 2.0

Table Shell Version: 2.0

Caidya Code: WWT21330

Date: 26Feb2025

## **Table of Contents**

| Approval and Signature Page | 3 |
|----------------------------------------------------|----|
| Format and Ordering of Treatment Groups | |
| General Display Conventions | |
| Sorting Conventions | |
| Display of Continuous Statistics | 5 |
| Display of Percentages | 5 |
| Display of P-Values | |
| Display of Dates in Subject Data Listings | |
| Display of Missing Values in Subject Data Listings | 6 |
| Modification History | |
| List of Tables | |
| List of Figures | 13 |
| List of Listings | 14 |
| Table Shells | |
| Figure Shells | |
| Listing Shells | |

Date: 26Feb2025

## **Approval and Signature Page**

Approved by:

| Name, Institution, and Job<br>Title | Signature | Date |
|---|---|---|
| Shuangli Guo<br>Senior Manager Biostatistics<br>Caidya | Signed by: Signer Name: Shuangli Guo Signing Reason: I am the author of this document Signing Time: 26-Feb-2025 7:28:54 PM GMT 3F1277AD321D4048BF564AE5BED08E47 | 26-Feb-2025 |
| Oliver Schonborn-<br>Kellenberger<br>Biostatistician<br>Werewolf Therapeutics, Inc. | Signiert von: Oliver Schönborn-Kellenberger Name des Unterzeichners: Oliver Schönborn-Kellenbergingiergrund: Ich genehmige dieses Dokument Signierzeit: 26-Feb-2025 7:59:53 PM GMT 988B94B1FDA24A35AEB8361DCA46EBF3 | 26-Feb-2025<br>erger |

Date: 26Feb2025

### **Format and Ordering of Treatment Groups**

The study includes Dose Escalation and Dose Expansion as the strategy below.



CPI = checkpoint inhibitor; MTD = maximum tolerated dose; Q2W = every 2 weeks; r/r = relapsed/refractory; SOC = standard of care.

Disposition, demographic, baseline characteristics, disease history, efficacy, and safety summaries will be presented as follows.

Dose Escalation will be presented by dose level – additional columns will be added if more dose levels/schedules are tested:

| WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|
| 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | Total |
| mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | |

### Dose Expansion will be presented by Arm:

| | | | | | Arm | ı A | Arm | В | Total |
|------|---|------|----------|----------|-----|---------|-------|---|-------|
| Maka | 7 | 7\ _ | Dationto | ما بدائد | | fanbiab | - CDT | | / |

Note: Arm A = Patients with indications for which a CPI is indicated/approved; Arm B = Patients with tumor types for which CPI therapy is not indicated/approved.

Overall response rate (ORR) and immune-overall response rate (iORR) in Dose Expansion will be further summarized by indication

| | Arm A | | | | Arm B | | | |
|---|---|---|---|---|---|---|---|---|
| | RCC | NSCLC | HNSCC | XXXXX | CC | FL | DLBCL | YYYYY |
| Note: Arm A = Patien | ts with in | dications | for which | a CPI i | s indica | ted/ap | proved; | Arm B = |
| Patients with tumor types for which CPI therapy is not indicated/approved. | | | | | | | | |
| Note: RCC = Renal Cell Carcinoma; NSCLC = Non-small Cell Lung Cancer; HNSCC = Head and | | | | | | | | |
| Neck Squamous Cell Carcinoma; XXXXXX =; CC = Colorectal Carcinoma; FL = Follicular | | | | | | | | |
| Lymphoma; DLBCL = Diffuse Large B-cell Lymphoma; YYYYYY = | | | | | | | | |

Column headers will be updated according to the indication in Arm A and B.

### **General Display Conventions**

Summary tables and subject data listings will be in landscape format. Table titles will be centered.

Date: 26Feb2025

### **Sorting Conventions**

For AE and MH summaries, Primary SOCs and PTs will be ordered by descending count in overall Total (last column in table display). Other summaries will follow table shells layout.

### **Display of Continuous Statistics**

Means and medians will be shown to one more decimal place, and the standard deviation will be shown to two more decimal places than the source data values. In cases where variables are derived and have floating point values (no fixed number of decimal places), an appropriate level of precision will be determined based on the context.

Statistics that cannot be derived will be shown as a dash ("-") in summary tables.

Two-Sided confidence intervals are displayed with a format such as "(xx.x, xx.x)." If a confidence interval cannot be produced due to insufficient data, then a dash ("-") will be shown in place of the entire confidence interval.

### **Display of Percentages**

The following conventions apply for percentages:

- Percentages will be displayed to one decimal place unless otherwise specified
- No percentage will be shown if the corresponding count is 0
- Percentages that are exactly equal to 100% will be displayed as "100%"
- Percentages that round down to 0.0% will be displayed as "<0.1%"
- Percentages that round up to 100.0% will be displayed as ">99.9%"

Percentages are shown in parentheses after the corresponding count such as "25 (5.2%)" where extra spaces are included after the left parenthesis to ensure that decimal places for all percentages align within the same column.

### **Display of P-Values**

Unless otherwise noted, p-values will be displayed as follows:

- P-values between 0.0001 and 0.9999 will be displayed in the format "0.xxxx"
- P-values that are exactly equal to 1 will be displayed as "1.0000"
- P-values <0.0001 will be displayed as "<0.0001"
- P-values >0.9999 and not exactly equal to 1 will be displayed as ">0.9999"

P-values that are descriptive and not associated with a formal test of hypothesis will not be flagged based on statistical significance. The following note will be shown in the table:

```
Note: P-values are for descriptive purposes and are not evaluated for statistical significance.
```

Unless otherwise noted, p-values that are statistically significant will be flagged with an asterisk. The table footnote is dependent on the setting, but the following example footnote is appropriate for many settings:

\* Statistically significant at the 0.05 level.

Date: 26Feb2025

### **Display of Dates in Subject Data Listings**

Dates will be shown in one of the following formats:

- YYYYMMDD for complete dates
- YYYYMM for dates with only a month and year
- YYYY for dates with only a year

Partial dates are not imputed for subject data listings even if such dates are imputed for statistical algorithms. Relative day (if shown) is only derived for complete dates.

Dates will be shown in ISO8601 format as follows:

- DDMMMYYYY for complete dates
- MMMYYYY for dates with only a month and year
- YYYY for dates with only a year

Partial dates are not imputed for subject data listings even if such dates are imputed for statistical algorithms. Relative day (if shown) is only derived for complete dates.

### **Display of Missing Values in Subject Data Listings**

For subject data listings, missing numeric values will be shown as a dash ("-"). Missing character values will be shown as blanks.

### **Modification History**

| Version | Date | Author | Changes from Previous Version |
|---|---|---|---|
| 0.1 | 19Dec2023 | Shuangli Guo | N/A – First Version |
| 0.2 | 12Jun2024 | Shuangli Guo | Add shift tables for Deauville Scale |
| 0.3 | 21Jun2024 | Shuangli Guo | Update footnote in TEAE table based on Werewolf's comments, correct typos |
| 1.0 | 21Jun2024 | Shuangli Guo | Accept changes in version 0.3 |
| 1.1 | 18Feb2025 | Shuangli Guo | Correct Typo Select the TFLs for aCSR based on WW request |
| 1.2 | 25Feb2025 | Shuangli Guo | Correct Typo<br>Add TFLs for free IL-12 PK summary |
| 2.0 | 26Feb2025 | Shuangli Guo | Accept changes/WW edits in draft 1.2 |

Protocol: WTX-330x2101 Date: 26Feb2025

### **List of Tables**

| 14.1 Study Population and Baseline |
|---|
| Table 14.1.1.1 Summary of Analysis Set - Dose Escalation Screened Subjects |
| Table 14.1.1.2.1 Summary of Analysis Set - Dose Expansion Screened Subjects |
| Table 14.1.1.2.2 Summary of Analysis Set - Dose Expansion by Indication Screened Subjects20 |
| Table 14.1.2.1 Summary of Subject Disposition - Dose Escalation Safety Analysis Set |
| Table 14.1.2.2 Summary of Subject Disposition - Dose Expansion Safety Analysis Set |
| Set |
| Table 14.1.3.2 Summary of Deviations from the Clinical Protocol - Dose Expansion Safety Analysis Set |
| 24 |
| Table 14.1.4.1 Summary of Demographic Characteristics - Dose Escalation Safety Analysis Set25 |
| Table 14.1.4.2 Summary of Demographic Characteristics - Dose Expansion Safety Analysis Set27 Table 14.1.5.1.1 Summary of Solid Tumor Disease Characteristics - Dose Escalation Safety Analysis |
| Set |
| Table 14.1.5.1.2 Summary of Solid Tumor Disease Characteristics - Dose Expansion Safety Analysis Set |
| Table 14.1.8.2.1 Summary of Concomitant Medications by WHO Drug ATC Category II and Preferred Term |
| - Dose Escalation Safety Analysis Set |
| Table 14.1.8.2.2 Summary of Concomitant Medications by WHO Drug ATC Category II and Preferred Term |
| - Dose Expansion Safety Analysis Set |
| Table 14.1.9.1 Summary of WTX-330 Exposure, Compliance and Dose Modification - Dose Escalation |
| Safety Analysis Set |
| Table 14.1.9.2 Summary of WTX-330 Exposure, Compliance and Dose Modification - Dose Expansion |
| Safety Analysis Set |
| 14.2 Analyses of Efficacy |
| Table 14.2.1.1 Summary of Best Overall Response, Objective Response Rate, and Clinical Benefit Rate |
| - Dose Escalation Efficacy Evaluable Analysis Set |
| Table 14.2.1.2.1 Summary of Best Overall Response, Objective Response Rate, and Clinical Benefit |
| Rate - Dose Expansion Efficacy Evaluable Analysis Set |
| Rate - Dose Expansion by Type of Disease (Solid Tumor) Efficacy Evaluable Analysis Set $\dots 48$ |

| 14.3 Summaries and Analyses of Safety | J |
|---|---|
| Table 14.3.1.1.1 Overall Summary of Treatment-Emergent Adverse Events - Dose Escalation Safety | |
| Analysis Set51 | 1 |
| Table 14.3.1.1.2 Overall Summary of Treatment-Emergent Adverse Events - Dose Expansion Safety | |
| Analysis Set | 2 |
| Table 14.3.2.1.1 Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred | _ |
| Term - Dose Escalation Safety Analysis Set | 3 |
| Table 14.3.2.1.2 Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred | |
| Term - Dose Expansion Safety Analysis Set | |
| Table 14.3.2.2.1 Summary of WTX-330-related Treatment-Emergent Adverse Events by System Organ Class | |
| and Preferred Term - Dose Escalation Safety Analysis Set | |
| Table 14.3.2.2.2 Summary of WTX-330-related Treatment-Emergent Adverse Events by System Organ Class | |
| and Preferred Term - Dose Expansion Safety Analysis Set | + |
| Organ Class and Preferred Term - Dose Escalation Safety Analysis Set | 1 |
| Table 14.3.2.3.2 Summary of Treatment-Emergent Adverse Events with Grade 3 or Higher by System | Т |
| Organ Class and Preferred Term - Dose Expansion Safety Analysis Set | 4 |
| Table 14.3.2.4.1 Summary of WTX-330-related Treatment-Emergent Adverse Events with Grade 3 or | • |
| Higher by System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set | 4 |
| Table 14.3.2.4.2 Summary of WTX-330-related Treatment-Emergent Adverse Events with Grade 3 or | |
| Higher by System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set55 | 5 |
| Table 14.3.2.5.1 Summary of Treatment-Emergent Adverse Events Leading to WTX-330 Withdrawal by | |
| System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set | 5 |
| Table 14.3.2.5.2 Summary of Treatment-Emergent Adverse Events Leading to WTX-330 Withdrawal by | |
| System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set $\dots \dots \dots$ | 5 |
| Table 14.3.2.6.1 Summary of WTX-330-related Treatment-Emergent Adverse Events Leading to WTX-330 | |
| Withdrawal by System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set $55$ | 5 |
| Table 14.3.2.6.2 Summary of WTX-330-related Treatment-Emergent Adverse Events Leading to WTX-330 | _ |
| Withdrawal by System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set55 | ) |
| Table 14.3.2.7.1 Summary of Treatment-Emergent Adverse Events Leading to WTX-330 Modification by | , |
| System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set | ) |
| Table 14.3.2.7.2 Summary of Treatment-Emergent Adverse Events Leading to WTX-330 Modification by | 6 |
| System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set $\dots$ 56 | J |

| Table 14.3.2.8.1 Summary of WTX-330-related Treatment-Emergent Adverse Events Leading to WTX-330 |
|---|
| Modification by System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set % |
| Table 14.3.2.8.2 Summary of WTX-330-related Treatment-Emergent Adverse Events Leading to WTX-330 |
| Modification by System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set § Table 14.3.2.9.1 Summary of Immune Related Treatment-Emergent Adverse Events by System Organ Class |
| and Preferred Term - Dose Escalation Safety Analysis Set |
| Table 14.3.2.9.2 Summary of Immune Related Treatment-Emergent Adverse Events by System Organ Class |
| and Preferred Term - Dose Expansion Safety Analysis Set |
| Table 14.3.2.10.1 Summary of Treatment-Emergent Adverse Events of Infusion Related Reaction by |
| System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set |
| System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set |
| Table 14.3.2.11.1 Summary of Treatment-Emergent Adverse Events of Cytokine Release Syndrome by |
| System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set |
| Table 14.3.2.11.2 Summary of Treatment-Emergent Adverse Events of Cytokine Release Syndrome by |
| System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set |
| Table 14.3.2.12.1 Summary of Treatment-Emergent Adverse Events of Special Interest by Special |
| Interest Category and Preferred Term - Dose Escalation Safety Analysis Set |
| Table 14.3.2.12.2 Summary of Treatment-Emergent Adverse Events of Special Interest by Special |
| Interest Category and Preferred Term - Dose Expansion Safety Analysis Set |
| Table 14.3.2.13.1 Summary of Treatment-Emergent Adverse Events by System Organ Class, Preferred |
| Term, and Maximum CTCAE/ASTCT Grade - Dose Escalation Safety Analysis Set |
| Term, and Maximum CTCAE/ASTCT Grade - Dose Expansion Safety Analysis Set |
| Table 14.3.2.14.1 Summary of WTX-330-related Treatment-Emergent Adverse Events by System Organ |
| Class, Preferred Term, and Maximum CTCAE/ASTCT Grade - Dose Escalation Safety Analysis Set |
| Table 14.3.2.14.2 Summary of WTX-330-related Treatment-Emergent Adverse Events by System Organ |
| Class, Preferred Term, and Maximum CTCAE/ASTCT Grade - Dose Expansion Safety Analysis Set |
| Table 14.3.2.15.1 Summary of Treatment-Emergent Adverse Events by Preferred Term - Dose Escalation |
| Safety Analysis Set |
| Table 14.3.2.15.2 Summary of Treatment-Emergent Adverse Events by Preferred Term - Dose Expansion |
| Safety Analysis Set |
| Table 14.3.3.1.1 Summary of Treatment-Emergent Serious Adverse Events by System Organ Class and |
| Preferred Term - Dose Escalation Safety Analysis Set |

| Table 14.3.3.1.2 Summary of Treatment-Emergent Serious Adverse Events by System Organ Class and |
|---|
| Preferred Term - Dose Expansion Safety Analysis Set |
| Table 14.3.3.2.1Summary of WTX-330-related Treatment-Emergent Serious Adverse Events by System |
| Organ Class and Preferred Term - Dose Escalation Safety Analysis Set $\dots \dots 63$ |
| Table 14.3.3.2.2 Summary of WTX-330-related Treatment-Emergent Serious Adverse Events by System |
| Organ Class and Preferred Term - Dose Expansion Safety Analysis Set |
| Table 14.3.3.3.1 Summary of Treatment-Emergent Serious Adverse Events by System Organ Class, |
| Preferred Term and Maximum CTCAE /ASTCT Grade - Dose Escalation Safety Analysis Set64 |
| Table 14.3.3.3.2 Summary of Treatment-Emergent Serious Adverse Events by System Organ Class, |
| Preferred Term and Maximum CTCAE /ASTCT Grade - Dose Expansion Safety Analysis Set64 |
| Table 14.3.3.4.1 Summary of WTX-330-related Treatment-Emergent Serious Adverse Events by System |
| Organ Class, Preferred Term and Maximum CTCAE /ASTCT Grade - Dose Escalation Safety Analysis Set 64 |
| Table 14.3.3.4.2 Summary of WTX-330-related Treatment-Emergent Serious Adverse Events by System |
| Organ Class, Preferred Term and Maximum CTCAE /ASTCT Grade - Dose Expansion Safety Analysis Set $64$ |
| Table 14.3.3.5.1 Summary of Treatment-Emergent Serious Adverse Events by Preferred Term - Dose |
| Escalation Safety Analysis Set |
| Table 14.3.3.5.2 Summary of Treatment-Emergent Serious Adverse Events by Preferred Term - Dose |
| Expansion Safety Analysis Set |
| Table 14.3.3.6.1 Summary of WTX-330-related Treatment-Emergent Serious Adverse Events by Preferred |
| Term - Dose Escalation Safety Analysis Set |
| Table 14.3.3.6.2 Summary of WTX-330-related Treatment-Emergent Serious Adverse Events by Preferred |
| Term - Dose Expansion Safety Analysis Set |
| Table 14.3.3.7.1 Summary of Treatment-Emergent Adverse Events Leading Death by System Organ Class |
| and Preferred Term - Dose Escalation Safety Analysis Set |
| Table 14.3.3.7.2 Summary of Treatment-Emergent Adverse Events Leading Death by System Organ Class |
| and Preferred Term - Dose Expansion Safety Analysis Set |
| Table 14.3.3.8.1 Summary of Death - Dose Escalation Safety Analysis Set |
| Table 14.3.3.8.2 Summary of Death - Dose Expansion Safety Analysis Set |
| Table 14.3.7.1.1 Summary of Hematology Laboratory by Visit - Dose Escalation Safety Analysis Set 68 |
| Table 14.3.7.1.2 Summary of Hematology Laboratory by Visit - Dose Expansion Safety Analysis Set 69 |
| Table 14.3.7.1.3 Shift of Hematology CTCAE Grade from Baseline to Worst Post-baseline - Dose |
| Escalation Safety Analysis Set |
| Table 14.3.7.1.4 Shift of Hematology CTCAE Grade from Baseline to Worst Post-baseline - Dose |
| Expansion Safety Analysis Set71 |

| Table 14.3.7.1.5 Shift of Hematology Tests without CTCAE Grade from Baseline to Lowest/Highest |
|---|
| Post-baseline - Dose Escalation Safety Analysis Set |
| Table 14.3.7.1.6 Shift of Hematology Tests without CTCAE Grade from Baseline to Lowest/Highest |
| Post-baseline - Dose Expansion Safety Analysis Set |
| Table 14.3.7.2.1 Summary of Chemistry Laboratory by Visit - Dose Escalation Safety Analysis Set74 |
| Table 14.3.7.2.2 Summary of Chemistry Laboratory by Visit - Dose Expansion Safety Analysis Set 74 |
| Table 14.3.7.2.3 Shift of Chemistry CTCAE Grade from Baseline to Worst Post-baseline - Dose |
| Escalation Safety Analysis Set |
| Table 14.3.7.2.4 Shift of Chemistry CTCAE Grade from Baseline to Worst Post-baseline - Dose |
| Expansion Safety Analysis Set |
| Table 14.3.7.2.5 Shift of Chemistry Tests without CTCAE Grade from Baseline to Lowest/Highest Post- |
| baseline - Dose Escalation Safety Analysis Set |
| Table 14.3.7.2.6 Shift of Chemistry Tests without CTCAE Grade from Baseline to Lowest/Highest Post- |
| baseline - Dose Expansion Safety Analysis Set |
| Table 14.3.7.2.7 Summary of Clinically Significant Liver Function Tests - Dose Escalation Safety |
| Analysis Set |
| Table 14.3.7.2.8 Summary of Clinically Significant Liver Function Tests - Dose Expansion Safety |
| Analysis Set |
| Table 14.3.7.3.1 Summary of Coagulation Laboratory by Visit - Dose Escalation Safety Analysis Set $78$ |
| Table 14.3.7.3.2 Summary of Coagulation Laboratory by Visit - Dose Expansion Safety Analysis Set 78 |
| Table 14.3.7.3.3 Shift of Coagulation CTCAE Grade from Baseline to Worst Post-baseline - Dose |
| Escalation Safety Analysis Set |
| Table 14.3.7.3.4 Shift of Coagulation CTCAE Grade from Baseline to Worst Post-baseline - Dose |
| Expansion Safety Analysis Set |
| Table 14.3.7.3.5 Shift of Coagulation Tests without CTCAE Grade from Baseline to Lowest/Highest |
| Post-baseline - Dose Escalation Safety Analysis Set |
| Table 14.3.7.3.6 Shift of Coagulation Tests without CTCAE Grade from Baseline to Lowest/Highest |
| Post-baseline - Dose Expansion Safety Analysis Set |
| Table 14.3.8.1 Summary of Vital Signs by Visit - Dose Escalation Safety Analysis Set80 |
| Table 14.3.8.2 Summary of Vital Signs by Visit - Dose Expansion Safety Analysis Set80 |
| Table 14.3.8.3 Summary of Vital Signs Clinically Significant on Treatment - Dose Escalation Safety |
| Analysis Set |
| Table 14.3.8.4 Summary of Vital Signs Clinically Significant on Treatment - Dose Expansion Safety |
| Analysis Set |

| able 14.3.9.1 Summary of Electrocardiograms by Visit - Dose Escalation Safety Analysis Set | 83 |
|---|---|
| able 14.3.9.2 Summary of Electrocardiograms by Visit - Dose Expansion Safety Analysis Set | 83 |
| able 14.3.9.3 Summary of QTcF Categories - Dose Escalation Safety Analysis Set | 84 |
| able 14.3.9.4 Summary of QTcF Categories - Dose Expansion Safety Analysis Set | 85 |
| able 14.4.1.1 Summary of WTX-330 Plasma Concentration (ug/mL) by Timepoint Pharmacokinetic | |
| malysis Set | 86 |
| able 14.4.1.2 Summary of Free IL-12 Plasma Concentration (pg/mL) by Timepoint Pharmacokinetic | |
| malysis Set | 87 |
| able 14.4.2.1 Summary of WTX-330 Pharmacokinetic Parameters Pharmacokinetic Analysis Set | 88 |
| able 14.4.2.2 Summary of Free IL-12 Pharmacokinetic Parameters Pharmacokinetic Analysis Set | 88 |
| able 14.4.3.1 Summary of Anti-drug Antibody for WTX-330 - Dose Escalation and Dose Expansion | |
| nti-Drug Antibody Analysis Set | 89 |

Date: 26Feb2025

### **List of Figures**

| Figure 14.4.1.1.1 Semi-logarithmic Plot and Linear Plot for Individual WTX-330 Plasma | |
|---|---|
| Concentrations versus Time at Cycle 1 - Dose Escalation Pharmacokinetic Analysis Set | 91 |
| Figure 14.4.1.1.2 Semi-logarithmic Plot and Linear Plot for Individual WTX-330 Plasma | |
| Concentrations versus Time at Cycle 2 - Dose Escalation Pharmacokinetic Analysis Set | 92 |
| Figure 14.4.1.1.3 Semi-logarithmic Plot and Linear Plot for Individual Free IL-12 Plasma | |
| Concentrations versus Time at Cycle 1 - Dose Escalation Pharmacokinetic Analysis Set | 92 |
| Figure 14.4.1.1.4 Semi-logarithmic Plot and Linear Plot for Individual Free IL-12 Plasma | |
| Concentrations versus Time at Cycle 2 - Dose Escalation Pharmacokinetic Analysis Set | 92 |
| Figure 14.4.1.2.1 Semi-logarithmic Plot and Linear Plot for Mean WTX-330 Plasma Concentrations | |
| versus Time at Cycle 1 - Dose Escalation Pharmacokinetic Analysis Set | 93 |
| Figure 14.4.1.2.2 Semi-logarithmic Plot and Linear Plot for Mean WTX-330 Plasma Concentrations | |
| versus Time at Cycle 2 - Dose Escalation Pharmacokinetic Analysis Set | 94 |
| Figure 14.4.1.2.3 Semi-logarithmic Plot and Linear Plot for Mean Free IL-12 Plasma Concentrations | |
| versus Time at Cycle 1 - Dose Escalation Pharmacokinetic Analysis Set | 94 |
| Figure 14.4.1.2.4 Semi-logarithmic Plot and Linear Plot for Mean Free IL-12 Plasma Concentrations | |
| versus Time at Cycle 2 - Dose Escalation Pharmacokinetic Analysis Set | 94 |

Date: 26Feb2025

### **List of Listings**

| Listing 16.2.2.1 Subject Disposition Safety Analysis Set | 96 |
|---|---|
| Listing 16.2.2.2 Safety and Survival Status Follow-Up Safety Analysis Set | 97 |
| Listing 16.2.2.3 Death Safety Analysis Set | 98 |
| Listing 16.2.3 Deviations from the Clinical Protocol Safety Analysis Set | 99 |
| Listing 16.2.4.1 Demographic Data Safety Analysis Set | |
| Listing 16.2.4.2 Baseline Characteristics Safety Analysis Set | . 101 |
| Listing 16.2.5 Study Drug Extent of Exposure and Compliance Safety Analysis Set | . 102 |
| Listing 16.2.6.1 Efficacy Parameters by RECIST 1.1 - Part 1 of 2 Evaluable Efficacy Analysis Set | 103 |
| Listing 16.2.6.2 Efficacy Parameters by iRECIST - Part 2 of 2 Evaluable Efficacy Analysis Set | . 104 |
| Listing 16.2.7.1 Treatment-Emergent Adverse Events Safety Analysis Set | . 105 |
| Listing 16.2.7.2 Serious Adverse Events Safety Analysis Set | . 106 |
| Listing 16.2.7.3 Treatment-Emergent Adverse Events Leading to Drug Withdrawal Safety Analysis Set | . 107 |
| Listing 16.2.7.4 Treatment-Emergent Adverse Events Leading to Drug Modification Safety Analysis S | |
| Listing 16.2.7.5 Treatment-Emergent Adverse Events of Special Interest Safety Analysis Set | |
| Listing 16.2.7.6 Dose Limiting Toxicity Dose Limiting Toxicity Evaluable Analysis Set | |
| Listing 16.2.7.7 Treatment Emergent Adverse Events Leading to Death Safety Analysis Set | |
| Listing 16.2.8.1 Hematology Tests with CTCAE Grade ≥ 3 Safety Analysis Set | |
| Listing 16.2.8.2.1 Serum Chemistry Tests with CTCAE Grade ≥ 3 Safety Analysis Set | |
| Listing 16.2.8.2.2 Liver Function Tests Safety Analysis Set | |
| Listing 16.2.8.3 Coagulation Tests with CTCAE Grade ≥ 3 Safety Analysis Set | |
| Listing 16.2.9 Vital Signs Clinically Notable Increase and/or Decrease Safety Analysis Set | |
| Listing 16.4.2.1 Medical History Safety Analysis Set | |
| Listing 16.4.2.2.1 Solid Tumor Cancer History - Part 1 of 2 Safety Analysis Set | |
| Listing 16.4.2.2.2 Solid Tumor Cancer History - Part 2 of 2 Safety Analysis Set | |
| Listing 16.4.3.1 Prior Systemic Anti-Cancer Therapies Safety Analysis Set | |
| Listing 16.4.3.2 Prior Radiation Therapy Safety Analysis Set | |
| Listing 16.4.3.3 Prior Cancer Surgery Safety Analysis Set | |
| Listing 16.4.4.1 Prior and Concomitant Medications Safety Analysis Set | |
| Listing 16.4.4.2 Prior and Concomitant Procedures Safety Analysis Set | |
| Listing 16.4.5.1.1 WTX-330 Administration - Part 1 of 2 Safety Analysis Set | . 125 |

| Listing 16.4.5.1.2 WTX-330 Administration - Part 2 of 2 Safety Analysis Set | 126 |
|---|---|
| Listing 16.4.5.2.1 Antineoplastic Therapy since Discontinuation of Study Treatment - Medication | |
| Safety Analysis Set | 127 |
| Listing 16.4.5.2.2 Antineoplastic Therapy since Discontinuation of Study Treatment - Radiation | |
| Safety Analysis Set | |
| Listing 16.4.5.2.3 Antineoplastic Therapy since Discontinuation of Study Treatment - Surgery Safe | _ |
| Analysis Set | |
| Listing 16.4.6.1.1 Target Lesion Safety Analysis Set | |
| Listing 16.4.6.1.2 Non-Target Lesion Safety Analysis Set | |
| Listing 16.4.6.1.3.1 New Target Lesion Safety Analysis Set | 132 |
| Listing 16.4.6.1.3.2 New Non-Target Lesion Safety Analysis Set | 133 |
| Listing 16.4.6.2 Disease Response - Solid Tumor Efficacy Evaluable Population | 134 |
| Listing 16.4.6.4 Prostate-specific Antigen (PSA) Safety Analysis Set | 135 |
| Listing 16.4.7 All Adverse Events Safety Analysis Set | 136 |
| Listing 16.4.8.1 Hematology Tests Safety Analysis Set | 137 |
| Listing 16.4.8.2 Serum Chemistry Tests Safety Analysis Set | 138 |
| Listing 16.2.8.3 Coagulation Tests Safety Analysis Set | 139 |
| Listing 16.4.8.4 Urinalysis Tests Safety Analysis Set | 140 |
| Listing 16.4.8.5 Thyroid Stimulating Hormone Safety Analysis Set | 141 |
| Listing 16.4.8.6 Pregnancy Test Safety Analysis Set | 142 |
| Listing 16.4.9.1 12-Lead ECG Safety Analysis Set | 144 |
| Listing 16.4.9.2 Vital Signs Safety Analysis Set | 145 |
| Listing 16.4.9.3 ECOG Performance Status Safety Analysis Set | 146 |
| Listing 16.4.9.4 Physical Examination Safety Analysis Set | 147 |
| Listing 16.4.10.1.1 WTX-330 Plasma Concentrations ( $\mu$ g/ml) Pharmacokinetic Analysis Set | 148 |
| Listing 16.4.10.1.2 Free IL-12 Plasma Concentrations (pg/ml) Pharmacokinetic Analysis Set | 149 |
| Listing 16.4.10.2.1 WTX-330 Pharmacokinetic Parameters Pharmacokinetic Analysis Set | 150 |
| Listing 16.4.10.2.1 Free IL-12 Pharmacokinetic Parameters Pharmacokinetic Analysis Set | 151 |
| Listing 16.4.10.3 Anti-Drug Antibody Anti-Drug Antibody Analysis Set | 152 |

Date: 26Feb2025

**Table Shells** 

Date: 26Feb2025

### 14.1 Study Population and Baseline

Date: 26Feb2025

Table 14.1.1.1 Summary of Analysis Set - Dose Escalation Screened Subjects

| | WTX-330<br>0.016<br>mg/kg<br>(N=x) | WTX-330<br>0.032<br>mg/kg<br>(N=x) | WTX-330<br>0.056<br>mg/kg<br>(N=x) | WTX-330<br>0.084<br>mg/kg<br>(N=x) | WTX-330<br>0.126<br>mg/kg<br>(N=x) | WTX-330<br>0.190<br>mg/kg<br>(N=x) | WTX-330<br>0.290<br>mg/kg<br>(N=x) | WTX-330<br>0.XXX<br>mg/kg<br>(N=x) | Total<br>(N=xx) |
|---|---|---|---|---|---|---|---|---|---|
| Screened subjects | | | | | | | | | XXX |
| Screen failure | | | | | | | | | XX |
| Enrolled subjects, n | X | X | Х | Х | Х | х | Х | Х | XX |
| Safety analysis set, n | X | X | X | X | Х | X | X | X | XX |
| Dose-determining analysis set, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Efficacy evaluable analysis set, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Pharmacokinetics analysis set, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Pharmacodynamics analysis set - Cytokines , n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX (XX.X) |
| Pharmacodynamics analysis set - Peripheral Immune Cells, n(%) | X (XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | XX(XX.X) |
| Anti-drug antibody analysis set, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |

Note: See SAP section 5 for the definition of each analysis set.

Note: N is the number of subjects in Safety Analysis Set. It is the denominator for the percentage.

Date: 26Feb2025

# Table 14.1.1.2.1 Summary of Analysis Set - Dose Expansion Screened Subjects

| | Arm A<br>(N=XX) | Arm B (N=XX) | Total<br>(N=XX) |
|---|---|---|---|
| Screened subjects | XX | XX | XX |
| Screen failure | xx | XX | XX |
| Enrolled subjects, n | xx | xx | XX |
| Safety analysis set, n | XX | XX | XX |
| Efficacy evaluable analysis set, n(%) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Pharmacokinetics analysis set, n(%) | XX(XX.X) | XX(XX.X) | XX(XX.X) |

Note: Arm A = Patients with indications for which a CPI is indicated/approved; Arm B = Patients with tumor types for which CPI therapy is not indicated/approved.

Note: See SAP section 5 for the definition of each analysis set.

Note: N is the number of subjects in Safety Analysis Set. It is the denominator for the percentage.

Date: 26Feb2025

Table 14.1.1.2.2

Summary of Analysis Set - Dose Expansion by Indication Screened Subjects

Arm A

Arm B

X(XX.X)

X(XX.X) X(XX.X)

| Screened subjects xx xx | | RCC (N=XX) | NSCLC<br>(N=XX) | HNSCC<br>(N=XX) | XXXXX<br>(N=XX) | CC<br>(N=X | | DLBCL<br>(N=XX) | YYYYY<br>(N=XX) |
|---|---|---|---|---|---|---|---|---|---|
| Enrolled subjects, n x x x x x x x x x x x x x x x x x x | Screened subjects | XX | XX | XX | XX | XX | XX 2 | XX | XX |
| Safety analysis set, n x x x x x x x x x x x | Screen failure | XX | XX | XX | xx | XX | XX 1 | XX | XX |
| | Enrolled subjects, n | х | x | x | x | х | . х | х | х |
| Efficacy evaluable analysis set, $n(%)$ $X(XX.X)$ $X(XX.X)$ $X(XX.X)$ $X(XX.X)$ $X(XX.X)$ $X(XX.X)$ $X(XX.X)$ | Safety analysis set, n | X | x | x | X | x | X | x | x |
| | Efficacy evaluable analysis set, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX | .X) X(XX.X) | X(XX.X) | X(XX.X) |

Note: Arm A = Patients with indications for which a CPI is indicated/approved; Arm B = Patients with tumor types for which CPI therapy is not indicated/approved.

X(XX.X)

Note: RCC = Renal Cell Carcinoma; NSCLC = Non-small Cell Lung Cancer; HNSCC = Head and Neck Squamous Cell Carcinoma; XXXXXX = \_\_\_; CC = Colorectal Carcinoma; FL = Follicular Lymphoma; DLBCL = Diffuse Large B-cell Lymphoma; YYYYYY = \_\_\_.

X(XX.X)

X(XX.X)

X(XX.X)

Note: See SAP section 5 for the definition of each analysis set.

Anti-drug antibody analysis set, n(%)

Note: N is the number of subjects in Safety Analysis Set. It is the denominator for the percentage.

X(XX.X)

Table 14.1.2.1 Summary of Subject Disposition - Dose Escalation Safety Analysis Set

| | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | |
| | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| Disposition Description | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=XX) |
| Ongoing WTX-330 treatment, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Discontinued WTX-330 treatment, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX (XX.X) |
| Reason for WTX-330 treatment discontinuation, n(%) | | | | | | | | | |
| Adverse event | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Death | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Physician decision | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Pregnancy | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Progressive disease | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Radiological | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Clinical | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Study terminated by sponsor | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Withdrawal of ICF | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX (XX.X) |
| Ongoing study, n(%) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Discontinued study, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Reason for study discontinuation, n(%) | | | | | | | | | |
| Completed study | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Withdrawal of consent by patient | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Lost to follow-up | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Death | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Sponsor terminated the study | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| COVID-19 related | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | XX (XX.X) |

Date: 26Feb2025

Table 14.1.2.2

Summary of Subject Disposition - Dose Expansion
Safety Analysis Set

| | Arm A | Arm B | Total |
|---|---|---|---|
| Disposition Description | (N=XX) | (N=XX) | (N=XX) |
| Ongoing WTX-330 treatment, n(%) | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| Discontinued WTX-330 treatment, n(%) | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| Reason for WTX-330 treatment discontinuation, n(%) | | | |
| Adverse event | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Death | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Physician decision | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Pregnancy | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Progressive disease | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Radiological | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Clinical | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Study terminated by sponsor | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Withdrawal of ICF | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Other | XX(XX.X) | XX (XX.X) | XX(XX.X) |
| Ongoing study, n(%) | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| Discontinued study, n(%) | XX(XX.X) | XX (XX.X) | XX(XX.X) |
| Reason for study discontinuation, n(%) | | | |
| Completed study | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Withdrawal of consent by patient | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Lost to follow-up | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Death | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Sponsor terminated the study | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| COVID-19 related | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Other | XX(XX.X) | XX(XX.X) | XX(XX.X) |

Note: Arm A = Patients with indications for which a CPI is indicated/approved; Arm B = Patients with tumor types for which CPI therapy is not indicated/approved.

Table 14.1.3.1

Summary of Deviations from the Clinical Protocol - Dose Escalation
Safety Analysis Set

| | WTX-330 | | WTX-330 | WTX-330 | WTX-330 | WTX-330 | | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | |
| | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| | (N=x) | (N=x) | (N=x) | (N=x) | (N=X) | (N=x) | (N=x) | (N=x) | (N=XX) |
| Subjects with any deviation, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Deviation category | | | | | | | | | |
| ICF/Subject information | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Ineligible subject enrolled | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| IMP dose error | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| IMP other error | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Prohibited medication | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| <pre><insert "0"="" all="" categories="" edc="" in="" non=""></insert></pre> | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| SAE or AESI reporting failure | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Subjects with any major deviation, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Deviation category | | | | | | | | | |
| ICF/Subject information | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Ineligible subject enrolled | X (XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X(XX.X) | | | | XX(XX.X) |
| IMP dose error | X (XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | | | | XX(XX.X) |
| <pre><insert "0"="" all="" categories="" edc="" in="" non=""></insert></pre> | X (XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | | | | XX(XX.X) |
| SAE or AESI reporting failure | X (XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | XX(XX.X) |
| Other | X (XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Subjects with any minor deviation, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Deviation category | | | | | | | | | |
| ICF/Subject information | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | XX(XX.X) |
| Ineligible subject enrolled | | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | | | | XX(XX.X) |
| IMP dose error | | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | | | | XX(XX.X) |
| <pre><insert "0"="" all="" categories="" edc="" in="" non=""></insert></pre> | | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | | | | XX(XX.X) |
| SAE or AESI reporting failure | | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | | | | XX(XX.X) |
| Other | | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | | | | XX (XX.X) |

Date: 26Feb2025

Table 14.1.3.2

Summary of Deviations from the Clinical Protocol - Dose Expansion

Safety Analysis Set

| | Arm A | Arm B | Total |
|---|---|---|---|
| | (N=XX) | (N=XX) | (N=XX) |
| Subjects with any deviation, n(%) | X (XX.X) | X(XX,X) | XX(XX.X) |
| Deviation category | | | |
| ICF/Subject information | X(XX.X) | X(XX.X) | XX(XX.X) |
| Ineligible subject enrolled | X(XX.X) | X(XX.X) | XX(XX.X) |
| IMP dose error | X(XX.X) | X(XX.X) | XX(XX.X) |
| IMP other error | X(XX.X) | X(XX.X) | XX(XX.X) |
| Prohibited medication | X(XX.X) | X(XX.X) | XX(XX.X) |
| <pre><insert "0"="" all="" categories="" edc="" in="" non=""></insert></pre> | X(XX.X) | X(XX.X) | XX(XX.X) |
| SAE or AESI reporting failure | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X (XX.X) | X(XX.X) | XX(XX.X) |
| Subjects with any major deviation, n(%) | X(XX.X) | X (XX.X) | XX(XX.X) |
| Deviation category | | | |
| ICF/Subject information | X(XX.X) | X (XX.X) | XX(XX.X) |
| Ineligible subject enrolled | X(XX.X) | X (XX.X) | XX(XX.X) |
| IMP dose error | X(XX.X) | X (XX.X) | XX(XX.X) |
| <pre><insert "0"="" all="" categories="" edc="" in="" non=""></insert></pre> | X(XX.X) | X (XX.X) | XX(XX.X) |
| SAE or AESI reporting failure | X(XX.X) | X (XX.X) | XX(XX.X) |
| Other | X (XX.X) | X(XX.X) | XX(XX.X) |
| Subjects with any minor deviation, n(%) | X (XX.X) | X (XX.X) | XX(XX.X) |
| Deviation category | | | |
| ICF/Subject information | X(XX.X) | X(XX.X) | XX(XX.X) |
| Ineligible subject enrolled | X(XX.X) | X(XX.X) | XX(XX.X) |
| IMP dose error | X(XX.X) | X(XX.X) | XX(XX.X) |
| <pre><insert "0"="" all="" categories="" edc="" in="" non=""></insert></pre> | X(XX.X) | X(XX.X) | XX(XX.X) |
| SAE or AESI reporting failure | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | XX(XX.X) |

Note: Arm A = Patients with indications for which a CPI is indicated/approved; Arm B = Patients with tumor types for which CPI therapy is not indicated/approved.

Table 14.1.4.1

Summary of Demographic Characteristics - Dose Escalation

Safety Analysis Set

| | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | |
| | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=X) | (N=X) | (N=X) | (N=xX) |
| Age (years) | | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Age group, n(%) | | | | | | | | | |
| <45 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| ≥45 - <65 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| ≥65 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Sex, n(%) | | | | | | | | | |
| Male | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Female | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| With childbearing potential | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Without childbearing potential | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Ethnicity, n(%) | | | | | | | | | |
| Hispanic or Latino | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Not Hispanic or Latino | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Not Reported | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Race [1], n(%) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | XX(XX.X) |
| American Indian or Alaskan Native | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Asian | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Black or African American | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | | XX(XX.X) |
| Native Hawaiian or Other Pacific | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Islander | | | | | | | | | |
| White | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Not Reported | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |

Protocol: WTX-330x2101

| Weight (kg) at baseline | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |
| Height (cm) at baseline | | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |
| ECOG performance status at baseline, n(%) | | | | | | | | | |
| 0 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| 1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |

<sup>[1]</sup> Subjects might report multiple races.

Table 14.1.4.2

Summary of Demographic Characteristics - Dose Expansion
Safety Analysis Set

| | Arm A | Arm B | Total |
|---|---|---|---|
| | (N=XX) | (N=XX) | (N=XX) |
| Age (years) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |
| ge group, n(%) | | | |
| <45 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| ≥45 - <65 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| ≥65 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Sex, n(%) | | | |
| Male | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Female | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| With childbearing potential | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Without childbearing potential | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| thnicity, n(%) | | | |
| Hispanic or Latino | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Not Hispanic or Latino | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Not Reported | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| ace [1], n(%) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| American Indian or Alaskan Native | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| Asian | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| Black or African American | XX(XX.X) | XX (XX.X) | XX(XX.X) |
| Native Hawaiian or Other Pacific Islander | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| White | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Reported | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Protocol: WTX-330x2101

Date: 26Feb2025

| Weight (kg) at baseline | | | |
|-------------------------------------------|-----------|----------|----------|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |
| Height (cm) at baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | xx.xx |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |
| ECOG performance status at baseline, n(%) | | | |
| 0 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| 1 | XX (XX.X) | XX(XX.X) | XX(XX.X) |

Note: Arm A = Patients with indications for which a CPI is indicated/approved; Arm B = Patients with tumor types for which CPI therapy is not indicated/approved.
[1] Subjects might report multiple races.

Table 14.1.5.1.1

Summary of Solid Tumor Disease Characteristics - Dose Escalation
Safety Analysis Set

| | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | |
| | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| | (N=x) | (N=x) | (N=X) | (N=x) | (N=x) | (N=X) | (N=x) | (N=X) | (N=xX) |
| Time since date of initial histopathological | | | | | | | | | |
| diagnosis (months) | | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX |
| <12 months, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| >=12 months - < 24 months, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| >=24 months - < 36 months, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| >=36 months, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Time since date of most recent disease recurrence/progression (months) | | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Cancer type, n(%) | | | | | | | | | |
| Adrenal cancer | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Basal cell skin cancer | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Bile duct cancer | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Bladder cancer | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Bone cancer | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Breast cancer | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | XX(XX.X) |
| <pre><insert cancer="" edc="" type=""></insert></pre> | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Primary site of solid tumor, n(%) | | | | | | | | | |
| Bone | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Breast | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | | XX (XX.X) |
| Bronchus | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | | XX (XX.X) |
| Cervix | X (XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | | XX (XX.X) |
| Colon | X (XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | | XX (XX.X) |
| Duodenum | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | | XX (XX.X) |

| <pre><insert "0"="" edc="" non="" records=""></insert></pre> | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| Any pathologic sub-type, n(%) | | | | | | | | | |
| Yes | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| No | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Stage of solid tumor at initial diagnosis, n | 1 (%) | | | | | | | | |
| 0 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| I | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| II | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| III | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| IV | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Stage of solid tumor at baseline, n(%) | | | | | | | | | |
| 0 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| I | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| II | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| III | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| IV | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX (XX.X) |
| Characterization of disease at study entry, | n (%) | | | | | | | | |
| Locally advanced | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Metastatic | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Metastatic site if metastatic | | | | | | | | | |
| Abdomen/Abdominal Wall | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Adrenal Glands | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| <pre><insert "0"="" edc="" non="" records=""></insert></pre> | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX (XX.X) |
| Any known genetic mutations, n(%) | | | | | | | | | |
| No | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Yes | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| BRAF | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| EGFR | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| HER2 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| KRAS | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| KIT | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| BRAF | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| EGFR | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| <pre><insert "0"="" edc="" non="" records=""></insert></pre> | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| MSI status, n(%) | | | | | | | | | |
| Not applicable | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Unknown | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Known | X (XX X) | X(XX X) | X (XX X) | X(XX X) | X(XX X) | X(XX X) | X(XX X) | X (XX X) | XX (XX X) |

Date: 26Feb2025

| MSI-H (microsatellite instability-high) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
|---|---|---|---|---|---|---|---|---|---|
| MSI-L (microsatellite instability-low) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| MSS (microsatellite stable) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| dMMR (mismatch repair deficient) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| pMMR (mismatch repair proficient) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| TMB status known?, n(%) | | | | | | | | | |
| Not Applicable | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| No | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Yes | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| High | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Intermediate | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Tumoral genetic characterization, n(%) | | | | | | | | | |
| Yes | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| No | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Not Applicable | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |

Note: Time since date of initial histopathological diagnosis (months) = (date of first dose - date of initial histopathological diagnosis)/30.4375. Time since date of most recent disease recurrence/progression (months) = (date of first dose - date of most recent disease recurrence/progression)/30.4375.
Table 14.1.5.1.2

Summary of Solid Tumor Disease Characteristics - Dose Expansion
Safety Analysis Set

| | Arm A | Arm B | Total |
|---|---|---|---|
| | (N=XX) | (N=XX) | (N=XX) |
| Time since date of initial histopathological diagnosis (months) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |
| <12 months, n(%) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| >=12 months - < 24 months, n(%) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| >=24 months - < 36 months, n(%) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| >=36 months, n(%) | XX(XX.X) | XX (XX.X) | XX(XX.X) |
| Time since date of most recent disease recurrence/progression (months) | | | |
| n | XX | XX | XX |
| Mean | xx.x | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX |
| Cancer type, n(%) | | | |
| Adrenal cancer | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Basal cell skin cancer | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Bile duct cancer | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Bladder cancer | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Bone cancer | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Breast cancer | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| <pre><insert "0"="" edc="" non="" records=""></insert></pre> | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Primary site of solid tumor, n(%) | | | |
| Bone | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Breast | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Bronchus | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Cervix | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Colon | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Duodenum | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <pre><insert "0"="" edc="" non="" records=""></insert></pre> | XX (XX.X) | XX (XX.X) | XX (XX.X) |

| Any pathologic sub-type, n(%) | | | |
|---|---|---|---|
| Yes | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| No | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Stage of solid tumor at initial diagnosis, n(%) | | | |
| 0 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| I | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| II | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| III | XX(XX.X) | XX (XX.X) | XX(XX.X) |
| IV | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| Stage of solid tumor at baseline, n(%) | | | |
| 0 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| I | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| II | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| III | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| IV | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| Characterization of disease at study entry, n(%) | | | |
| Locally advanced | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| Metastatic | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| Metastatic site if metastatic | | | |
| Abdomen/Abdominal Wall | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| Adrenal Glands | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| <pre><insert "0"="" edc="" non="" records=""></insert></pre> | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Any known genetic mutations, n(%) | | | |
| No | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Yes | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| BRAF | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| EGFR | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| HER2 | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| KRAS | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| KIT | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| BRAF | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| EGFR | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| <pre><insert "0"="" edc="" non="" records=""></insert></pre> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| MSI status, n(%) | | | |
| Not applicable | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Unknown | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Known | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| MSI-H (microsatellite instability-high) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| MSI-L (microsatellite instability-low) | XX(XX.X) | XX(XX.X) | XX(XX.X) |

Date: 26Feb2025

| MSS (microsatellite stable) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
|----------------------------------------|-----------|----------|----------|
| dMMR (mismatch repair deficient) | XX(XX,X) | XX(XX.X) | XX(XX.X) |
| pMMR (mismatch repair proficient) | XX(XX,X) | XX(XX.X) | XX(XX.X) |
| Other | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| TMB status known?, n(%) | | | |
| Not Applicable | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| No | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Yes | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| High | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Intermediate | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Other | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| Tumoral genetic characterization, n(%) | | | |
| Yes | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| No | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Not Applicable | XX(XX.X) | XX(XX.X) | XX(XX.X) |

Note: Arm A = Patients with indications for which a CPI is indicated/approved; Arm B = Patients with tumor types for which CPI

therapy is not indicated/approved.

Note: Time since date of initial histopathological diagnosis (months) = (date of first dose - date of initial histopathological diagnosis)/30.4375. Time since date of most recent disease recurrence/progression (months) = (date of first dose - date of most recent disease recurrence/progression)/30.4375.

Date: 26Feb2025

Table 14.1.8.2.1

Summary of Concomitant Medications by WHO Drug ATC Category II and Preferred Term - Dose Escalation Safety Analysis Set

| | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | |
| ATC Category II | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| Preferred Term | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=XX) |
| Subjects with concomitant medications, n(%) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| ATC category II #1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred name #1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred name #2 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| <insert></insert> | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| ATC category II #2 | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | XX(XX.X) |
| Preferred name #1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred name #2 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| <insert></insert> | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |

# <insert>

Note: Prior Medications are coded with WHODRUG Global B3 March 2023.

Note: Concomitant medication is the medication that is used on/after the first dose of WTX-330.

Date: 26Feb2025

Table 14.1.8.2.2

Summary of Concomitant Medications by WHO Drug ATC Category II and Preferred Term - Dose Expansion
Safety Analysis Set

| ATC Category II | Arm A | Arm B | Total |
|---|---|---|---|
| Preferred Term | (N=XX) | (N=XX) | (N=XX) |
| Subjects with concomitant medications, n(%) | X (XX.X) | X (XX.X) | XX (XX.X) |
| ATC category II #1 | X (XX.X) | X (XX.X) | XX(XX.X) |
| Preferred name #1 | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred name #2 | X(XX.X) | X(XX.X) | XX(XX.X) |
| <insert></insert> | X (XX.X) | X(XX.X) | XX(XX.X) |
| ATC category II #2 | X (XX.X) | X (XX.X) | XX(XX.X) |
| Preferred name #1 | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred name #2 | X(XX.X) | X(XX.X) | XX(XX.X) |
| <insert></insert> | X(XX.X) | X(XX.X) | XX(XX.X) |

#### <insert>

Note: Arm A = Patients with indications for which a CPI is indicated/approved; Arm B = Patients with tumor types for which CPI therapy is not indicated/approved.

Note: Prior Medications are coded with WHODRUG Global B3 March 2023.

Note: Concomitant medication is the medication that is used on/after the first dose of WTX-330.

Table 14.1.9.1

Summary of WTX-330 Exposure, Compliance and Dose Modification - Dose Escalation Safety Analysis Set

| N=x (N=x) | | | | | | | | | | _ |
|---|---|---|---|---|---|---|---|---|---|---|
| mg/kg mg/k | | | | | | | | | | |
| N=x (N=x) | | | | | | | | | | |
| Duration of exposure [a], weeks n | | | , , | | | | | | | Total |
| Median | | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=xX) |
| Mean Standard Deviation XX.X XX | Duration of exposure [a], weeks | | | | | | | | | |
| Standard Deviation | n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Median Min, Max XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX. | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | Standard Deviation | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Duration of exposure categories, n(%) <pre></pre> | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| <pre></pre> | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| >=4 weeks - < 12 weeks X(XX.X) X(XX.X)< | Duration of exposure categories, n(%) | | | | | | | | | |
| >=12 weeks X(XX.X) X( | <4 weeks | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Number of treatment cycle started n | >=4 weeks - < 12 weeks | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| n xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx </td <td>&gt;=12 weeks</td> <td>X(XX.X)</td> <td>X(XX.X)</td> <td>X(XX.X)</td> <td>X(XX.X)</td> <td>X(XX.X)</td> <td>X(XX.X)</td> <td>X(XX.X)</td> <td>X(XX.X)</td> <td>XX(XX.X)</td> | >=12 weeks | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Mean xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x <th< td=""><td>Number of treatment cycle started</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></th<> | Number of treatment cycle started | | | | | | | | | |
| Standard Deviation xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx <td>n</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> | n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Median Min, Max XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX. | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X |
| Min, Max xx, xx xx, xx xx, xx xx, xx xx, xx xx, xx xx, xx xx, xx xx, xx xx, xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx <th< td=""><td>Standard Deviation</td><td>XX.XX</td><td>xx.xx</td><td>XX.XX</td><td>XX.XX</td><td>XX.XX</td><td>XX.XX</td><td>XX.XX</td><td>XX.XX</td><td>xx.xx</td></th<> | Standard Deviation | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx |
| Cumulative dose [b], mg/kg n | Median | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X |
| n xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx </td <td>Min, Max</td> <td>xx, xx</td> <td>XX, XX</td> <td>XX, XX</td> <td>XX, XX</td> <td>XX, XX</td> <td>XX, XX</td> <td>xx, xx</td> <td>xx, xx</td> <td>XX, XX</td> | Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx | XX, XX |
| Mean xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x <th< td=""><td>Cumulative dose [b], mg/kg</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></th<> | Cumulative dose [b], mg/kg | | | | | | | | | |
| Standard Deviation xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx <td>n</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> | n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Median Min, Max xx.x | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X |
| Min, Max | Standard Deviation | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx |
| Average dose intensity [c], (mg/kg)/cycle n | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| n xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx </td <td>Min, Max</td> <td>XX, XX</td> <td>XX, XX</td> <td>XX, XX</td> <td>XX, XX</td> <td>XX, XX</td> <td>XX, XX</td> <td>xx, xx</td> <td>xx, xx</td> <td>XX, XX</td> | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx | XX, XX |
| Mean xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x <th< td=""><td>Average dose intensity [c], (mg/kg)/cycle</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></th<> | Average dose intensity [c], (mg/kg)/cycle | | | | | | | | | |
| Standard Deviation xx.xx | n | XX | XX | XX | xx | xx | XX | XX | XX | XX |
| Median xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx | Mean | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx | Standard Deviation | XX.XX | XX.XX | xx.xx | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx |
| Min, Max xx, xx xx, xx xx, xx xx, xx xx, xx xx, xx xx | Median | xx.x | xx.x | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X | xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

| Treatment compliance [d], % | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| Treatment compliance categories, n(%) | | | | | | | | | |
| <80% | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| >=80% -<120% | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| >=120% | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | XX(XX.X) |
| Subjects with infusion interrupted, n(%) | | | | | | | | | |
| 0 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | | | | | XX(XX.X) |
| 1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | | | | | XX(XX.X) |
| 2 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| >=3 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | XX(XX.X) |
| Reason for infusion interruption [e] n(%) | | | | | | | | | |
| Infusion reaction | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Adverse event other than infusion reaction | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Subjects with Dose Adjusted [e], n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | XX(XX.X) |
| Dose missed | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Dose reduced | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Dose discontinued | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | | | | | XX(XX.X) |
| Dose interrupted | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | XX(XX.X) |
| Reason for dose missed [e] n(%) | | | | | | | | | |
| Adverse event | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| PI/Sponsor decision | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | XX(XX.X) |
| Reason for dose reduced [e] n(%) | | | | | | | | | |
| Adverse event | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| PI/Sponsor decision | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Reason for dose discontinued [e] n(%) | | | | | | | | | |
| Adverse event | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| PI/Sponsor decision | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |

| Reason for dose interrupted [e] n(%) | | | | | | | |
|---|---|---|---|---|---|---|---|
| Adverse event | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) X(XX.X) XX(XX.X) |
| PI/Sponsor decision | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) X(XX.X) XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) X(XX.X) XX(XX.X) |

<sup>[</sup>a] Duration of exposure = (the date of last WTX-330 does - the date of first WTX-330 dose + 14)/7.

<sup>[</sup>b] Cumulative Dose of WTX-330 (mg/kg) = sum of the individual Total Dose Administered being reported in CRFs.

<sup>[</sup>c] Average Dose Intensity ((mg/kg)/cycle) is calculated by Cumulative Dose /Number of treatment cycles started.

<sup>[</sup>d] Treatment compliance (%) = 100\*(Cumulative Dose/Total Planned Dose).

<sup>[</sup>e] Categories are not mutually exclusive.

Table 14.1.9.2

Summary of WTX-330 Exposure, Compliance and Dose Modification - Dose Expansion Safety Analysis Set

| | Arm A | Arm B | Total |
|------------------------------------------|----------|---------|----------|
| | (N=XX) | (N=XX) | (N=XX) |
| Duration of exposure [a], weeks | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |
| Ouration of exposure categories, n(%) | | | |
| <4 weeks | X(XX.X) | X(XX.X) | XX(XX.X) |
| >=4 weeks - < 12 weeks | X(XX.X) | X(XX.X) | XX(XX.X) |
| >=12 weeks | X (XX.X) | X(XX.X) | XX(XX.X) |
| Number of treatment cycle started | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |
| Cumulative dose [b], mg/kg | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Average dose intensity [c],(mg/kg)/cycle | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |

| reatment compliance [d], % | | | |
|--------------------------------------------|----------|----------|-----------|
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |
| reatment compliance categories, n(%) | | | |
| <80% | X (XX.X) | X(XX.X) | XX(XX.X) |
| >=80% -<120% | X(XX.X) | X(XX.X) | XX(XX.X) |
| >=120% | X (XX.X) | X(XX.X) | XX(XX.X) |
| ubjects with infusion interrupted, n(%) | | | |
| 0 | X (XX.X) | X(XX.X) | XX(XX.X) |
| 1 | X (XX.X) | X(XX.X) | XX(XX.X) |
| 2 | X (XX.X) | X(XX.X) | XX(XX.X) |
| >=3 | X (XX.X) | X(XX.X) | XX(XX.X) |
| eason for infusion interruption [e] n(%) | | | |
| Infusion reaction | X(XX.X) | X(XX.X) | XX(XX.X) |
| Adverse event other than infusion reaction | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X (XX.X) | X(XX.X) | XX(XX.X) |
| ubjects with Dose Adjusted [e], n(%) | X (XX.X) | X(XX.X) | XX(XX.X) |
| Dose missed | X(XX.X) | X(XX.X) | XX(XX.X) |
| Dose reduced | X(XX.X) | X(XX.X) | XX(XX.X) |
| Dose discontinued | X(XX.X) | X(XX.X) | XX(XX.X) |
| Dose interrupted | X (XX.X) | X(XX.X) | XX(XX.X) |
| eason for dose missed [e] n(%) | | | |
| Adverse event | X(XX.X) | X(XX.X) | XX(XX.X) |
| PI/Sponsor decision | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X (XX.X) | X(XX.X) | XX(XX.X) |
| eason for dose reduced [e] n(%) | | | |
| Adverse event | X (XX.X) | X(XX.X) | XX(XX.X) |
| PI/Sponsor decision | X (XX.X) | X (XX.X) | XX(XX.X) |
| Other | X (XX.X) | X(XX.X) | XX(XX.X) |
| eason for dose discontinued [e] n(%) | | | |
| Adverse event | X (XX.X) | X(XX.X) | XX(XX.X) |
| PI/Sponsor decision | X (XX.X) | X (XX.X) | XX (XX.X) |
| ri/spolisor decision | | | |

Date: 26Feb2025

| Reason for dose interrupted [e] n(%) | | | |
|--------------------------------------|---------|---------|----------|
| Adverse event | X(XX.X) | X(XX.X) | XX(XX.X) |
| PI/Sponsor decision | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | XX(XX.X) |

Note: Arm A = Patients with indications for which a CPI is indicated/approved; Arm B = Patients with tumor types for which CPI therapy is not indicated/approved.

- [a] Duration of exposure = (the date of last WTX-330 does the date of first WTX-330 dose + 14)/7.
- [b] Cumulative Dose of WTX-330 (mg/kg) = sum of the individual Total Dose Administered being reported in CRFs.
- [c] Average Dose Intensity ((mg/kg)/cycle) is calculated by Cumulative Dose /Number of treatment cycles started.
- [d] Treatment compliance (%) = 100\*(Cumulative Dose/Total Planned Dose).
- [e] Categories are not mutually exclusive.

Date: 26Feb2025

# 14.2 Analyses of Efficacy

Date: 26Feb2025

Table 14.2.1.1

Summary of Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Dose Escalation

Efficacy Evaluable Analysis Set

| | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | |
| | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=xX) |
| RECIST 1.1 | | | | | | | | | |
| BOR, n(%) | | / | 4 | / | | / | 4 | | |
| Complete Response (CR) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Partial Response (PR) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Stable Disease (SD) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Progressive Disease (PD) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Not Evaluable | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| ORR n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| CBR at 3 month, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| CBR at 6 month, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| CBR at 9 month, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| irecist | | | | | | | | | |
| iBOR, n(%) | | | | | | | | | |
| iCR | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| iPR | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| iSD | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| iUPD | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| iCPD | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Not Evaluable | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| iORR, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| 95% CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| iCBR at 3 month, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| 95% CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| iCBR at 6 month, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| iCBR at 9 month, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |

Note: Best overall response (BOR) of CR and PR per RECIST 1.1 needs to be confirmed in a subsequent assessment (≥ 4 weeks). Immune Best overall response (iBOR) per iRECIST 1.1 is the best response among all visits according to the following sequence: Immune Complete Response (iCR), Immune Partial Response (iPR), Immune Stable Disease (iSD), Immune Confirmed Progressive Disease (iCPD), Immune Unconfirmed Progressive Disease (iUPD), Not Evaluable.

Date: 26Feb2025

Note: Overall response rate (ORR or iORR) is defined as the proportion of patients achieving CR and/or PR in RECIST 1.1 or iCR and/or iPR in iRECIST.

Note: Clinical Benefit Rate (CBR or iCBR) is defined as the proportion of subjects achieving clinical benefit, which is defined as the time from the date of last CR/PR/SD per RECIST or iCR/iPR/iSD per iRECIST to the date of first dose is at least 3, 6, or 9 months.

Date: 26Feb2025

Table 14.2.1.2.1

Summary of Best Overall Response, Objective Response Rate, and Clinical Benefit Rate - Dose Expansion

Efficacy Evaluable Analysis Set

| | Arm A | Arm B [1] | Total |
|--------------------------|-----------|-----------|-----------|
| | (N=XX) | (N=XX) | (N=XX) |
| ECIST 1.1 | | | |
| BOR, n(%) | | | |
| Complete Response (CR) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Partial Response (PR) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Stable Disease (SD) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Progressive Disease (PD) | X (XX.X) | X(XX.X) | XX(XX.X) |
| Not Evaluable | X(XX.X) | X (XX.X) | XX(XX.X) |
| ORR n(%) | X(XX.X) | X(XX.X) | XX(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| CBR at 3 month, n(%) | X(XX.X) | X (XX.X) | XX(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| CBR at 6 month, n(%) | X(XX.X) | X(XX.X) | XX(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| CBR at 9 month, n(%) | X(XX.X) | X(XX.X) | XX(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| RECIST | | | |
| iBOR, n(%) | | | |
| iCR | X(XX.X) | X(XX.X) | XX(XX.X) |
| iPR | X (XX.X) | X (XX.X) | XX(XX.X) |
| iSD | X(XX.X) | X (XX.X) | XX(XX.X) |
| iUPD | X(XX.X) | X (XX.X) | XX(XX.X) |
| iCPD | X(XX.X) | X(XX.X) | XX(XX.X) |
| Not Evaluable | X(XX.X) | X(XX.X) | XX(XX.X) |
| iORR, n(%) | X(XX.X) | X(XX.X) | XX(XX.X) |
| 95% CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| iCBR at 3 month, n(%) | X (XX.X) | X(XX.X) | XX(XX.X) |
| 95% CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| iCBR at 6 month, n(%) | X(XX.X) | X(XX.X) | XX(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| iCBR at 9 month, n(%) | X (XX.X) | X(XX.X) | XX(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |

Note: Arm A = Patients with indications for which a CPI is indicated/approved; Arm B = Patients with tumor types for which CPI therapy is not indicated/approved.

Note: Best overall response (BOR) of CR and PR per RECIST 1.1 needs to be confirmed in a subsequent assessment ( $\geq$  4 weeks). Immune Best overall response (iBOR) per iRECIST 1.1 is the best response among all visits according to the following sequence: Immune

Date: 26Feb2025

Complete Response (iCR), Immune Partial Response (iPR), Immune Stable Disease (iSD), Immune Confirmed Progressive Disease (iCPD), Immune Unconfirmed Progressive Disease (iUPD), Not Evaluable.

Note: Overall response rate (ORR or iORR) is defined as the proportion of patients achieving CR and/or PR in RECIST 1.1 or iCR and/or iPR in iRECIST.

Note: Clinical Benefit Rate (CBR or iCBR) is defined as the proportion of subjects achieving clinical benefit, which is defined as the time from the date of last CR/PR/SD per RECIST or iCR/iPR/iSD per iRECIST to the date of first dose is at least 3, 6, or 9 months.

[1] Include solid tumor only.

Date: 26Feb2025

Table 14.2.1.2.2

Summary of Best Overall Response, Objective Response Rate, and Clinical Benefit Rate
- Dose Expansion by Type of Disease (Solid Tumor)

Efficacy Evaluable Analysis Set

| | | Arm | A | | Arm | В |
|---|---|---|---|---|---|---|
| | RCC (N=x) | NSCLC (N=x) | HNSCC (N=x) | XXXXX (N=x) | CC (N=x) | YYYYY (N=x) |
| RECIST 1.1 | | | | | <u> </u> | |
| BOR, n(%) | | | | | | |
| Complete Response (CR) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) |
| Partial Response (PR) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| Stable Disease (SD) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) |
| Progressive Disease (PD) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) |
| Not Evaluable | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| ORR n(%) | X(XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | X(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | xx.x,xx.x |
| CBR at 3 month, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| CBR at 6 month, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | xx.x,xx.x | XX.X,XX.X |
| CBR at 9 month, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| irecist | | | | | | |
| iBOR, n(%) | | | | | | |
| iCR | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) |
| iPR | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) |
| iSD | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) |
| iUPD | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) |
| iCPD | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) |
| Not Evaluable | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) |
| iORR, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) |
| 95% CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | xx.x,xx.x | xx.x,xx.x | XX.X,XX.X |
| iCBR at 3 month, n(%) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | X(XX.X) |
| 95% CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| iCBR at 6 month, n(%) | X (XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | X (XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |
| iCBR at 9 month, n(%) | X (XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | X (XX.X) |
| 95% exact CI, % | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X |

Note: Arm A = Patients with indications for which a CPI is indicated/approved; Arm B = Patients with tumor types for which CPI therapy is not indicated/approved; RCC = Renal Cell Carcinoma; NSCLC = Non-small Cell Lung Cancer; HNSCC = Head and Neck Squamous Cell Carcinoma; XXXXXX = \_\_\_; CC = Colorectal Carcinoma; YYYYYY = \_\_\_.

Date: 26Feb2025

Note: Best overall response (BOR) of CR and PR per RECIST 1.1 needs to be confirmed in a subsequent assessment ( $\geq$  4 weeks). Immune Best overall response (iBOR) per iRECIST 1.1 is the best response among all visits according to the following sequence: Immune Complete Response (iCR), Immune Partial Response (iPR), Immune Stable Disease (iSD), Immune Confirmed Progressive Disease (iCPD), Immune Unconfirmed Progressive Disease (iUPD), Not Evaluable.

Note: Overall response rate (ORR or iORR) is defined as the proportion of patients achieving CR and/or PR in RECIST 1.1 or iCR and/or iPR in iRECIST.

Note: Clinical Benefit Rate (CBR or iCBR) is defined as the proportion of subjects achieving clinical benefit, which is defined as the time from the date of last CR/PR/SD per RECIST or iCR/iPR/iSD per iRECIST to the date of first dose is at least 3, 6, or 9 months.

Date: 26Feb2025

# 14.3 Summaries and Analyses of Safety

Date: 26Feb2025

Table 14.3.1.1.1

Overall Summary of Treatment-Emergent Adverse Events - Dose Escalation
Safety Analysis Set

| | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | |
| | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| Subjects Who Had Any, n(%) | (N=x) | (N=x) | (N=X) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=xX) |
| TEAEs | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| TEAEs Related to WTX-330 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Grade 3 or Higher TEAEs | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Grade 3 or Higher TEAEs Related to WTX-330 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Serious TEAEs | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Serious TEAEs Related to WTX-330 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX (XX.X) |
| TEAEs Leading to WTX-330 Withdrawal | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| WTX-330-Related TEAEs Leading to WTX-330 Withdrawal | X (XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | XX (XX.X) |
| TEAEs Leading to WTX-330 Modification | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Dose Delayed | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Dose Interrupted | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Dose Reduced | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Infusion Rate Reduced | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| WTX-330-Related TEAEs Leading to WTX-330 Modification | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | XX(XX.X) |
| TEAEs of Special Interest | X (XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | XX(XX.X) |
| Immune Related TEAEs | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Infusion Related Reaction | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Cytokine Release Syndrome | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| DLT | X (XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | XX(XX.X) |
| TEAE Leading to Death | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |

Note: A TEAE is defined as an AEs that emerges or worsens (ie increase in CTCAE grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

Note: Adverse Events are graded with CTCAE Grade 5.0, except for Cytokine Release Syndrome which is graded with ASTCT Grade.

Note: Each subject is counted only once in each category. TEAEs related to study drug are events reported with 'Definitely Related', 'Probably', 'Possibly' or missing in the relationship.

Date: 26Feb2025

Table 14.3.1.1.2

Overall Summary of Treatment-Emergent Adverse Events - Dose Expansion Safety Analysis Set

| | Arm A | Arm B | Total |
|---|---|---|---|
| Subjects Who Had Any, n(%) | (N=XX) | (N=XX) | (N=XX) |
| TEAES | X (XX.X) | X(XX.X) | XX(XX.X) |
| TEAEs Related to WTX-330 | X (XX.X) | X(XX.X) | XX(XX.X) |
| Grade 3 or Higher TEAEs | X (XX.X) | X(XX.X) | XX(XX.X) |
| Grade 3 or Higher TEAEs Related to WTX-330 | X(XX.X) | X(XX.X) | XX(XX.X) |
| Serious TEAEs | X (XX.X) | X (XX.X) | XX(XX.X) |
| Serious TEAEs Related to WTX-330 | X(XX.X) | X(XX.X) | XX(XX.X) |
| TEAEs Leading to WTX-330 Withdrawal | X (XX.X) | X (XX.X) | XX(XX.X) |
| WTX-330-Related TEAEs Leading to WTX-330 Withdrawal | X (XX.X) | X(XX.X) | XX(XX.X) |
| TEAEs Leading to WTX-330 Modification | X(XX.X) | X(XX.X) | XX(XX.X) |
| Dose Delayed | X (XX.X) | X(XX.X) | XX(XX.X) |
| Dose Interrupted | X(XX.X) | X(XX.X) | XX(XX.X) |
| Dose Reduced | X (XX.X) | X(XX.X) | XX(XX.X) |
| Infusion Rate Reduced | X (XX.X) | X(XX.X) | XX(XX.X) |
| WTX-330-Related TEAEs Leading to WTX-330 Modification | X (XX.X) | X(XX.X) | XX(XX.X) |
| TEAEs of Special Interest | X (XX.X) | X (XX.X) | XX(XX.X) |
| Immune Related TEAEs | X(XX.X) | X(XX.X) | XX(XX.X) |
| Infusion Related Reaction | X (XX.X) | X(XX.X) | XX(XX.X) |
| Cytokine Release Syndrome | X(XX.X) | X(XX.X) | XX(XX.X) |
| TEAE Leading to Death | X (XX.X) | X(XX.X) | XX(XX.X) |

Note: Arm A = Patients with indications for which a CPI is indicated/approved; Arm B = Patients with tumor types for which CPI therapy is not indicated/approved.

Note: A TEAE is defined as an AEs that emerges or worsens (ie increase in CTCAE grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

Note: Adverse Events are graded with CTCAE Grade 5.0, except for Cytokine Release Syndrome which is graded with ASTCT Grade.

Note: Each subject is counted only once in each category. TEAEs related to study drug are events reported with 'Definitely Related', 'Probably', 'Possibly' or missing in the relationship.

Date: 26Feb2025

Table 14.3.2.1.1

Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set

| | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | |
| System Organ Class/ | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| Preferred Term | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=XX) |
| Patients with Any Event, n(%) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | XX (XX.X) |
| System Organ Class #1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | XX(XX.X) |
| Preferred Term #1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred Term #2 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| <insert></insert> | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| System Organ Class #2 | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | XX(XX.X) |
| Preferred Term #1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred Term #2 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| <insert></insert> | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |

<insert>

Note: Adverse Events are coded with MedDRA version 26.0.

Note: A TEAE is defined as an AEs that emerges or worsens (i.e. increase in CTCAE grade/ASTCT Grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

Note: Each subject is counted only once in each category. Table is sorted by System Organ Class count in total, and Preferred Term count in total within each System Organ Class.

# Programming Note:

Sort by SOC count in total, and PT count in total within each SOC

Date: 26Feb2025

Repeat table 14.3.2.1.1 for the following tables, except for the column header and footnote for Dose Expansion.

#### Table 14.3.2.1.2

Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set

## Table 14.3.2.2.1

Summary of WTX-330-related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set

Programming Note: Add "Note: TEAEs related to study drug are events reported with 'Definitely Related', 'Probably', 'Possibly' or missing in the relationship."

## Table 14.3.2.2.2

Summary of WTX-330-related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set

Programming Note: Add "Note: TEAEs related to study drug are events reported with 'Definitely Related', 'Probably', 'Possibly' or missing in the relationship."

#### Table 14.3.2.3.1

Summary of Treatment-Emergent Adverse Events with Grade 3 or Higher by System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set

## Table 14.3.2.3.2

Summary of Treatment-Emergent Adverse Events with Grade 3 or Higher by System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set

#### Table 14.3.2.4.1

Summary of WTX-330-related Treatment-Emergent Adverse Events with Grade 3 or Higher by System Organ Class and Preferred Term - Dose Escalation
Safety Analysis Set

Programming Note: Add "Note: TEAEs related to study drug are events reported with 'Definitely Related', 'Probably', 'Possibly' or missing in the relationship."


Date: 26Feb2025

#### Table 14.3.2.4.2

Summary of WTX-330-related Treatment-Emergent Adverse Events with Grade 3 or Higher by System Organ Class and Preferred Term - Dose Expansion

Safety Analysis Set

Programming Note: Add "Note: TEAEs related to study drug are events reported with 'Definitely Related', 'Probably', 'Possibly' or missing in the relationship."

#### Table 14.3.2.5.1

Summary of Treatment-Emergent Adverse Events Leading to WTX-330 Withdrawal by System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set

#### Table 14.3.2.5.2

Summary of Treatment-Emergent Adverse Events Leading to WTX-330 Withdrawal by System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set

#### Table 14.3.2.6.1

Summary of WTX-330-related Treatment-Emergent Adverse Events Leading to WTX-330 Withdrawal by System Organ Class and Preferred Term - Dose Escalation
Safety Analysis Set

Programming Note: Add "Note: TEAEs related to study drug are events reported with 'Definitely Related', 'Probably', 'Possibly' or missing in the relationship."

## Table 14.3.2.6.2

Summary of WTX-330-related Treatment-Emergent Adverse Events Leading to WTX-330 Withdrawal by System Organ Class and Preferred Term - Dose Expansion
Safety Analysis Set

Date: 26Feb2025

#### Table 14.3.2.7.1

Summary of Treatment-Emergent Adverse Events Leading to WTX-330 Modification by System Organ Class and Preferred Term - Dose Escalation
Safety Analysis Set

#### Table 14.3.2.7.2

Summary of Treatment-Emergent Adverse Events Leading to WTX-330 Modification by System Organ Class and Preferred Term - Dose Expansion
Safety Analysis Set

#### Table 14.3.2.8.1

Summary of WTX-330-related Treatment-Emergent Adverse Events Leading to WTX-330 Modification by System Organ Class and Preferred Term - Dose Escalation
Safety Analysis Set

Programming Note: Add "Note: TEAEs related to study drug are events reported with 'Definitely Related', 'Probably', 'Possibly' or missing in the relationship."

#### Table 14.3.2.8.2

Summary of WTX-330-related Treatment-Emergent Adverse Events Leading to WTX-330 Modification by System Organ Class and Preferred Term - Dose Expansion
Safety Analysis Set

Programming Note: Add "Note: TEAEs related to study drug are events reported with 'Definitely Related', 'Probably', 'Possibly' or missing in the relationship."

#### Table 14.3.2.9.1

Summary of Immune Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set

# Table 14.3.2.9.2

Summary of Immune Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set

Date: 26Feb2025

## Table 14.3.2.10.1

Summary of Treatment-Emergent Adverse Events of Infusion Related Reaction by System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set

# Table 14.3.2.10.2

Summary of Treatment-Emergent Adverse Events of Infusion Related Reaction by System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set

# Table 14.3.2.11.1

Summary of Treatment-Emergent Adverse Events of Cytokine Release Syndrome by System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set

## Table 14.3.2.11.2

Summary of Treatment-Emergent Adverse Events of Cytokine Release Syndrome by System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set

Date: 26Feb2025

Table 14.3.2.12.1

Summary of Treatment-Emergent Adverse Events of Special Interest by Special Interest Category and Preferred Term - Dose Escalation

Safety Analysis Set

| | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | |
| Special Interest Category/ | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| Preferred Term | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=xX) |
| Patients with Any Event, n(%) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Special Interest Category#1 | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred Term #1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred Term #2 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| <insert></insert> | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Special Interest Category#2 | X (XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | XX(XX.X) |
| Preferred Term #1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred Term #2 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| <insert></insert> | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |

#### <insert>

Note: Adverse Events are coded with MedDRA version 26.0.

Note: A TEAE is defined as an AEs that emerges or worsens (i.e. increase in CTCAE grade/ASTCT Grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

Note: Each subject is counted only once in each category. The table is sorted by Special Interest Category count in total, and Preferred Term count in total within each Special Interest Category.

# Programming Note:

Sort by Special Interest Category count in total, and PT count in total within each Special Interest Category
Special Interest Category include >=Grade 2 CRS, >= Grade 3 Oral Mucositis, Hy's Law or >= Grade 3 increased ALT or AST

Date: 26Feb2025

Table 14.3.2.12.2

Summary of Treatment-Emergent Adverse Events of Special Interest by Special Interest Category and Preferred Term - Dose Expansion Safety Analysis Set

| Special Interest Category/ | Arm A | Arm B | Total |
|-------------------------------|-----------|----------|-----------|
| Preferred Term | (N=XX) | (N=XX) | (N=XX) |
| Patients with Any Event, n(%) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| Special Interest Category#1 | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| Preferred Term #1 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Preferred Term #2 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| <insert></insert> | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| Special Interest Category#2 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Preferred Term #1 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Preferred Term #2 | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| <insert></insert> | XX(XX.X) | XX(XX.X) | XX(XX.X) |

<insert>

Note: Arm A = Patients with indications for which a CPI is indicated/approved; Arm B = Patients with tumor types for which CPI therapy is not indicated/approved.

Note: Adverse Events are coded with MedDRA version 26.0.

Note: A TEAE is defined as an AEs that emerges or worsens (i.e. increase in CTCAE grade/ASTCT Grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

Note: Each subject is counted only once in each category. The table is sorted by Special Interest Category count in total, and Preferred Term count in total within each Special Interest Category.

# Programming Note:

Sort by Special Interest Category count in total, and PT count in total within each Special Interest Category
Special Interest Category include >= Grade 2 CRS, >= Grade 3 Oral Mucositis, Hy's Law or >= Grade 3 increased ALT or AST

Date: 26Feb2025

# Table 14.3.2.13.1 Summary of Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum CTCAE/ASTCT Grade - Dose Escalation Safety Analysis Set

Dose Escalation - WTX-330 0.016 mg/kg (N=xx)

| System Organ Class/ | | | Maximum CTCAE/ | ASTCT Grade | | | |
|---|---|---|---|---|---|---|---|
| Preferred Term/ | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 | Grade 3+ | Total |
| Patients with Any Event, n(%) | X(XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | XX(XX.X) |
| System Organ Class #1 | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | XX(XX.X) |
| Preferred Term #1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred Term #2 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| <insert></insert> | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| System Organ Class #2 | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | XX(XX.X) |
| Preferred Term #1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred Term #2 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| <insert></insert> | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |

Note: Adverse Events are coded with MedDRA version 26.0 and graded with CTCAE Grade 5.0, except for Cytokine Release Syndrome which is graded with ASTCT Grade.

Note: A TEAE is defined as an AEs that emerges or worsens (i.e. increase in CTCAE grade/ASTCT Grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

Note: Each subject is counted only once at maximum CTCAE Grade in each category. Table is sorted by System Organ Class count in total, and Preferred Term count in total within each System Organ Class.

# **Programming note:**

• Repeat all dose levels and total on a new page.

Date: 26Feb2025

Repeat table 14.3.2.13.1 for the following tables, except for the column header and footnote for Dose Expansion.

Table 14.3.2.13.2

Summary of Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum CTCAE/ASTCT Grade - Dose Expansion Safety Analysis Set

Table 14.3.2.14.1

Summary of WTX-330-related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum CTCAE/ASTCT Grade - Dose Escalation
Safety Analysis Set

Programming Note: Add "Note: TEAEs related to study drug are events reported with 'Definitely Related', 'Probably', 'Possibly' or missing in the relationship."

Table 14.3.2.14.2

Summary of WTX-330-related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum CTCAE/ASTCT Grade - Dose Expansion Safety Analysis Set

Date: 26Feb2025

Table 14.3.2.15.1

Summary of Treatment-Emergent Adverse Events by Preferred Term - Dose Escalation
Safety Analysis Set

| Preferred Term | WTX-330<br>0.016<br>mg/kg<br>(N=x) | WTX-330<br>0.032<br>mg/kg<br>(N=x) | WTX-330<br>0.056<br>mg/kg<br>(N=x) | WTX-330<br>0.084<br>mg/kg<br>(N=x) | WTX-330<br>0.126<br>mg/kg<br>(N=x) | WTX-330<br>0.190<br>mg/kg<br>(N=x) | WTX-330<br>0.290<br>mg/kg<br>(N=x) | WTX-330<br>0.XXX<br>mg/kg<br>(N=x) | Total (N=xX) |
|---|---|---|---|---|---|---|---|---|---|
| Patients with Any Event, n(%) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred Term #1 | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred Term #2 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred Term #3 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Preferred Term #4 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| <insert></insert> | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |

Note: Adverse Events are coded with MedDRA version 26.0.

Note: A TEAE is defined as an AEs that emerges or worsens (i.e. increase in CTCAE grade/ASTCT grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

Note: Each subject is counted only once in each category. The table is sorted by Preferred Term count in total.

Repeat table 14.3.2.15.1 for the following tables, except for the column header and footnote for Dose Expansion.

Table 14.3.2.15.2 Summary of Treatment-Emergent Adverse Events by Preferred Term - Dose Expansion Safety Analysis Set

Date: 26Feb2025

Repeat table 14.3.2.1a for the following tables, except for the column header and footnote for Dose expansion.

## Table 14.3.3.1.1

Summary of Treatment-Emergent Serious Adverse Events by System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set

#### Table 14.3.3.1.2

Summary of Treatment-Emergent Serious Adverse Events by System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set

Table 14.3.3.2.1Summary of WTX-330-related Treatment-Emergent Serious Adverse Events by System Organ Class and Preferred Term - Dose Escalation
Safety Analysis Set

Programming Note: Add "Note: TEAEs related to study drug are events reported with 'Definitely Related', 'Probably', 'Possibly' or missing in the relationship."

#### Table 14.3.3.2.2

Summary of WTX-330-related Treatment-Emergent Serious Adverse Events by System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set

Date: 26Feb2025

Repeat table 14.3.2.13.1 for the following tables, except for the column header and footnote for Dose Expansion.

#### Table 14.3.3.3.1

Summary of Treatment-Emergent Serious Adverse Events by System Organ Class, Preferred Term and Maximum CTCAE /ASTCT Grade - Dose Escalation
Safety Analysis Set

## Table 14.3.3.3.2

Summary of Treatment-Emergent Serious Adverse Events by System Organ Class, Preferred Term and Maximum CTCAE /ASTCT Grade - Dose Expansion
Safety Analysis Set

## Table 14.3.3.4.1

Summary of WTX-330-related Treatment-Emergent Serious Adverse Events by System Organ Class, Preferred Term and Maximum CTCAE /ASTCT Grade - Dose Escalation
Safety Analysis Set

Programming Note: Add "Note: TEAEs related to study drug are events reported with 'Definitely Related', 'Probably', 'Possibly' or missing in the relationship."

#### Table 14.3.3.4.2

Summary of WTX-330-related Treatment-Emergent Serious Adverse Events by System Organ Class, Preferred Term and Maximum CTCAE /ASTCT Grade - Dose Expansion
Safety Analysis Set

Date: 26Feb2025

Repeat table 14.3.2.15.1 for the following tables, except for the column header and footnote for Dose Expansion.

Table 14.3.3.5.1

Summary of Treatment-Emergent Serious Adverse Events by Preferred Term - Dose Escalation Safety Analysis Set

Table 14.3.3.5.2

Summary of Treatment-Emergent Serious Adverse Events by Preferred Term - Dose Expansion Safety Analysis Set

Table 14.3.3.6.1

Summary of WTX-330-related Treatment-Emergent Serious Adverse Events by Preferred Term - Dose Escalation Safety Analysis Set

Programming Note: Add "Note: TEAEs related to study drug are events reported with 'Definitely Related', 'Probably', 'Possibly' or missing in the relationship."

Table 14.3.3.6.2

Summary of WTX-330-related Treatment-Emergent Serious Adverse Events by Preferred Term - Dose Expansion Safety Analysis Set

Date: 26Feb2025

Repeat table 14.3.2.1.1 for the following tables, except for the column header and footnote for Dose Expansion.

## Table 14.3.3.7.1

Summary of Treatment-Emergent Adverse Events Leading Death by System Organ Class and Preferred Term - Dose Escalation Safety Analysis Set

# Table 14.3.3.7.2

Summary of Treatment-Emergent Adverse Events Leading Death by System Organ Class and Preferred Term - Dose Expansion Safety Analysis Set

Date: 26Feb2025

Table 14.3.3.8.1
Summary of Death - Dose Escalation
Safety Analysis Set

| | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | |
| | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=xX) |
| Death on Study, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Primary Cause of Death | | | | | | | | | |
| Disease Progression | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Adverse Event | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Unknown | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Death within 30 Days of last study drug, n(%) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | XX (XX.X) |
| Primary Cause of Death | | | | | | | | | |
| Disease Progression | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Adverse Event | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Unknown | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Other | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Death after 30 Days of last study drug, $n(%)$ | X(XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | XX (XX.X) |
| Primary Cause of Death | | | | | | | | | |
| Disease Progression | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Adverse Event | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | XX(XX.X) |
| Unknown | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | XX(XX.X) |
| Other | X (XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | XX(XX.X) |

Repeat table 14.3.3.8.1 for the following tables, except for the column header and footnote for Dose Expansion.

Table 14.3.3.8.2 Summary of Death - Dose Expansion Safety Analysis Set
Date: 26Feb2025

Table 14.3.7.1.1

Summary of Hematology Laboratory by Visit - Dose Escalation
Safety Analysis Set

Test (SI unit): Hemoglobin (g/L)

| | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | |
| | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=xX) |
| Baseline | | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Cycle 1 Day X | | | | | | | | | |
| Absolute Value | | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Change from Baseline | | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

<insert Visit>

Note: Baseline is defined as the last non-missing value prior to the first WTX-330 dose.

#### **Programming instruction:**

Each parameter starts from a new page, including Red blood cell (RBC) count, hemoglobin (Hb), hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH); white blood cell (WBC) count and differentials, absolute lymphocyte count (ALC), and absolute neutrophil count (ANC), platelet count.

Date: 26Feb2025

Repeat table 14.3.7.1.1 for the following tables, except for the column header and footnote.

Table 14.3.7.1.2 Summary of Hematology Laboratory by Visit - Dose Expansion Safety Analysis Set

Date: 26Feb2025

Table 14.3.7.1.3

Shift of Hematology CTCAE Grade from Baseline to Worst Post-baseline - Dose Escalation Safety Analysis Set

Test: Anemia (Hypo-Hemoglobin)

| | _ | | Wo | rst Post-bas | eline CTCAE ( | Grade, n(%) | | |
|---|---|---|---|---|---|---|---|---|
| | Baseline<br>CTCAE Grade | Missing | 0 | 1 | 2 | 3 | 4 | Total |
| WTX-330 0.016 mg/kg (N=xx) | Missing | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | 0 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | 1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | 2 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | 3 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | 4 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Total | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| WTX-330 0.032 mg/kg (N=xx) | Missing | X(XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) |
| | 0 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | 1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | 2 | X(XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | 3 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | 4 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Total | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| <insert dose="" levels=""></insert> | | | | | | | | |
| Total (N=xx) | Missing | X (XX.X) | X (XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) |
| | 0 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | 1 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | 2 | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | 3 | X(XX.X) | X(XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | X(XX.X) |
| | 4 | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Total | X(XX.X) | X(XX.X) | X (XX.X) | X (XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |

Note: Baseline is defined to be the last non-missing value prior to the first WTX-330 dose.

Programming instruction:

Each parameter starts from a new page.

Date: 26Feb2025

Repeat table 14.3.7.1.3 for the following tables, except for the column header.

Table 14.3.7.1.4

Shift of Hematology CTCAE Grade from Baseline to Worst Post-baseline - Dose Expansion Safety Analysis Set

Programming instruction: Replace dose levels with Arm A and Arm B Add footnote for Dose expansion.

Date: 26Feb2025

Table 14.3.7.1.5

Shift of Hematology Tests without CTCAE Grade from Baseline to Lowest/Highest Post-baseline - Dose Escalation
Safety Analysis Set

Test: Red blood cells (RBC) count

| | | | | Baseline n(%) | | |
|---|---|---|---|---|---|---|
| | Lowest/Highest Post-baseline | Missing | Low | Normal | High | Total |
| WTX-330 0.016 mg/kg | (N=xx) Lowest Post-baseline Value | | | | | |
| | Missing | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Low | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Normal | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | High | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Total | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Highest Post-baseline Value | | | | | |
| | Missing | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Low | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Normal | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | High | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Total | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| <pre><insert dose="" levels=""></insert></pre> | | | | | | |
| Total (N=xx) | Lowest Post-baseline Value | | | | | |
| | Missing | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Low | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Normal | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | High | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Total | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Highest Post-baseline Value | | | | | |
| | Missing | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Low | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Normal | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | High | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |
| | Total | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) |

Note: Baseline is defined to be the last non-missing value prior to the first WTX-330 dose.

Programming instruction:

Each parameter starts from a new page.

Date: 26Feb2025

Repeat table 14.3.7.1.5 for the following tables, except for the column header and footnote for Dose Expansion.

Table 14.3.7.1.6
Shift of Hematology Tests without CTCAE Grade from Baseline to Lowest/Highest Post-baseline - Dose Expansion Safety Analysis Set

Programming instruction: Replace dose levels with Arm A and Arm B Add footnote for Dose expansion.

Date: 26Feb2025

Repeat table 14.3.7.1.1 for the following tables, except for the column header and footnote for Dose Expansion.

Table 14.3.7.2.1 Summary of Chemistry Laboratory by Visit - Dose Escalation Safety Analysis Set

Programming instruction:

Each parameter starts from a new page, including Calcium, magnesium, potassium, sodium, bicarbonate, chloride phosphate, albumin, total blood urea nitrogen (BUN), C-reactive protein (CRP), creatinine, urate, estimated glomerular filtration rate, glucose, Alanine transaminase (ALT), aspartate transaminase (AST), bilirubin, alkaline phosphatase (ALP), lactic acid dehydrogenase (LDH), gamma-glutamyl transferase (GGT)

Table 14.3.7.2.2 Summary of Chemistry Laboratory by Visit - Dose Expansion Safety Analysis Set

Programming instruction:

Each parameter starts from a new page, including Calcium, magnesium, potassium, sodium, bicarbonate, chloride phosphate, albumin, total blood urea nitrogen (BUN), C-reactive protein (CRP), creatinine, urate, estimated glomerular filtration rate, glucose, Alanine transaminase (ALT), aspartate transaminase (AST), bilirubin, alkaline phosphatase (ALP), lactic acid dehydrogenase (LDH), gamma-glutamyl transferase (GGT)

Date: 26Feb2025

Repeat table 14.3.7.1.3 for the following tables, except for the column header and footnote for Dose Expansion.

Table 14.3.7.2.3

Shift of Chemistry CTCAE Grade from Baseline to Worst Post-baseline - Dose Escalation Safety Analysis Set

Table 14.3.7.2.4

Shift of Chemistry CTCAE Grade from Baseline to Worst Post-baseline - Dose Expansion Safety Analysis Set

Repeat table 14.3.7.1.5 for the following tables, except for the column header and footnote for Dose Expansion.

Table 14.3.7.2.5

Shift of Chemistry Tests without CTCAE Grade from Baseline to Lowest/Highest Post-baseline - Dose Escalation Safety Analysis Set

Table 14.3.7.2.6

Shift of Chemistry Tests without CTCAE Grade from Baseline to Lowest/Highest Post-baseline - Dose Expansion Safety Analysis Set

Date: 26Feb2025

Table 14.3.7.2.7

Summary of Clinically Significant Liver Function Tests - Dose Escalation Safety Analysis Set

| | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | |
| | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=xX) |
| Aspartate Aminotransferase (AST),n (%) | | | | | | | | | |
| > 3 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| > 5 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| > 10 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| > 20 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Alanine Aminotransferase (ALT),n (%) | | | | | | | | | |
| > 3 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| > 5 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| > 10 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| > 20 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| AST or ALT, n (%) | | | | | | | | | |
| > 3 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| > 5 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| > 10 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| > 20 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Total Bilirubin (TBL),n (%) | | | | | | | | | |
| > 1.5 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| > 2 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Alkaline Phosphatase (ALP),n (%) | | | | | | | | | |
| > 1.5 x ULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| (AST or ALT) and TBL,n (%) | | | | | | | | | |
| AST or ALT>3xULN and TBL>1.5xULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| AST or ALT>3xULN and TBL>2xULN | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |

Date: 26Feb2025

Repeat table 14.3.7.2.7 for the following tables, except for the column header and footnote for Dose Expansion.

Table 14.3.7.2.8

Summary of Clinically Significant Liver Function Tests - Dose Expansion Safety Analysis Set

Date: 26Feb2025

Repeat table 14.3.7.1.1 for the following tables, except for the column header and footnote for Dose Expansion.

Table 14.3.7.3.1

Summary of Coagulation Laboratory by Visit - Dose Escalation Safety Analysis Set

Programming instruction:

Each parameter starts from a new page, including Prothrombin time (PT) or International normalized ratio (INR), and Partial thromboplastin time (PTT) or Activated partial thromboplastin time (APTT).

Table 14.3.7.3.2

Summary of Coagulation Laboratory by Visit - Dose Expansion Safety Analysis Set

Programming instruction:

Each parameter starts from a new page, including Prothrombin time (PT) or International normalized ratio (INR), and Partial thromboplastin time (PTT) or Activated partial thromboplastin time (APTT).

Date: 26Feb2025

Repeat table 14.3.7.1.3 for the following tables, except for the column header and footnote for Dose Expansion.

Table 14.3.7.3.3

Shift of Coagulation CTCAE Grade from Baseline to Worst Post-baseline - Dose Escalation Safety Analysis Set

Table 14.3.7.3.4

Shift of Coagulation CTCAE Grade from Baseline to Worst Post-baseline - Dose Expansion Safety Analysis Set

Repeat table 14.3.7.1.5 for the following tables, except for the column header and footnote for Dose Expansion.

Table 14.3.7.3.5

Shift of Coagulation Tests without CTCAE Grade from Baseline to Lowest/Highest Post-baseline - Dose Escalation Safety Analysis Set

Table 14.3.7.3.6

Shift of Coagulation Tests without CTCAE Grade from Baseline to Lowest/Highest Post-baseline - Dose Expansion Safety Analysis Set

Date: 26Feb2025

Repeat table 14.3.7.1.1 for the following table, except for the column header and footnote for Dose Expansion.

Table 14.3.8.1 Summary of Vital Signs by Visit - Dose Escalation Safety Analysis Set

Table 14.3.8.2 Summary of Vital Signs by Visit - Dose Expansion Safety Analysis Set

Date: 26Feb2025

Table 14.3.8.3

Summary of Vital Signs Clinically Significant on Treatment - Dose Escalation Safety Analysis Set

| | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | _ |
| | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| Abnormal Categories, n(%) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=xX) |
| Systolic BP | | | | | | | | | |
| ≥180mmHg and an increase ≥20mmHg from baseline | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| ≤90mmHg and a decrease ≥20mmHg from baseline | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Diastolic BP | | | | | | | | | |
| ≥105mmHg and an increase ≥15mmHg from baseline | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| $\leq$ 50mmHg and a decrease $\geq$ 15mmHg from baseline | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Weight | | | | | | | | | |
| Increase of ≥10% from baseline | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Decrease of ≥10% from baseline | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | XX (XX.X) |
| Heart rate | | | | | | | | | |
| | 37 (3737 37) | V (VV V) | V (VV V) | V (VV V) | V (VV V) | 37 /3737 37 \ | 37 (3737 37) | 37 /3737 37) | 3/3/ /3/3/ 3/\ |
| ≥120bpm with an increase ≥15bpm from baseline | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | X (XX.X) | XX (XX.X) |
| ≤50bpm and a decrease ≥15bpm from baseline | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Temperature | | | | | | | | | |
| >38° C | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| <35° C | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |

Date: 26Feb2025

Repeat table 14.3.8.3 for the following table, except for the column header and footnote for Dose Expansion.

Table 14.3.8.4

Summary of Vital Signs Clinically Significant on Treatment - Dose Expansion Safety Analysis Set

Date: 26Feb2025

Repeat table 14.3.7.1.1 for the following table, except for the column header and footnote for Dose Expansion.

Table 14.3.9.1 Summary of Electrocardiograms by Visit - Dose Escalation Safety Analysis Set

Table 14.3.9.2 Summary of Electrocardiograms by Visit - Dose Expansion Safety Analysis Set

Date: 26Feb2025

Table 14.3.9.3

Summary of QTcF Categories - Dose Escalation
Safety Analysis Set

| | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | |
| | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| QTcF Categories, n(%) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=xX) |
| Baseline | | | | | | | | | |
| QTcF >450 msec | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| QTcF >480 msec | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| QTcF >500 msec | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Highest Post-Baseline | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| QTcF >450 msec | | | | | | | | | |
| QTcF >480 msec | | | | | | | | | |
| QTcF >500 msec | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Highest Change from Baseline | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| >30 msec | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| >60 msec | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| Cycle x Day y, Timepoint | | | | | | | | | |
| QTcF >450 msec | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| QTcF >480 msec | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| QTcF >500 msec | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) |
| <pre><insert and="" timepoints="" visits=""></insert></pre> | | | | | | | | | |

### Programming notes:

The categories ("QTc > 450m msec", "QTc > 480m msec", "QTc > 500m msec", ">30 msec", ">60 msec") are non-mutually exclusive categories.

Date: 26Feb2025

Repeat table 14.3.9.3 for the following table, except for the column header and footnote for Dose Expansion.

Table 14.3.9.4 Summary of QTcF Categories - Dose Expansion Safety Analysis Set

Date: 26Feb2025

Dose Escalation: WTX-330 0.016 mg/kg (N=x)

| | | | | | | Coefficient of |
|---|---|---|---|---|---|---|
| | | Mean (Standard | | | Geometric | variation for |
| Timepoints | n | Deviation) | Median | Min, Max | Mean | Geometric Mean |
| Cycle 1 Day 1 | | | | | | |
| Pre-dose | XX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | XX.XX |
| Immediately after (±5 minutes) WTX-330 infusion | XX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | XX.XX |
| 4 hours (±30 minutes) post start of WTX-330 infusion | XX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | XX.XX |
| 8 hours (±30 minutes) post start of WTX-330 infusion | XX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | XX.XX |
| 24 hours (±2 hours) post start of WTX-330 infusion | XX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | XX.XX |
| 48 hours (±2 hours) post start of WTX-330 infusion | XX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | XX.XX |
| 168 hours (±4 hours) post start of WTX-330 Infusion | XX | xx.x(xx.xx) | XX.X | xx,xx | XX.X | XX.XX |
| Cycle 1 Day 15 | | | | | | |
| Pre-dose | XX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | xx.xx |
| Immediately after (±5 minutes) WTX-330 infusion | XX | xx.x(xx.xx) | XX.X | xx,xx | XX.X | XX.XX |
| Cycle 1 Day 21 | | | | | | |
| Pre-dose | xx | xx.x(xx.xx) | XX.X | xx,xx | XX.X | xx.xx |
| Immediately after (±5 minutes) WTX-330 infusion | XX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | xx.xx |
| 4 hours (±30 minutes) post start of WTX-330 infusion | XX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | xx.xx |
| 8 hours (±30 minutes) post start of WTX-330 infusion | XX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | xx.xx |
| 24 hours (±2 hours) post start of WTX-330 infusion | XX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | xx.xx |
| 48 hours (±2 hours) post start of WTX-330 infusion | XX | xx.x(xx.xx) | XX.X | XX,XX | XX.X | xx.xx |
| 168 hours (±4 hours) post start of WTX-330 Infusion | XX | xx.x(xx.xx) | XX.X | xx,xx | XX.X | XX.XX |
| Cycle X Day Y | | | | | | |
| Pre-dose | XX | xx.x(xx.xx) | XX.X | xx,xx | XX.X | XX.XX |

## Programming Note:

Each Dose Escalation dose level will start from a new page.

Vendor data will need to be divided by 1000 to report in CSR as ug/mL.

Date: 26Feb2025

The following table will be displayed as Table 14.4.1.1

Table 14.4.1.2 Summary of Free IL-12 Plasma Concentration (pg/mL) by Timepoint Pharmacokinetic Analysis Set

Programming Note:

Units for Free IL-12, use pg/ml - multiply vendor conc by 1000

Date: 26Feb2025

Table 14.4.2.1
Summary of WTX-330 Pharmacokinetic Parameters
Pharmacokinetic Analysis Set

Visit: Cycle 1 Day 1

| | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | WTX-330 | |
|---|---|---|---|---|---|---|---|---|---|
| | 0.016 | 0.032 | 0.056 | 0.084 | 0.126 | 0.190 | 0.290 | 0.XXX | |
| | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | mg/kg | Total |
| Parameter (unit) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=x) | (N=xX) |
| C <sub>max</sub> (ug/mL) | | | | | | | | | |
| n | X | X | X | X | X | X | X | X | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX |
| Geometric Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CV for Geometric Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| T <sub>max</sub> (hours) | | | | | | | | | |
| n | X | X | X | X | X | X | X | X | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX |

<insert Parameter>

Nore: CV = Coefficient of variation.

Programming Note:

Includes all PK parameters

Repeat table for Cycle 2 Day 1

T<sub>max</sub> and T<sub>last</sub> summary will no include Geometric Mean, Coefficient of variation

The following table will be displayed as Table 14.4.2.1,

**Table** 14.4.2.2

Summary of Free IL-12 Pharmacokinetic Parameters Pharmacokinetic Analysis Set

#### Programming Note:

Units for Free IL-12, use pg/ml - multiply vendor conc by 1000


Date: 26Feb2025

Table 14.4.3.1

Summary of Anti-drug Antibody for WTX-330 - Dose Escalation and **Dose Expansion**Anti-Drug Antibody Analysis Set

| | WTX-330<br>0.016<br>mg/kg<br>(N=x) | WTX-330<br>0.032<br>mg/kg<br>(N=x) | WTX-330<br>0.056<br>mg/kg<br>(N=x) | WTX-330<br>0.084<br>mg/kg<br>(N=x) | WTX-330<br>0.126<br>mg/kg<br>(N=x) | WTX-330<br>0.190<br>mg/kg<br>(N=x) | WTX-330<br>0.290<br>mg/kg<br>(N=x) | WTX-330<br>0.XXX<br>mg/kg<br>(N=x) | Total<br>(N=xX) |
|---|---|---|---|---|---|---|---|---|---|
| ADA at Baseline, n(%) | | | | | | | | | |
| Positive | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Negative | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Unknown | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| ADA at Post-Baseline, n(%) | | | | | | | | | |
| At least one positive | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| All negative | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Unknown | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Treatment-induced ADA, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Treatment-boosted ADA, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |
| Treatment-unaffected ADA, n(%) | X(XX.X) | X(XX.X) | X(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) | XX(XX.X) |

Note: Treatment-induced ADA is defined as those patients with no ADA at baseline and one or more post-treatment (Cycle 1 Day 15 and later) ADA-positive sample. Treatment-boosted ADA is defined as patients with a positive baseline ADA result who had one or more post-treatment (Cycle 1 Day 15 and later) ADA result with a higher titer than that of the baseline ADA sample. Treatment-unaffected ADA, defined as patients with a positive baseline ADA result who had post-treatment (Cycle 1 Day 15 and later) ADA result with a lower titer than that of the baseline ADA sample in all visits.

Note: Dose escalation and dose expansion are summarized together by dose level.

#### Programming Note:

Combine Dose Escalation and Dose Expansion and summary the results by dose level

Date: 26Feb2025

## Figure Shells

Date: 26Feb2025

Figure 14.4.1.1.1

Semi-logarithmic Plot and Linear Plot for Individual WTX-330 Plasma Concentrations versus Time at Cycle 1 - Dose Escalation Pharmacokinetic Analysis Set



- Different WTX-330 dose levels used different colors. Add legend to indicate dose level by color
- Each subject will be plotted in one line

Date: 26Feb2025

Repeat Figure 14.4.1.1.1 for the following figures, except for the Treatment.

#### Figure 14.4.1.1.2

Semi-logarithmic Plot and Linear Plot for Individual WTX-330 Plasma Concentrations versus Time at Cycle 2 - Dose Escalation Pharmacokinetic Analysis Set

#### Figure 14.4.1.1.3

Semi-logarithmic Plot and Linear Plot for Individual Free IL-12 Plasma Concentrations versus Time at Cycle 1 - Dose Escalation Pharmacokinetic Analysis Set

#### Programming Note:

Units for Free IL-12, use pg/ml - multiply vendor conc by 1000

#### Figure 14.4.1.1.4

Semi-logarithmic Plot and Linear Plot for Individual Free IL-12 Plasma Concentrations versus Time at Cycle 2 - Dose Escalation Pharmacokinetic Analysis Set

#### Programming Note:

Units for Free IL-12, use pg/ml - multiply vendor conc by 1000

Date: 26Feb2025

Figure 14.4.1.2.1

Semi-logarithmic Plot and Linear Plot for Mean WTX-330 Plasma Concentrations versus Time at Cycle 1 - Dose Escalation
Pharmacokinetic Analysis Set



Note: The error bars indicate the standard error (SE).

- Different WTX-330 dose levels used different colors in Dose Escalation. Add legend to indicate dose level by color
- Add  $\pm$  SE in the plot (not SD)

Date: 26Feb2025

Repeat Figure 14.4.1.2.1 for the following figures, except for the Treatment.

#### Figure 14.4.1.2.2

Semi-logarithmic Plot and Linear Plot for Mean WTX-330 Plasma Concentrations versus Time at Cycle 2 - Dose Escalation Pharmacokinetic Analysis Set

#### Figure 14.4.1.2.3

Semi-logarithmic Plot and Linear Plot for Mean Free IL-12 Plasma Concentrations versus Time at Cycle 1 - Dose Escalation Pharmacokinetic Analysis Set

### Programming Note:

Units for Free IL-12, use pg/ml - multiply vendor conc by 1000

#### Figure 14.4.1.2.4

Semi-logarithmic Plot and Linear Plot for Mean Free IL-12 Plasma Concentrations versus Time at Cycle 2 - Dose Escalation Pharmacokinetic Analysis Set

#### Programming Note:

Units for Free IL-12, use pg/ml - multiply vendor conc by 1000

Date: 26Feb2025

#### **Listing Shells**

#### **Programming Note:**

The data will be listed in each listing based on the following sequence if the cohort is available (new dose levels might be added upon protocol amendment):

Dose Escalation: WTX-330 0.016 mg/kg Dose Escalation: WTX-330 0.032 mg/kg Dose Escalation: WTX-330 0.056 mg/kg Dose Escalation: WTX-330 0.084 mg/kg Dose Escalation: WTX-330 0.126 mg/kg Dose Escalation: WTX-330 0.190 mg/kg Dose Escalation: WTX-330 0.290 mg/kg Dose Escalation: WTX-330 0.XXX mg/kg

Dose Expansion (Arm A): Head and Neck Squamous Cell Carcinoma

Dose Expansion (Arm A): Non-small Cell Lung Cancer

Dose Expansion (Arm A): Renal Cell Carcinoma

Dose Expansion (Arm A): XXXXXXXXXXXXXXXXX

Dose Expansion (Arm B): Colorectal Carcinoma

Dose Expansion (Arm B): Diffuse Large B-cell Lymphoma

Dose Expansion (Arm B): Follicular Lymphoma

Dose Expansion (Arm B): YYYYYYYYYYYYYY

Date: 26Feb2025

#### Listing 16.2.2.1 Subject Disposition Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level and/or Arm/Disease)

| Discontinuation<br>(Study Day)<br>DDMMMYYY (XX) | Reason for Study Discontinuation Withdrawal of consent by the patient |
|---|---|
| DDMMMYYY (XX) | Withdrawal of concent by the nationt |
| | withdrawar or consent by the pattern |
| DDMMMYYY (XX) | Loss to follow-up |
| DDMMMYYY (XX) | Complete the Study |
| DDMMMYYY (XX) | Study termination by Sponsor |
| DDMMMYYY (XX) | COVID-19 Related: MH #2 |
| DDMMMYYY (XX) | Other: XXXXXX |
| DDMMMYYY (XX) | Death |
| DDMMMYYY (XX) | Complete the Study |
| | DDMMMYYY (XX) DDMMMYYY (XX) DDMMMYYY (XX) DDMMMYYY (XX) DDMMMYYY (XX) |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: PD = Progressive Disease.

- \* Sorting order is by Subject ID
- \* Repeat each dose level and/or arm on a separate page.
- \* if 'Did the Subject Complete the Study?' = Yes, please assign 'Complete the Study' for reason for study Discontinuation

Date: 26Feb2025

## Listing 16.2.2.2 Safety and Survival Status Follow-Up Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level and/or Arm/Disease)

| | | | Date of Last Known | New Surgery or Therapy?: | Continuing |
|---|---|---|---|---|---|
| Subject | Date of Contact | Subject | to Be Alive | Radiotherapy/Antineoplastic | in Survival |
| ID/Age/Sex | (Study Day) | Status | (Study Day) | Surgery/Anticancer Medications | Monitoring? |
| XXXX-XX/xx/M | DDMMMYYYY (xx) | Alive | DDMMMYYY (XX) | No | Yes |
| | DDMMMYYYY (xx) | Lost to follow up | | | |
| XXXX-XX/xx/F | DDMMMYYYY (xx) | Alive | DDMMMYYY (XX) | Yes: XXXXXXXXXX/ /XXXXXXXXXXXXXXXX | Yes |
| | DDMMMYYYY (xx) | Alive | DDMMMYYY (XX) | Yes: / / XXXXXXXXXXXXXXXX | Yes |
| | DDMMMYYYY (xx) | Dead | | | |
| XXXX-XX/xx/M | DDMMMYYYY (xx) | Alive | DDMMMYYY (XX) | No | Yes |
| | DDMMMYYYY (xx) | Alive | DDMMMYYY (XX) | Yes: XXXXXXXXXX/ / | Yes |
| | DDMMMYYYY (xx) | Lost to follow up | | | |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

### **Programming Note:**

\* Sorting order is by Subject ID, and Date of Contact.

Date: 26Feb2025

## Listing 16.2.2.3 Death Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level and/or Arm/Disease)

| Subject | Date of Death | |
|---|---|---|
| ID/Age/Sex | (Study Day) Primary Reason for Death | Death Period |
| XXXX-XXX/xx/M | DDMMMYYYY (xx) Disease Progression | Death within 30 Days of last study drug |
| XXXX-XXX/xx/F | DDMMMYYYY (xx) Adverse Event: #1, #4 | Death within 30 Days of last study drug |
| XXXX-XXX/xx/F | DDMMMYYYY (xx) Unknown | Death within 30 Days of last study drug |
| XXXX-XXX/xx/M | DDMMMYYYY (xx) Other: XXXXXXXXXXXXXXXX | Death after 30 Days of last study drug |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

- \* Sorting order is by Subject ID.
- \* Repeat each dose level and/or arm on a separate page.

Date: 26Feb2025

## Listing 16.2.3 Deviations from the Clinical Protocol Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level and/or Arm/Disease)

| | Date of Protocol | | | |
|---|---|---|---|---|
| Subject | Deviation | | | |
| ID/Age/Sex | (Study Day) | Protocol Deviation Term | Protocol Category | Major/Minor |
| XXXX-XXX/xx/M | DDMMMYYYY (xx) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXX | Minor |
| XXXX-XXX/xx/F | DDMMMYYYY (xx) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Minor |
| XXXX-XXX/xx/F | DDMMMYYYY (xx) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Minor |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

#### **Programming Note:**

\* Sorting order is by Subject ID, Date of Protocol Deviation.

Date: 26Feb2025

#### Listing 16.2.4.1 Demographic Data Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level and/or Arm/Disease)

| Subject | Date of Birth/ | Age | | Childbearing | | |
|---|---|---|---|---|---|---|
| ID/Age/Sex | Age | Group | Sex | Potential? | Ethnicity | Race |
| XXXX-XXX/xx/I | M DDMMMYYYY/28 | <45 | Male | | Hispanic or Latino | American Indian or Alaskan Native |
| XXXX-XXX/xx/I | F DDMMMYYYY/37 | <45 | Male | | Not Hispanic or Latino | Asian |
| XXXX-XXX/xx/I | F DDMMMYYYY/40 | <45 | Female | Yes | Not Reported | Black or African American |
| XXXX-XXX/xx/1 | DDMMMYYYY/56 | ≥45-<65 | Male | | Unknown | Native Hawaiian or Other Pacific Islander |
| XXXX-XXX/xx/I | F DDMMMYYYY/70 | ≥65 | Female | No | Not Hispanic or Latino | White |
| XXXX-XXX/xx/1 | DDMMMYYYY/48 | ≥45-<65 | Male | | Not Hispanic or Latino | Not Reported |
| XXXX-XXX/xx/I | F DDMMMYYYY/80 | ≥65 | Female | No | Not Hispanic or Latino | White |
| XXXX-XXX/xx/N | DDMMMYYYY/66 | ≥65 | Male | | Not Reported | White |

<sup>\*</sup> Sorting order is by Subject ID

Date: 26Feb2025

# Listing 16.2.4.2 Baseline Characteristics Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level and/or Arm/Disease)

| Subject | Weight | Height | Hepatitis | Hepatitis | ECOG Performance |
|---------------|--------|--------|-----------|-----------|------------------|
| ID/Age/Sex | (kg) | (cm) | B Virus | C Virus | Status |
| XXXX-XXX/xx/M | XXX.X | XXX.X | Positive | Negative | 0 |
| XXXX-XXX/xx/F | XXX.X | XXX.X | Negative | Negative | 0 |
| XXXX-XXX/xx/F | XXX.X | XXX.X | Negative | Negative | 1 |
| XXXX-XXX/xx/M | XXX.X | XXX.X | Negative | Negative | 1 |
| XXXX-XXX/xx/F | XXX.X | XXX.X | Negative | Positive | 1 |
| XXXX-XXX/xx/M | XXX.X | XXX.X | Negative | Positive | 1 |
| XXXX-XXX/xx/M | XXX.X | XXX.X | Negative | Negative | 0 |
| XXXX-XXX/xx/F | XXX.X | XXX.X | Positive | Negative | 0 |
| | | | | _ | |

Note: Baseline is defined to be the last non-missing value prior to the first WTX-330 dose.

<sup>\*</sup> Sorting order is by Subject ID

Date: 26Feb2025

## Listing 16.2.5 Study Drug Extent of Exposure and Compliance Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level and/or Arm/Disease)

| | | Number Of | Total | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Duration of | Treatment | Planned | Cumulative | Treatment | Average Dose | Infusion | |
| Subject | Exposure | Cycle | Dose | Dose | Compliance | Intensity | Interruption | Subject with Dose |
| ID/Age/Sex | (week) | Started | (mg/kg) | (mg/kg) | (%) | ((mg/kg)/cycle) | Events | Adjustment |
| XXXX-XXX/xx/M | XXX | XX | XXX | XXX | XXX.X | XXX.X | 0 | No |
| XXXX-XXX/xx/F | XXX | XX | XXX | XXX | XXX.X | XXX.X | 0 | Yes/Missed |
| XXXX-XXX/xx/F | XXX | XX | XXX | XXX | XXX.X | XXX.X | 1 | Yes/Missed, Reduced |
| XXXX-XXX/xx/M | XXX | XX | XXX | XXX | XXX.X | XXX.X | 2 | Yes/Missed, Discontinued |
| XXXX-XXX/xx/F | XXX | XX | XXX | XXX | XXX.X | XXX.X | >=3 | No |
| XXXX-XXX/xx/M | XXX | XX | XXX | XXX | XXX.X | XXX.X | 2 | Yes/Missed, Reduced, |
| | | | | | | | | Interrupted, Discontinued |
| XXXX-XXX/xx/M | XXX | XX | XXX | XXX | XXX.X | XXX.X | >=3 | No |
| XXXX-XXX/xx/F | XXX | XX | XXX | XXX | XXX.X | XXX.X | 2 | Yes/ Missed |

Note: Duration of exposure (weeks) is (the date of last administration of WTX-330 - the date of first administration of WTX-330 + 14)/7.

Note: Total Planned Dose (mg/kg) is calculated by the sum of the individual Planned Dose Level being reported in eCRFs.

Note: Cumulative Dose (mg/kg) is calculated by sum of the individual Total Dose Administered being reported in eCRFs.

Note: Treatment compliance (%) is 100\*(Cumulative Dose/Total Planned Dose).

Note: Average Dose Intensity((mg/kg)/cycle) is calculated by Cumulative Dose/number of treatment cycles started (any amount of the study drug was administered).

- \* Sorting order is by Subject ID
- \* "Subject with Dose Adjustment" will be derived by concatenate all WTX-330 Administration records (remove duplicated dose adjustment)

Date: 26Feb2025

## Listing 16.2.6.1 Efficacy Parameters by RECIST 1.1 - Part 1 of 2 Evaluable Efficacy Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level and/or Arm/Disease)

| | | Duration of | | |
|---|---|---|---|---|
| Best Overall | Objective | Clinical Benefit | Response | Progression-Free |
| Response | Response | at Month 3/6/9 | (month) | Survival (month) |
| CR | Yes | Yes/Yes/Yes | XXX.X* | XXX.X* |
| SD | No | Yes/Yes/Yes | | XXX.X |
| SD | No | No/No/No | | XXX.X |
| PR | Yes | Yes/Yes/Yes | XXX.X | XXX.X* |
| PD | No | No/No/No | | XXX.X |
| SD | No | Yes/No/No | | XXX.X |
| SD | No | Yes/Yes/No | | XXX.X* |
| NE | No | No/No/No | | XXX.X |
| | Response CR SD SD PR PD SD SD SD | ResponseResponseCRYesSDNoSDNoPRYesPDNoSDNoSDNo | Response Response at Month 3/6/9 CR Yes Yes/Yes/Yes SD No Yes/Yes/Yes SD No No/No/No PR Yes Yes/Yes/Yes PD No No/No/No SD No Yes/No/No SD No Yes/Yes/No | Best Overall<br>ResponseObjective<br>ResponseClinical Benefit<br>at Month 3/6/9Response<br>(month)CRYesYes/Yes/YesXXX.X*SDNoYes/Yes/YesSDNoNo/No/NoPRYesYes/Yes/YesXXX.XPDNoNo/No/NoSDNoYes/No/NoSDNoYes/Yes/No |

Note: CR = Complete Response; PR = Partial Response; SD = Stable Disease; PD = Progressive Disease; NE = Not Evaluable.

Note: CR or PR of best overall response needs to be confirmed in a subsequent assessment at least 28 days apart. See the definition of each parameter in SAP section 8.2.

Note: \* indicates the censor.

#### **Programming Note:**

\* Sorting order is by Subject ID
Date: 26Feb2025

# Listing 16.2.6.2 Efficacy Parameters by iRECIST - Part 2 of 2 Evaluable Efficacy Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | Best | | | | | | |
|---|---|---|---|---|---|---|---|
| | Percentage | | | | Duration of | | |
| | of TL from | | Objective | Clinical Benefit | Response | Progression- | Overall |
| Subject | Baseline | Best Overall | Response | at Month 3/6/9 | (iDOR) | Free Survival | Survival |
| ID/Age/Sex | (%) | Response (iBOR) | (iOR) | (iCB) | (month) | (iPFS) (month) | (month) |
| XXXX-XXX/xx/M | XX.X | iCR | Yes | Yes/Yes/Yes | XXX.X* | XXX.X* | XXX.X* |
| XXXX-XXX/xx/F | XX.X | iSD | No | Yes/Yes/Yes | | XXX.X | XXX.X |
| XXXX-XXX/xx/F | XX.X | iSD | No | No/No/No | | XXX.X | XXX.X |
| M/xx/XXX-XXXX | XX.X | iPR | Yes | Yes/Yes/Yes | XXX.X | XXX.X | XXX.X* |
| XXXX-XXX/xx/F | XX.X | iCPD | No | No/No/No | | XXX.X | XXX.X |
| M/xx/XXX-XXXX | XX.X | iUPD | No | Yes/No/No | | XXX.X | XXX.X |
| M/xx/XXX-XXXX | XX.X | iSD | No | Yes/No/No | | XXX.X* | XXX.X* |
| XXXX-XXX/xx/F | XX.X | iSD | No | Yes/Yes/No | | XXX.X* | XXX.X* |
| XXXX-XXX/xx/M | | NE | No | No/No/No | | XXX.X | XXX.X* |

Note: TL = Target Lesion; iCR = Immune Complete Response; iPR = Immune Partial Response; iSD = Immune Stable Disease; iUPD = Immune Unconfirmed Progressive Disease; iCPD = Immune Confirmed Progressive Disease; NE = Not Evaluable.

Note: Best overall response of each subject is the best tumor response among all visits according to the following sequence: iCR, iPR, iSD, iCPD, iUPD, NE. See the definition of each parameter in SAP section 8.2.

Note: \* indicates the censor.

## **Programming Note:**

\* Sorting order is by Subject ID

Date: 26Feb2025

# Listing 16.2.7.1 Treatment-Emergent Adverse Events Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | Start Date | irAE?/ | | Relation to | |
|---|---|---|---|---|---|---|
| | System Organ Class/ | (Study Day)/ | AESI?/ | CRS?/Serious?/ | WTX-330/ | Outcome/ |
| Subject | Preferred Term/ | Stop Date | IRR?/ | NCI-CTCAE | Action Taken with | Concomitant or Additional |
| ID/Age/Sex | Verbatim | (Study Day) | DLT? | Grade/ASTCT Grade | WTX-330 | Treatment Given |
| XXXX-XXX/ | XXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/No/ | No/No/ | Unlikely/ | Recovered/ |
| xx/<br>M | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Ongoing | No/No | 2/ | Dose Not Changed | Concurrent Procedure |
| | xxxxxxxxxxxxxxxxxxx/ | DDMMMYYY (xx)/ | Yes/Yes/ | No/No/ | Unrelated/ | Recovered with Sequelae/ |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | DDMMMYYY (xx)/ | No/No | 1/ | Dose Interrupted | Concurrent Procedure |
| | xxxxxxxxxxxxxxxxx/ | DDMMMYYY (xx)/ | No/Yes/ | Yes/Yes/ | Probable/ | Not Recovered/ |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Ongoing | Yes/No | 4/ | Dose Reduced | Concomitant Medication |
| XXXX-XXX/ | XXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/No/ | Yes/No/ | Definite/ | Recovered with Sequelae/ |
| XX/<br>F | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx) | Yes/Yes | 1/ | Drug Withdrawn | Other:XXX |
| | XXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/No/ | No/Yes/ | Possible/ | Fatal/ |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx) | No/No | 5/ | Not Applicable | None |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Adverse Events are coded with MedDRA version 26.0. Adverse Events are graded with CTCAE Grade 5.0, except for Cytokine Release Syndrome which is graded with ASTCT Grade.

Note: A TEAE is defined as an AEs that emerges or worsens (i.e. increase in CTCAE grade/ASTCT Grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

Note: irAE = Immune Related Adverse Event; AESI = Adverse Event of Special Interest; IRR = Infusion Related Reaction; CRS = Cytokine Release Syndrome; DLT = Dose Limiting Toxicity; ASTCT = American Society for Transplantation and Cellular Therapy; Recovered = Recovered/Resolved; Not Recovered = Not Recovered/Not Resolved; Recovered with Sequelae = Recovered/Resolved with Sequelae.

## **Programming Note:**

Date: 26Feb2025

### Listing 16.2.7.2 Serious Adverse Events Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | Start Date | irAE?/ | CRS?/Serious?/ | Relation to | |
|---|---|---|---|---|---|---|
| | System Organ Class/ | (Study Day)/ | AESI?/ | NCI-CTCAE | WTX-330/ | Serious |
| Subject | Preferred Term/ | Stop Date | IRR?/ | Grade/ASTCT | Action Taken with | Adverse Event |
| ID/Age/Sex | Verbatim | (Study Day) | DLT? | Grade | WTX-330 | Category |
| XXXX-XXX/ | XXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/No/ | No/Yes/ | Unlikely/ | Required inpatient |
| xx/ | XXXXXXXXXXXXXXXXXXX/ | Ongoing | No/No | 2/ | Dose Not Changed | hospitalization or |
| М | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | prolongation of existing<br>hospitalization |
| | xxxxxxxxxxxxxxxxxxx/ | DDMMMYYY (xx)/ | Yes/Yes/ | No/Yes/ | Unrelated/ | Life Threatening |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | DDMMMYYY (xx)/ | No/No | 4/ | Dose Interrupted | |
| XXXX-XXX/<br>xx/<br>M | XXXXXXXXXXXXXXXXXXXXXXXXXXXX/<br>XXXXXXXXX | DDMMMYYY (xx)/<br>Ongoing | No/Yes/<br>Yes/No | Yes/Yes/<br>4/ | Probable/<br>Dose Reduced | Life Threatening;<br>Congenital Anomaly or Birth<br>Defect |
| XXXX-XXX/ | XXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/No/ | Yes/Yes/ | Definite/ | Other Medically Important |
| XX/<br>F | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx) | Yes/Yes | 3/ | Drug Withdrawn | Serious Event |
| | xxxxxxxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxxx | DDMMMYYY (xx)/<br>DDMMMYYY (xx) | No/No/<br>No/No | No/Yes/<br>5/ | Possible/<br>Not Applicable | Results in Death |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Adverse Events are coded with MedDRA version 26.0. Adverse Events are graded with CTCAE Grade 5.0, except for Cytokine Release Syndrome which is graded with ASTCT Grade.

Note: A TEAE is defined as an AEs that emerges or worsens (i.e. increase in CTCAE grade/ASTCT Grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

Note: irAE = Immune Related Adverse Event; AESI = Adverse Event of Special Interest; IRR = Infusion Related Reaction; CRS = Cytokine Release Syndrome; DLT = Dose Limiting Toxicity; ASTCT = American Society for Transplantation and Cellular Therapy; Recovered = Recovered/Resolved; Not Recovered = Not Recovered/Not Resolved; Recovered with Sequelae = Recovered/Resolved with Sequelae.

## **Programming Note:**

Date: 26Feb2025

# Listing 16.2.7.3 Treatment-Emergent Adverse Events Leading to Drug Withdrawal Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | Start Date | irAE?/ | CRS?/Serious?/ | Relation to | |
|---|---|---|---|---|---|---|
| | System Organ Class/ | (Study Day)/ | AESI?/ | NCI-CTCAE | WTX-330/ | Outcome/ |
| ~ 1 ! . | | | | | / | |
| Subject | Preferred Term/ | Stop Date | IRR?/ | Grade/ASTCT | Action Taken with | Concomitant or Additional |
| ID/Age/Sex | Verbatim | (Study Day) | DLT? | Grade | WTX-330 | Treatment Given |
| XXXX-XXX/ | XXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/No/ | No/No/ | Unlikely/ | Recovered/ |
| xx/ | XXXXXXXXXXXXXXXXX/ | Ongoing | No/No | 2/ | Drug Withdrawn | Concurrent Procedure |
| M | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | |
| XXXX-XXX/ | XXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | Yes/Yes/ | No/No/ | Unrelated/ | Recovered with Sequelae/ |
| xx/ | XXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/No | 1/ | Drug Withdrawn | Concurrent Procedure |
| М | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | |
| | XXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/Yes/ | Yes/Yes/ | Probable/ | Not Recovered/ |
| | XXXXXXXXXXXXXXXXXXX/ | Ongoing | Yes/No | 4/ | Drug Withdrawn | Concomitant Medication |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | |
| XXXX-XXX/ | xxxxxxxxxxxxxxxxxxx/ | DDMMMYYY (xx)/ | No/No/ | Yes/No/ | Definite/ | Recovered with Sequelae/ |
| XX/ | XXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx) | Yes/Yes | 1/ | Drug Withdrawn | Other:XXX |
| F | XXXXXXXXXXXXXXXXXXXXXX | | 100, 100 | -/ | | <del> </del> |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Adverse Events are coded with MedDRA version 26.0. Adverse Events are graded with CTCAE Grade 5.0, except for Cytokine Release Syndrome which is graded with ASTCT Grade.

Note: A TEAE is defined as an AEs that emerges or worsens (i.e. increase in CTCAE grade/ASTCT Grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

Note: irAE = Immune Related Adverse Event; AESI = Adverse Event of Special Interest; IRR = Infusion Related Reaction; CRS = Cytokine Release Syndrome; DLT = Dose Limiting Toxicity; ASTCT = American Society for Transplantation and Cellular Therapy; Recovered = Recovered/Resolved; Not Recovered = Not Recovered/Not Resolved; Recovered with Sequelae = Recovered/Resolved with Sequelae.

## **Programming Note:**

Date: 26Feb2025

## Listing 16.2.7.4 Treatment-Emergent Adverse Events Leading to Drug Modification Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| · | · | Start Date | irAE?/ | CRS?/Serious?/ | Relation to | Outcome/ |
|---|---|---|---|---|---|---|
| | System Organ Class/ | (Study Day)/ | AESI?/ | NCI-CTCAE | WTX-330/ | Concomitant or |
| Subject | Preferred Term/ | Stop Date | IRR?/ | Grade/ASTCT | Action Taken with | Additional Treatment |
| ID/Age/Sex | Verbatim | (Study Day) | DLT? | Grade | WTX-330 | Given |
| XXXX-XXX/ | XXXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/No/ | No/No/ | Unlikely/ | Recovered/ |
| xx/ | XXXXXXXXXXXXXXXXXXX/ | Ongoing | No/No | 2/ | Infusion Rate Reduced | Concurrent Procedure |
| М | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | |
| | XXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | Yes/Yes/ | No/No/ | Unrelated/ | Recovered with Sequelae/ |
| | XXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/No | 1/ | Dose Interrupted | Concurrent Procedure |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | |
| | XXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/Yes/ | Yes/Yes/ | Probable/ | Not Recovered/ |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Ongoing | Yes/No | 4/ | Dose Reduced | Concomitant Medication |
| XXXX-XXX/ | XXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/No/ | Yes/No/ | Definite/ | Recovered with Sequelae/ |
| XX/<br>F | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | DDMMMYYY (xx) | Yes/Yes | 1/ | Drug Withdrawn | Other:XXX |
| | XXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/No/ | No/Yes/ | Possible/ | Recovered with Sequelae/ |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx) | No/No | 3/ | Dose Delayed | None |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Adverse Events are coded with MedDRA version 26.0. Adverse Events are graded with CTCAE Grade 5.0, except for Cytokine Release Syndrome which is graded with ASTCT Grade.

Note: A TEAE is defined as an AEs that emerges or worsens (i.e. increase in CTCAE grade/ASTCT Grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

Note: irAE = Immune Related Adverse Event; AESI = Adverse Event of Special Interest; IRR = Infusion Related Reaction; CRS = Cytokine Release Syndrome; DLT = Dose Limiting Toxicity; ASTCT = American Society for Transplantation and Cellular Therapy; Recovered = Recovered/Resolved; Not Recovered = Not Recovered/Not Resolved; Recovered with Sequelae = Recovered/Resolved with Sequelae.

- \* Sorting order is by Subject ID, Start Date, System Organ Class and Preferred Term.
- \* WTX-330 Dose Delayed/ Dose Interrupted/Dose Reduced/Infusion Rate Reduced/Treatment Held

Date: 26Feb2025

# Listing 16.2.7.5 Treatment-Emergent Adverse Events of Special Interest Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | System Organ Class/ | Start Date<br>(Study Day)/ | irAE?/<br>AESI?/ | CRS?/Serious?/<br>NCI-CTCAE | Relation to<br>WTX-330/ | Outcome/<br>Concomitant or Additional |
|---|---|---|---|---|---|---|
| Subject | Preferred Term/ | Stop Date | IRR?/ | Grade/ASTCT | Action Taken with | Treatment Given/Special |
| ID/Age/Sex | Verbatim | (Study Day) | DLT? | Grade | WTX-330 | Interest Category |
| XXXX-XXX/ | XXXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/Yes/ | No/No/ | Unlikely/ | Recovered/ |
| XX/<br>F | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Ongoing | No/No | 2/ | Infusion Rate Reduced | Concurrent Procedure/<br>>=Grade 2 CRS |
| XXXX-XXX/<br>XX/<br>M | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/<br>DDMMMYYY (xx)/ | Yes/Yes/<br>No/No | Yes/No/<br>1/ | Unrelated/<br>Dose Interrupted | Recovered with Sequelae / Concurrent Procedure/ >=Grade 2 CLS |
| XXXX-XXX/<br>XX/<br>F | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | DDMMMYYY (xx)/<br>DDMMMYYY (xx) | No/Yes/<br>Yes/No | No/Yes/<br>5/ | Probable/<br>Dose Reduced | Fatal/<br>None/<br>Hy's Law |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Adverse Events are coded with MedDRA version 26.0. Adverse Events are graded with CTCAE Grade 5.0, except for Cytokine Release Syndrome which is graded with ASTCT Grade.

Note: A TEAE is defined as an AEs that emerges or worsens (i.e. increase in CTCAE grade/ASTCT Grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

Note: irAE = Immune Related Adverse Event; AESI = Adverse Event of Special Interest; IRR = Infusion Related Reaction; CRS = Cytokine Release Syndrome; DLT = Dose Limiting Toxicity; ASTCT = American Society for Transplantation and Cellular Therapy; Recovered = Recovered/Resolved; Not Recovered = Not Recovered/Not Resolved; Recovered with Sequelae = Recovered/Resolved with Sequelae.

## **Programming Note:**

Date: 26Feb2025

# Listing 16.2.7.6 Dose Limiting Toxicity Dose Limiting Toxicity Evaluable Analysis Set

| Dose Escalat | se Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease) | | | | | |
|---|---|---|---|---|---|---|
| | | Start Date | irAE?/ | | Relation to | Outcome/ |
| | System Organ Class/ | (Study Day)/ | AESI?/ | CRS?/Serious?/ | WTX-330/ | Concomitant or Additional |
| Subject | Preferred Term/ | Stop Date | IRR?/ | NCI-CTCAE | Action Taken with | Treatment Given/Dose |
| ID/Age/Sex | Verbatim | (Study Day) | DLT? | Grade/ASTCT Grade | WTX-330 | Limiting Toxicity Details |
| XXXX-XXX/ | XXXXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/No/ | No/No/ | Unlikely/ | Recovered/ |
| XX/<br>F | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Ongoing | No/Yes | 2/ | Infusion Rate<br>Reduced | Concurrent Procedure/ Any >= Grade 3 cytokine release syndrome (CRS) or capillary leak syndrome (CLS) |
| XXXX-XXX/<br>XX/<br>M | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/<br>DDMMMYYY (xx)/ | Yes/No/<br>No/ Yes | Yes/No/<br>1/ | Unrelated/<br>Dose Interrupted | Recovered with Sequelae / Concurrent Procedure/ Any Grade 2 non-hematological central nervous system (CNS) |
| XXXX-XXX/<br>XX/<br>F | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/<br>DDMMMYYY (xx) | No/Yes/<br>Yes/ Yes | No/Yes/<br>3/ | Probable/<br>Dose Reduced | Fatal/ None/ Any >= Grade 4 hematological adverse event |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Adverse Events are coded with MedDRA version 26.0. Adverse Events are graded with CTCAE Grade 5.0, except for Cytokine Release Syndrome which is graded with ASTCT Grade.

Note: irAE = Immune Related Adverse Event; AESI = Adverse Event of Special Interest; IRR = Infusion Related Reaction; CRS = Cytokine Release Syndrome; DLT = Dose Limiting Toxicity; ASTCT = American Society for Transplantation and Cellular Therapy; Recovered = Recovered/Resolved; Not Recovered = Not Recovered/Not Resolved; Recovered with Sequelae = Recovered/Resolved with Sequelae.

## **Programming Note:**

Date: 26Feb2025

# Listing 16.2.7.7 Treatment Emergent Adverse Events Leading to Death Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| Subject<br>ID/Age/Sex | System Organ Class/<br>Preferred Term/<br>Verbatim | Start Date<br>(Study Day)/<br>Stop Date<br>(Study Day) | irAE?/<br>AESI?/<br>IRR?/<br>DLT? | CRS?/Serious?/<br>NCI-CTCAE<br>Grade/ASTCT<br>Grade | Relation to<br>WTX-330/<br>Action Taken with<br>WTX-330 | Outcome/<br>Concomitant or Additional<br>Treatment Given |
|---|---|---|---|---|---|---|
| XXXX-XXX/<br>XX/<br>F | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/<br>Ongoing | No/No/<br>No/Yes | No/Yes/<br>5/ | Unlikely/<br>Infusion Rate Reduced | Fatal/<br>Concurrent Procedure |
| XXXX-XXX/<br>XX/<br>M | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/<br>DDMMMYYY(xx) | Yes/No/<br>No/ Yes | Yes/Yes/<br>5/ | Unrelated/<br>Dose Interrupted | Fatal/<br>Other:XXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/<br>DDMMMYYY (xx) | No/Yes/<br>Yes/ Yes | No/Yes/<br>5/ | Probable/<br>Dose Reduced | Fatal/<br>None |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Adverse Events are coded with MedDRA version 26.0. Adverse Events are graded with CTCAE Grade 5.0, except for Cytokine Release Syndrome which is graded with ASTCT Grade.

Note: A TEAE is defined as an AEs that emerges or worsens (i.e. increase in CTCAE grade/ASTCT Grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

Note: irAE = Immune Related Adverse Event; AESI = Adverse Event of Special Interest; IRR = Infusion Related Reaction; CRS = Cytokine Release Syndrome; DLT = Dose Limiting Toxicity; ASTCT = American Society for Transplantation and Cellular Therapy.

## **Programming Note:**

Date: 26Feb2025

# Listing 16.2.8.1 Hematology Tests with CTCAE Grade ≥ 3 Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | | | | Reference | | | |
|---|---|---|---|---|---|---|---|---|
| Subject | | | Collection Date Time | Change from | | Reference | Range | CTCAE |
| ID/Age/Sex | Test | Visit | (Study Day) | Baseline | Units | Range | Indicator | Grade |
| XXXX-XXX/XX/M | Hemoglobin | Screening | DDMMMYYYY HH:MM (XX) | XX.X | XX | XXX,XXX | Low | 1 |
| | | C1D1* | DDMMMYYYY HH:MM (XX) | XX.X* | XX | XXX,XXX | Normal | 0 |
| | | C1D8 | DDMMMYYYY HH:MM (XX) | XX.X/XX.X | XX | XXX,XXX | High | 2 |
| | | <insert></insert> | | | | | | |
| | <insert></insert> | | | | | | | |

### XXXX-XXX/XX/F

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Lab data is graded with CTCAE version 5.0.

Note: \* indicates baseline value.

- \* Sorting order is by Subject ID, Test, Collection date.
- \* if a subject with a test with CTCAE grade>=3, all visits of the test will be listed.

Date: 26Feb2025

# Listing 16.2.8.2.1 Serum Chemistry Tests with CTCAE Grade $\geq$ 3 Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | | | | Reference | | | |
|---|---|---|---|---|---|---|---|---|
| Subject | | | Collection Date Time | Change from | | Reference | Range | CTCAE |
| ID/Age/Sex | Test | Visit | (Study Day)/ | Baseline | Units | Range | Indicator | Grade |
| XXXX-XXX/XX/M | ALT | Screening | DDMMMYYYY HH:MM (XX) | XX.X | XX | XXX <b>,</b> XXX | Low | 1 |
| | | C1D1* | DDMMMYYYY HH:MM (XX) | XX.X* | XX | XXX,XXX | Normal | 0 |
| | | C1D8 | DDMMMYYYY HH:MM (XX) | XX.X/XX.X | XX | XXX,XXX | High | 2 |
| | | <insert></insert> | | | | | | |
| | <insert></insert> | | | | | | | |

### XXXX-XXX/XX/F

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Lab data is graded with CTCAE version 5.0.

Note: \* indicates baseline value.

- \* Sorting order is by Subject ID, Test, Collection date.
- \* if a subject with a test with CTCAE grade>=3, all visits of the test will be listed.

Date: 26Feb2025

### Listing 16.2.8.2.2 Liver Function Tests Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | | Aspartate | Alanine | Alkaline | Total |
|---|---|---|---|---|---|---|
| Subject | | Collection Date Time | Aminotransferase | Aminotransferase | Phosphatase | Bilirubin |
| ID/Age/Sex | Visit | (Study Day)/ | (AST) (XULN) | (ALT) (XULN) | (ALP) (XULN) | (xULN) |
| XXXX-XXX/XX/M | Screening | DDMMMYYYY HH:MM (XX) | 3 | 3 | 1.5 | 2 |
| | C1D1* | DDMMMYYYY HH:MM (XX) | 1.2 | 1.2 | 1.3 | 1.0 |
| | C1D8 | DDMMMYYYY HH:MM (XX) | 5.1 | 4.2 | 1.2 | 3 |
| | <insert></insert> | | | | | |

### XXXX-XXX/XX/M

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: \* indicates baseline value.

- \* Sorting order is by Subject ID, Collection date.
- \* if a subject with AST>=3, ALT>=3, or Total Bilirubin>=1.5, then all visits of these tests will be listed.

Date: 26Feb2025

# Listing 16.2.8.3 Coagulation Tests with CTCAE Grade $\geq$ 3 Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | | Result/ | | | | Reference | |
|---|---|---|---|---|---|---|---|---|
| Subject<br>ID/Age/Sex | Test | Visit | Collection Date Time (Study Day)/ | Change from<br>Baseline | Units | Reference<br>Range | Range<br>Indicator | CTCAE<br>Grade |
| XXXX-XXX/XX/M | Partial thromboplastin time | Screening | DDMMMYYYY HH:MM (XX) | XX.X | XX | XXX,XXX | Low | 1 |
| | | C1D1* | DDMMMYYYY HH:MM (XX) | XX.X* | XX | XXX,XXX | Normal | 0 |
| | | C1D8 | DDMMMYYYY HH:MM (XX) | XX.X/XX.X | XX | XXX,XXX | High | 2 |
| | | <insert></insert> | | | | | | |

<insert>

XXXX-XXX/XX/F

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Lab data is graded with CTCAE version 5.0.

Note: \* indicates baseline value.

- \* Sorting order is by Subject ID, Test, Collection date.
- \* if a subject with a test with CTCAE grade>=3, all visits of the test will be listed.

Date: 26Feb2025

# Listing 16.2.9 Vital Signs Clinically Notable Increase and/or Decrease Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| Subject<br>ID/Age/Sex | Test | Visit | Vital Signs Date Time<br>(Study Day)/ | Result/Change<br>from Baseline | Units | Increase or<br>Decrease [1] |
|---|---|---|---|---|---|---|
| XXXX-XXX/xx/F | Systolic blood pressure | Screening | DDMMMYYYY HH:MM (XX) | XX.X | XX | |
| | | C1D1* | DDMMMYYYY HH:MM (XX) | XX.X* | XX | |
| | | C1D2 | DDMMMYYYY HH:MM (XX) | XX.X/XX.X | XX | |
| | | C1D3 | DDMMMYYYY HH:MM (XX) | XX.X/XX.X | XX | |
| | | C1D8 | DDMMMYYYY HH:MM (XX) | XX.X/XX.X | XX | Increase |
| | | C1D15 | DDMMMYYYY HH:MM (XX) | XX.X/XX.X | XX | |
| | | C1D22 | DDMMMYYYY HH:MM (XX) | XX.X/XX.X | XX | |
| | | <insert></insert> | | | | |

<insert>

XXXX-XXX/xx/M

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: \* indicates baseline value.

[1] See SAP section 9.7 for the category.

- \* Sorting order is by Subject ID, Test, Collection date.
- \* if a subject with a test meeting the following category, all visits of the test will be listed.
  - Clinically notable elevated values:
    - o Systolic BP: ≥ 180 mmHg and an increase ≥ 20 mmHg from baseline
    - o Diastolic BP:  $\geq$  105 mmHg and an increase  $\geq$  15 mmHg from baseline
    - o Weight: Increase of ≥ 10% from baseline
    - Heart rate:  $\ge 120$  bpm with an increase of  $\ge 15$  bpm from baseline
    - o Temperature:  $> 38^{\circ}$  C
  - Clinically notable decrease values:
    - o Systolic BP: ≤90 mmHg and a decrease ≥ 20 mmHg from baseline
    - o Diastolic BP:  $\leq$  50 mmHg and a decrease  $\geq$  15 mmHg from baseline
    - Weight: decrease of  $\geq 10\%$  from baseline
    - Heart rate:  $\leq$  50 bpm and a decrease  $\geq$  15 bpm from baseline
    - Temperature: < 35° C

Date: 26Feb2025

### Listing 16.4.2.1 Medical History Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| Subject | Medical History | | | Date of Onset | End Date |
|---|---|---|---|---|---|
| ID/Age/Sex | Description | System Organ Class | Preferred Term | (Study Day) | (Study Day) |
| XXXX-XXX/xx/M | XXXXXXXXXXXXXX | XXXXXXXXXXXXXX | XXXXXXXXXXXXXX | DDMMMYYY (xx) | DDMMMYYY (xx) |
| | XXXXXXXXXXXXX | XXXXXXXXXXXXX | XXXXXXXXXXXXXX | DDMMMYYY (xx) | Ongoing |
| | XXXXXXXXXXXXX | XXXXXXXXXXXXX | XXXXXXXXXXXXXX | DDMMMYYY (xx) | YYYY |
| XXXX-XXX/xx/F | XXXXXXXXXXXXX | XXXXXXXXXXXXX | XXXXXXXXXXXXXX | Unknown | Unknown |
| | XXXXXXXXXXXXX | XXXXXXXXXXXXXX | XXXXXXXXXXXXXX | DDMMMYYY (xx) | DDMMMYYY (xx) |
| | XXXXXXXXXXXXXX | XXXXXXXXXXXXXX | XXXXXXXXXXXXXX | YYYY | Ongoing |
| | XXXXXXXXXXXXXX | XXXXXXXXXXXXXX | XXXXXXXXXXXXXX | MMMYYY | YYYY |
| | XXXXXXXXXXXXXX | XXXXXXXXXXXXXX | XXXXXXXXXXXXXX | DDMMMYYY (xx) | MMMYYY |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Medical history was coded with MedDRA version 26.0.

## **Programming Note:**

\* Sorting order is by Subject ID, System Organ Class, Preferred Term.

Date: 26Feb2025

# Listing 16.4.2.2.1 Solid Tumor Cancer History - Part 1 of 2 Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | Stage of | | | | | |
|---|---|---|---|---|---|---|---|
| | Date of Initial | Solid Tumor | Date of most Recent | | | | |
| | Histopathological | at Initial | Disease Recurrence/ | | | | |
| Subject | Diagnosis | Diagnosis/ | Progression | Cancer | Pathologic | Primary Site | Disease |
| ID/Age/Sex | (Study Day) | Current | (Study Day) | Type | Sub-type? | of Tumor | Measurable? |
| XXXX-XXX/xx/M | DDMMMYYY (xx) | 0/II | DDMMMYYY (xx) | Adrenal Cancer | No | Bone | Yes |
| XXXX-XXX/xx/F | DDMMMYYY (xx) | II/III | DDMMMYYY (xx) | Basal Cell Skin Cancer | No | Brain | No |
| XXXX-XXX/xx/F | DDMMMYYY (xx) | II/IV | DDMMMYYY (xx) | Bile Duct Cancer | No | Breast | Yes |
| XXXX-XXX/xx/F | DDMMMYYY (xx) | I/III | DDMMMYYY (xx) | Bladder Cancer | Yes: XXXX | Bronchus | Yes |
| XXXX-XXX/xx/F | DDMMMYYY (xx) | 0/IV | DDMMMYYY (xx) | Other: XXXXX | No | Cervix | No |
| XXXX-XXX/xx/M | DDMMMYYY (xx) | 0/II | DDMMMYYY (xx) | Endometrial Cancer | Yes: XXXX | Colon | No |
| XXXX-XXX/xx/M | DDMMMYYY (xx) | II/II | DDMMMYYY (xx) | Esophageal Cancer | No | Other: XXXXX | Yes |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

<sup>\*</sup> Sorting order is by Subject ID

Date: 26Feb2025

# Listing 16.4.2.2.2 Solid Tumor Cancer History - Part 2 of 2 Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | Genetic Analysis | MSI status | Characterization of | TMB Status | | Tumoral Genetic |
|---|---|---|---|---|---|---|
| Subject | Performed?/ | known?/ | Disease at Study | Known?/ Actual | | Characterization?/if Yes, |
| ID/Age/Sex | if Yes, Mutations | if Yes, Status | Entry | Mutation Burden | Unresectable | Specify Most Recent |
| XXXX-XXX/xx/M | No | Not Applicable | Locally Advanced | Not Applicable | Yes | No |
| XXXX-XXX/xx/F | Yes/BRAF | No | Metastatic: XXXXXX | No | No | Yes/XXXXXXXXXXXXXXX |
| XXXX-XXX/xx/F | Yes/EGFR, HER2 | Yes/MSI-H | Locally Advanced | Yes: High/xxx | Yes | No |
| XXXX-XXX/xx/F | Yes/KIT,<br>PDGFRA,PIK3CA | Yes/MSI-L | Metastatic: XXXXXX | Yes: Other/xxx | Yes | Yes/XXXXXXXXXXXXXXXX |
| XXXX-XXX/xx/F | Yes/NRAS | Yes/MSS | Locally Advanced | No | No | No |
| XXXX-XXX/xx/M | Yes/VHL | Yes/pMMR | Metastatic: XXXXXX | Yes:<br>Intermediate/xxx | No | No |
| XXXX-XXX/xx/M | Yes/Other: XXXX | No | Locally Advanced | Not Applicable | Yes | Yes/XXXXXXXXXXXXXXX |

<sup>\*</sup> Sorting order is by Subject ID

Date: 26Feb2025

# Listing 16.4.3.1 Prior Systemic Anti-Cancer Therapies Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | Line of | | | | | |
|---|---|---|---|---|---|---|
| | Therapy/ | | ATC Category II/ | | | |
| Subject | Therapy | | Preferred Name | Start Date/ | Therapy setting/ | Primary Reason for |
| ID/Age/Sex | Number | Type of Therapy | Therapy Name/ | End Date | Best Overall Response | Stopping Treatment |
| XXXX-XXX/xx/F | 1/1 | Immunotherapy | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>MMYYYY | Advanced/Metastatic<br>Partial Response | Treatment Completed |
| | 1/2 | Chemotherapy | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>DDMMMYYYY | Palliative/<br>Progression Of Disease | Progressive Disease |
| | 2/1 | Other: XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY/<br>YYYY | Other: XXXXXXXXXXXXX/ Stable Disease | Toxicity |
| XXXX-XXX/xx/M | 1/1 | Hormonal Therapy | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Unknown/<br>Unknown | Palliative/<br>Complete Response | Adverse Event |
| | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | MMYYYY/<br>DDMMMYYYY | Other: XXXXXXXXXXXX/<br>Not Applicable | Other: XXXXX |

Note: Medications are coded with WHODRUG Global B3 March 2023.

## **Programming Note:**

\* Sorting order is by Subject ID, Therapy Number, Therapy Name.

Date: 26Feb2025

### Listing 16.4.3.2 Prior Radiation Therapy Safety Analysis Set

| | Dose level or Arm/Disease | Subject | | | |
|---|---|---|---|---|---|
| Cohort | | ID/Age/Sex | Site of Radiation | Start Date | End Date |
| Dose Escalation | WTX-330 0.016 mg/kg | XXXX-XXX/xx/F | Adrenal Gland | DDMMMYYYY | DDMMMYYYY |
| | | | Bile duct | DDMMMYYYY | DDMMMYYYY |
| | | | Bronchus | YYYY | YYYY |
| | | XXXX-XXX/xx/M | Gall bladder | Unknown | Unknown |
| | | | Large Intestine | DDMMMYYYY | DDMMMYYYY |
| | | XXXX-XXX/xx/M | Other: XXXXXXXX | DDMMMYYYY | DDMMMYYYY |

Programming Note:\* Sorting order is by Cohort, Dose level or Arm/Disease, Subject ID, Start Date, Site of Radiation.

Date: 26Feb2025

### Listing 16.4.3.3 Prior Cancer Surgery Safety Analysis Set

| Cohort | Dose level or Arm/Disease | Subject<br>ID/Age/Sex | Surgical Procedure Name | Date of Surgery |
|---|---|---|---|---|
| Dose Escalation | WTX-330 0.016 mg/kg | XXXX-XXX/xx/F | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY<br>DDMMMYYYY<br>YYYY |
| | | XXXX-XXX/xx/M | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Unknown<br>DDMMMYYYY |
| | | XXXX-XXX/xx/M | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | DDMMMYYYY |

Programming Note:\* Sorting order is by Cohort, Dose level or Arm/Disease, Subject ID, Date of Surgery.

Date: 26Feb2025

# Listing 16.4.4.1 Prior and Concomitant Medications Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | ATC Category II/ | | Dose/ | |
|---|---|---|---|---|---|
| Subject | Prior or | Preferred Name/ | Start Date (Study Day)/ | Unit/ | |
| ID/Age/Sex | Concomitant | Medication Name | End Date (Study Day) | Route | Indication |
| XXXX-XXX/xx/F | Prior | XXXXXXXXXXXXXXXXXXXXXXXXXXXXX/<br>XXXXXXXX | DDMMMYYY (XX)/<br>Ongoing | XX/<br>XXXXX/<br>XXXXXX | Adverse Event: #x,#y, |
| | Concomitant | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (XX)/<br>DDMMMYYY (XX) | XX/<br>XXXXX<br>Other: XXXXXX | Medical History: #x,#y,#z |
| | Concomitant | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (XX)/<br>DDMMMYYY (XX) | XX/<br>XXXXX/<br>XXXXXXXXXX | Premedication |
| XXXX-XXX/xx/M | Concomitant | XXXXXXXXXXXXXXXXXXXXXXXXXXXX/<br>XXXXXXXXX | DDMMMYYY (XX)/<br>DDMMMYYY (XX) | XX/<br>XXXXX/<br>XXXXXXXX | Prophylactic Use |
| | Concomitant | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (XX)/<br>DDMMMYYY (XX) | XX/<br>XXXXX/<br>XXXXXXXXXX | Other: XXXXXX |
| XXXX-XXX/xx/F | Prior | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (XX)/<br>DDMMMYYY (XX) | XX/<br>Other/<br>XXXXXXXXXXXXXX | Medical History: #x,#y,#z |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Medications are coded with WHODRUG Global B3 March 2023.

Note: Prior medication is the medication that stopped before the first dose of WTX-330. Concomitant medication is the medication that is used on/after the first dose of WTX-330.

## **Programming Note:**

\* Sorting order is by Subject ID, Prior or Concomitant, ATC Category II.

Date: 26Feb2025

# Listing 16.4.4.2 Prior and Concomitant Procedures Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| Subject<br>ID/Age/Sex | Prior or<br>Concomitant | System Organ Class/<br>Preferred Term/<br>Name of Procedure | Start Date (Study Day)/<br>Stop Date (Study Day) | Indication |
|---|---|---|---|---|
| XXXX-XXX/xx/F | Prior | XXXXXXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/<br>DDMMMYYY (xx) | Adverse Event: #x, #y |
| | Concomitant | xxxxxxxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxxx | DDMMMYYY (xx)/<br>DDMMMYYY (xx) | Medical History: #x, #y |
| | Concomitant | xxxxxxxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxxx | DDMMMYYY (xx)/<br>DDMMMYYY (xx) | Prophylaxis |
| XXXX-XXX/xx/M | Prior | xxxxxxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxxxx | DDMMMYYY (xx)/<br>DDMMMYYY (xx) | Diagnostic/Exploratory |
| | Concomitant | xxxxxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxxxxx | DDMMMYYY (xx)/<br>DDMMMYYY (xx) | Treatment Of Underlying Disease |
| XXXX-XXX/xx/F | Concomitant | XXXXXXXXXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX | DDMMMYYY (xx)/<br>DDMMMYYY (xx) | Other: XXXXXXXXXX |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Prior procedure was coded with MedDRA version 26.0.

Note: Prior procedure is the procedure that stopped before the first dose of WTX-330. Concomitant procedure is the procedure that is performed on/after the first dose of WTX-330.

## **Programming Note:**

\* Sorting order is by Subject ID, Start Date.

Date: 26Feb2025

# Listing 16.4.5.1.1 WTX-330 Administration - Part 1 of 2 Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | WTX-330 | Preinfusion | Infusion Start | Infusion End | Planned | Planned |
|---|---|---|---|---|---|---|---|
| Subject | | Administered/ | Medication Taken?/ | Date Time | Date Time | Dose Level | Infusion |
| ID/Age/Sex | Visit | Reason Not Done | If Yes, Specify | (Study Day) | (Study Day) | (mg/kg) | Volume (mL) |
| XXXX-XXX/xx/F | C1D1 | Yes | Yes/XXXXXXXXXXXXX | DDMMMYYY HH:MM (XX) | DDMMMYYY HH:MM(XX) | XX | XXX |
| | C1D15 | No, COVID-19 Related | No | | | XX | XXX |
| | C2D1 | Yes | No | DDMMMYYY HH:MM (XX) | DDMMMYYY HH:MM(XX) | XX | XXX |
| | C2D15 | Yes | Yes/XXXXXXXXXXXXX | DDMMMYYY HH:MM (XX) | DDMMMYYY HH:MM(XX) | XX | XXX |
| | C3D1 | Yes | Yes/XXXXXXXXXXXXX | DDMMMYYY HH:MM (XX) | DDMMMYYY HH:MM(XX) | XX | XXX |
| | C3D15 | No, Other: XXX | No | | | XX | XXX |
| | <insert></insert> | | | DDMMMYYY HH:MM (XX) | DDMMMYYY HH:MM(XX) | XX | XXX |
| XXXX-XXX/xx/M | C1D1 | Yes | Yes/XXXXXXXXXXXXXX | DDMMMYYY HH:MM (XX) | DDMMMYYY HH:MM(XX) | XX | XXX |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

## **Programming Note:**

\* Sorting order is by Subject ID, Visit.

Date: 26Feb2025

### Listing 16.4.5.1.2 WTX-330 Administration - Part 2 of 2 Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | | Infusion | | | | _ |
|---|---|---|---|---|---|---|---|
| | | WTX-330 | Interrupted?/ | Time of | Actual Dose | | |
| Subject | | Administered/ | Reason for | Interruption/ | (mg/kg)/Total | Dose Adjustment?/ | Reason for |
| ID/Age/Sex | Visit | Reason Not Done | Interruption | Restart Time | Volume (mL) | Adjustment Type | Adjustment |
| XXXX-XXX/xx/F | C1D1 | Yes | No | | XX/XXX | No | _ |
| | C1D15 | No,COVID-19 Related | | | | | |
| | C2D1 | Yes | No | | XX/XXX | Yes/ Dose Missed | Adverse Event: #x |
| | C2D15 | Yes | Yes/Infusion<br>Reaction | HH:MM/HH:MM | XX/XXX | No | |
| | C3D1 | Yes | No | | XX/XXX | Yes/Dose Reduced | PI/Sponsor Decision |
| | C3D15<br><insert></insert> | No,Other: XXX | | | | | |
| XXXX-XXX/xx/M | C1D1 | Yes | Yes/Other: XXXXXX | HH:MM/No | XX/XXX | Yes/Dose<br>Discontinued | Other: XXXXXXXX |

Programming Note:
\* Sorting order is by Subject ID, Visit.

Date: 26Feb2025

Listing 16.4.5.2.1

Antineoplastic Therapy since Discontinuation of Study Treatment - Medication Safety Analysis Set

| Cohort | Dose level or Arm/Disease | Subject<br>ID/Age/Sex | Line of<br>Therapy | Agent | Therapy Start<br>Date | Therapy Stop<br>Date |
|---|---|---|---|---|---|---|
| Dose Escalation | WTX-330 0.016 mg/kg | XXXX-XXX/xx/M | 1 | XXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY | DDMMMYYYY |
| | | | | XXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY | DDMMMYYYY |
| | | | 2 | XXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY | Ongoing |
| | | | | XXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY | DDMMMYYYY |
| | | | 3 | XXXXXXXXXXXXXXXXXXXX | DDMMMYYYY | DDMMMYYYY |
| | XXXX-XXX | XXXX-XXX/xx/F | 1 | xxxxxxxxxxxxxxxxx | DDMMMYYYY | DDMMMYYYY |

<sup>\*</sup> Sorting order is by Cohort, Dose level or Arm/Disease, Subject ID, Line of Therapy, Agent.

Date: 26Feb2025

Listing 16.4.5.2.2

Antineoplastic Therapy since Discontinuation of Study Treatment - Radiation Safety Analysis Set

| Cohort | Dose level or Arm/Disease | Subject<br>ID/Age/Sex | Site of Radiation | Start Date | End Date |
|---|---|---|---|---|---|
| Dose Escalation | WTX-330 0.016 mg/kg | XXXX-XXX/xx/M | Adrenal Gland | DDMMMYYYY | DDMMMYYYY |
| | | | Bile duct | DDMMMYYYY | DDMMMYYYY |
| | | | Bronchus | YYYY | YYYY |
| | | XXXX-XXX/xx/M | Gall bladder | Unknown | Unknown |
| | | | Large Intestine | DDMMMYYYY | DDMMMYYYY |
| | | XXXX-XXX/xx/F | Other: XXXXXXXX | DDMMMYYYY | DDMMMYYYY |

<sup>\*</sup> Sorting order is by Cohort, Dose level or Arm/Disease, Subject ID, Start Date, Site of Radiation.

Date: 26Feb2025

### Listing 16.4.5.2.3 Antineoplastic Therapy since Discontinuation of Study Treatment - Surgery Safety Analysis Set

| Cohort | Dose level or Arm/Disease | Subject<br>ID/Age/Sex | Surgical Procedure Name | Date of Surgery |
|---|---|---|---|---|
| Dose Escalation | WTX-330 0.016 mg/kg | XXXX-XXX/xx/F | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY<br>DDMMMYYYY<br>YYYY |
| | | XXXX-XXX/xx/M | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Unknown<br>DDMMMYYYY |
| | | XXXX-XXX/xx/M | XXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY |

Programming Note:\* Sorting order is by Cohort, Dose level or Arm/Disease, Subject ID, Date of Surgery.

Date: 26Feb2025

Listing 16.4.6.1.1 Target Lesion Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | Date of | | | | | Short Axis and/or | Target |
|---|---|---|---|---|---|---|---|---|
| Subject | | Assessment | Lesion | | Location of | | Longest | Lesion |
| ID/Age/Sex | Visit | (Study Day) | # | Site/organ | the Lesion | Method | diameter (mm)[1] | Status |
| XXXX-XXX/xx/F | Screening | DDMMMYYY (XX) | 1 | Adrenal Gland | XXXXXXXXX | CTwC | XXX.X | |
| | | | 2 | Bronchus | XXXXXXXXX | CTwC | XXX.X | |
| | | | 3 | Bone | XXXXXXXXX | CTwC | XXX.X | |
| | Week 8 | DDMMMYYY (XX) | 1 | Adrenal Gland | XXXXXXXXX | CTwC | XXX.X | No change |
| | | | 2 | Bronchus | XXXXXXXXX | CTwC | XXX.X | No change |
| | | | 3 | Bone | XXXXXXXXX | CTwC | XXX.X | No change |
| XXXX-XXX/xx/M | Screening | DDMMMYYY (XX) | 1 | Kidney | XXXXXXXXX | Other:XX | XXX.X | |
| | | | 2 | Other:XXX | XXXXXXXXX | MRIwC | XXX.X | |
| | Week 8 | DDMMMYYY (XX) | 1 | Kidney | XXXXXXXXX | Other:XX | XXX.X | No change |
| | | | 2 | Other:XXX | XXXXXXXXX | MRIwC | XXX.X | No change |
| | Week 16 | DDMMMYYY (XX) | 1 | Kidney | XXXXXXXXX | Other:XX | XXX.X | Merged |
| | | | 2 | Other:XXX | XXXXXXXXX | MRIwC | NE | Absent |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: CTwC = CT scan with contrast; CTw/oC = CT scan without contrast; MRIwC = MRI scan with contrast; MRIw/oC = MRI scan without contrast; NE = Not evaluable.

[1] For the subjects with solid tumor, the results will be Lymph Node/Short Axis or Non-Lymph Node/Longest diameter; For the subjects with Lymphoma, the results will be Lymph Node/Short Axis and Lymph Node/Longest diameter. The results will be separated with "/".

## **Programming Note:**

\* Sorting order is by Subject ID, Visit, Lesion #

Date: 26Feb2025

Listing 16.4.6.1.2 Non-Target Lesion Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | Date of | | | | | Status of |
|---|---|---|---|---|---|---|---|
| Subject | | Assessment | Lesion | | Location of | | Non-Target |
| ID/Age/Sex | Visit | (Study Day) | # | Site/organ | the Lesion | Method | Lesion |
| XXXX-XXX | Screening | DDMMMYYY (XX) | 1 | Adrenal Gland | XXXXXXXXX | CTwC | |
| | | | 2 | Bronchus | XXXXXXXXX | CTwC | |
| | | | 3 | Bone | XXXXXXXXX | Bone Scan | |
| | Week 8 | DDMMMYYY (XX) | 1 | Adrenal Gland | XXXXXXXXX | CTwC | Absent |
| | | | 2 | Bronchus | XXXXXXXXX | CTwC | UPD |
| | | | 3 | Bone | XXXXXXXXX | Bone Scan | NE |
| XXXX-XXX | Screening | DDMMMYYY (XX) | 1 | Kidney | XXXXXXXXX | Other:XX | |
| | | | 2 | Other:XXX | XXXXXXXXX | MRIwC | |
| | Week 8 | DDMMMYYY (XX) | 1 | Kidney | XXXXXXXXX | Other:XX | No Increase |
| | | | 2 | Other:XXX | XXXXXXXXX | MRIwC | No Increase |
| | Week 16 | DDMMMYYY (XX) | 1 | Kidney | XXXXXXXXX | Other:XX | Increase |
| | | | 2 | Other:XXX | XXXXXXXXX | MRIwC | Increase |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: CTwC = CT scan with contrast; CTw/oC = CT scan without contrast; MRIwC = MRI scan with contrast; MRIw/oC = MRI scan without contrast; UPD=Unequivocal Progression; NE=Not Evaluable.

## **Programming Note:**

\* Sorting order is by Subject ID, Visit, Lesion #

Date: 26Feb2025

### Listing 16.4.6.1.3.1 New Target Lesion Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | Date of | | | | | Short Axis or | New Target |
|---|---|---|---|---|---|---|---|---|
| Subject | | Assessment | Lesion | | Location of | | Longest | Lesion |
| ID/Age/Sex | Visit | (Study Day) | # | Site/organ | the Lesion | Method | Diameter (mm) | Status |
| XXXX-XXX/xx/F | Week 8 | DDMMMYYY (XX) | 1 | Bronchus | XXXXXXXXX | CTwC | XXX.X | NA, New |
| | Week 16 | DDMMMYYY (XX) | 1 | Bronchus | XXXXXXXXX | CTwC | XXX.X | No Change |
| | Week 24 | DDMMMYYY (XX) | 1 | Bronchus | XXXXXXXXX | CTwC | XXX.X | Split |
| XXXX-XXX/xx/M | Week 8 | DDMMMYYY (XX) | 1 | Kidney | XXXXXXXXX | Other:XX | XXX.X | NA, New |
| | | | 2 | Other:XXX | XXXXXXXXX | MRIwC | XXX.X | NA, New |
| | Week 16 | DDMMMYYY (XX) | 1 | Kidney | XXXXXXXXX | Other:XX | XXX.X | Merged |
| | | | 2 | Other:XXX | XXXXXXXXX | MRIwC | NE | Absent |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: CTwC = CT scan with contrast; CTw/oC = CT scan without contrast; MRIwC = MRI scan with contrast; MRIw/oC = MRI scan without contrast; NE = Not evaluable.

## **Programming Note:**

\* Sorting order is by Subject ID, Visit, Lesion #

Date: 26Feb2025

### Listing 16.4.6.1.3.2 New Non-Target Lesion Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | Date of | | | | | New Status of |
|---|---|---|---|---|---|---|---|
| Subject | | Assessment | Lesion | | Location of | | Non-Target |
| ID/Age/Sex | Visit | (Study Day) | # | Site/organ | the Lesion | Method | Lesion |
| XXXX-XXX/xx/F | Week 8 | DDMMMYYY (XX) | 1 | Adrenal Gland | XXXXXXXXX | CTwC | NA, New |
| | Week 16 | DDMMMYYY (XX) | 1 | Bronchus | XXXXXXXXX | CTwC | UPD |
| | Week 24 | DDMMMYYY (XX) | 1 | Bone | XXXXXXXXX | Bone Scan | NE |
| XXXX-XXX/xxM | Week 8 | DDMMMYYY (XX) | 1 | Kidney | XXXXXXXXX | Other:XX | NA, New |
| | | | 2 | Other:XXX | XXXXXXXXX | MRIwC | NA, New |
| | Week 16 | DDMMMYYY (XX) | 1 | Kidney | XXXXXXXXX | Other:XX | No Increase |
| | | | 2 | Other:XXX | XXXXXXXXX | MRIwC | No Increase |
| | Week 24 | DDMMMYYY (XX) | 1 | Kidney | XXXXXXXXX | Other:XX | Increase |
| | | | 2 | Other:XXX | XXXXXXXXX | MRIwC | Increase |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: CTwC = CT scan with contrast; CTw/oC = CT scan without contrast; MRIwC = MRI scan with contrast; MRIw/oC = MRI scan without contrast; UPD = Unequivocal Progression; NE = Not Evaluable.

<sup>\*</sup> Sorting order is by Subject ID, Visit, Lesion #

Date: 26Feb2025

Listing 16.4.6.2

Disease Response - Solid Tumor

Efficacy Evaluable Population

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| Subject<br>ID/Age/Sex | Visit | Date of<br>Assessment<br>(Study Day) | Target<br>Lesion<br>Response | Sum of Target Lesion (mm)/ % Change from Baseline/ % Change from Nadir | Non-Target<br>Lesion<br>Response | Any New | | Overall<br>RECIST 1.1<br>Response | Overall<br>iRECIST<br>Response |
|---|---|---|---|---|---|---|---|---|---|
| XXXX-XXX/xx/F | Screening | DDMMMYYY (XX) | | XXX.X | | | | | |
| | Week 8 | DDMMMYYY (XX) | PR | xxx.x/xx.x/xx.x | NCRNPD | No | | PR* | iPR* |
| | Week 16 | DDMMMYYY (XX) | PR | xxx.x/xx.x/xx.x | NCRNPD | No | | PR | iPR |
| | Uns. | DDMMMYYY (XX) | PR | xxx.x/xx.x/xx.x | NCRNPD | No | | PR | iPR |
| | Week 24 | DDMMMYYY (XX) | PR | xxx.x/xx.x/xx.x | NCRNPD | No | | PR | iPR |
| | Week 32 | DDMMMYYY (XX) | PD | xxx.x/xx.x/xx.x | NE | Yes | 1 | PD | iUPD |
| XXXX-XXX/xx/M | Screening | DDMMMYYY (XX) | | xxx.x | | | | | |
| | Week 8 | DDMMMYYY (XX) | SD | xxx.x/xx.x/xx.x | NCRNPD | No | | SD* | iSD* |
| | Week 16 | DDMMMYYY (XX) | SD | xxx.x/xx.x/xx.x | NCRNPD | Yes | 1 | PD | iUPD |
| | Week 24 | DDMMMYYY (XX) | PD | xxx.x/xx.x/xx.x | CR | Yes | 1 | PD | iCPD |
| | Week 32 | DDMMMYYY (XX) | PD | xxx.x/xx.x/xx.x | CR | Yes | 3 | PD | iCPD |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: CR = Complete Response; PR = Partial Response; SD = Stable Disease; PD = Progressive Disease; NE=Not Evaluable; NCRNPD=Non-CR/Non-PD; iCR = Immune Complete Response; iPR = Immune Partial Response; iSD = Immune Stable Disease; iUPD = Immune Unconfirmed Progressive Disease; iCPD = Immune Confirmed Progressive Disease.

Note: \* indicates the first best overall response.

- \* Sorting order is by Subject ID, Visit.
- \* Flag the first best overall response

Date: 26Feb2025

# Listing 16.4.6.4 Prostate-specific Antigen (PSA) Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| Subject<br>ID/Age/Sex | Visit | Collection Date Time (Study Day)/ | PSA Sample<br>Collected? | Result<br>(ng/mL) | PSA Tumor Marker Response |
|---|---|---|---|---|---|
| | | | | . 3 . | rsa rumor marker kesponse |
| XXXX-XXX/xx/F | Screening | DDMMMYYYY HH:MM (XX) | Yes | XXX.X | |
| | Week 8 | DDMMMYYYY HH:MM (XX) | Yes | XXX.X | Non-response/Non-Progression |
| | Week 16 | DDMMMYYYY HH:MM (XX) | Yes | XXX.X | Non-response/Non-Progression |
| | Uns. | | No, COVID-19 Related | | |
| | Week 24 | DDMMMYYYY HH:MM (XX) | Yes | XXX.X | Progression |
| | Week 32 | DDMMMYYYY HH:MM (XX) | Yes | XXX.X | Progression |
| XXX-XXX/xx/M | Screening | DDMMMYYYY HH:MM (XX) | Yes | xxx.x | |
| | Week 8 | | No, Other: XXXXXXX | | |
| | Week 16 | DDMMMYYYY HH:MM (XX) | Yes | XXX.X | 50% decrease from baseline |
| | Week 24 | DDMMMYYYY HH:MM (XX) | Yes | XXX.X | 50% decrease from baseline |
| | Week 32 | DDMMMYYYY HH:MM (XX) | Yes | XXX.X | Not Evaluable |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Nore: Progression is defined as  $\geq$ = 25% increase and  $\geq$ =2 ng/mL increase from nadir.

## **Programming Note:**

\* Sorting order is by Subject ID, Visit.

Date: 26Feb2025

### Listing 16.4.7 All Adverse Events Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | Start Date | / | | | |
|---|---|---|---|---|---|---|
| | | (Study Day)/ | irAE?/ | CRS?/Serious?/ | Relation to | |
| | System Organ Class/ | Stop Date | AESI?/ | NCI-CTCAE | WTX-330/ | Outcome/ |
| Subject | Preferred Term/ | (Study Day)/ | IRR?/ | Grade/ASTCT | Action Taken with | Concomitant or Additional |
| ID/Age/Sex | Verbatim | TEAE? | DLT? | Grade | WTX-330 | Treatment Given |
| XXXX- | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/ | No/No/ | No/No/ | Unlikely/ | Recovered/ |
| XXX/xx/F | XXXXXXXXXXXXXXXXX/ | Ongoing/ | No/No | 2/ | Dose Not Changed | Concurrent Procedure |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | No | | | | |
| | xxxxxxxxxxxxxxxxxxx/ | DDMMMYYY (xx)/ | Yes/Yes/ | No/No/ | Unrelated/ | Recovered with Sequelae/ |
| | XXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/No | 1/ | Dose Interrupted | Concurrent Procedure |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes | | | | |
| | XXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/Yes/ | Yes/Yes/ | Probable/ | Not Recovered/ |
| | XXXXXXXXXXXXXXXXX/ | Ongoing/ | Yes/No | 4/ | Dose Reduced | Concomitant Medication |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes | | | | |
| XXXX- | xxxxxxxxxxxxxxxxxxx/ | DDMMMYYY (xx)/ | No/No/ | Yes/No/ | Definite/ | Recovered with Sequelae/ |
| XXX/xx/M | XXXXXXXXXXXXXXXXXX/ | DDMMMYYY(xx)/ | Yes/Yes | 1/ | Drug Withdrawn | Other:XXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes | | | | |
| | XXXXXXXXXXXXXXXXXXXX/ | DDMMMYYY (xx)/ | No/No/ | No/Yes/ | Possible/ | Fatal/ |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYY (xx)/ | No/No | 5/ | Not Applicable | None |
| | XXXXXXXXXXXXXXXXXXXXXX | Yes | -, | *, | 11 | |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Adverse Events are coded with MedDRA version 26.0. Adverse Events are graded with CTCAE Grade 5.0, except for Cytokine Release Syndrome which is graded with ASTCT Grade.

Note: A TEAE is defined as an AEs that emerges or worsens (i.e. increase in CTCAE grade/ASTCT Grade) on/after the first WTX-330 dose and within 30 days of the last WTX-330 dose or the start of a new cancer regimen, whichever occurs earlier.

Note: irAE = Immune Related Adverse Event; AESI = Adverse Event of Special Interest; IRR = Infusion Related Reaction; CRS = Cytokine Release Syndrome; DLT = Dose Limiting Toxicity; ASTCT = American Society for Transplantation and Cellular Therapy; Recovered = Recovered/Resolved; Not Recovered = Not Recovered/Not Resolved; Recovered with Sequelae = Recovered/Resolved with Sequelae.

## **Programming Note:**

Date: 26Feb2025

### Listing 16.4.8.1 Hematology Tests Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | | | | Reference | | | |
|---|---|---|---|---|---|---|---|---|
| Subject<br>ID/Age/Sex | Test | Visit | Collection Date Time<br>(Study Day) | Change from<br>Baseline | Units | Reference<br>Range | Range<br>Indicator | CTCAE<br>Grade |
| XXXX-XXX/xx/F | Hemoglobin | Screening | DDMMMYYYY HH:MM (XX) | XX.X | XX | XXX,XXX | Low | 1 |
| | | C1D1 | DDMMMYYYY HH:MM (XX) | XX.X* | XX | XXX,XXX | Normal | 0 |
| | | C1D8 | DDMMMYYYY HH:MM (XX) | XX.X/XX.X | XX | XXX,XXX | High | 2 |
| | | <insert></insert> | | | | | | |

<insert>

XXXX-XXX/xx/M

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Lab data is graded with CTCAE version 5.0.

Note: \* indicates baseline value.

## **Programming Note:**

\* Sorting order is by Subject ID, Test, Collection date.

Date: 26Feb2025

### Listing 16.4.8.2 Serum Chemistry Tests Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | | | Result/ | | | Reference | |
|---|---|---|---|---|---|---|---|---|
| Subject | | | Collection Date Time | Change from | | Reference | Range | CTCAE |
| ID/Age/Sex | Test | Visit | (Study Day)/ | Baseline | Units | Range | Indicator | Grade |
| XXXX-XXX/xx/F | ALT | Screening | DDMMMYYYY HH:MM (XX) | XX.X | XX | XXX,XXX | Low | 1 |
| | | C1D1 | DDMMMYYYY HH:MM (XX) | XX.X* | XX | XXX,XXX | Normal | 0 |
| | | C1D8 | DDMMMYYYY HH:MM (XX) | XX.X/XX.X | XX | XXX,XXX | High | 2 |
| | | <insert></insert> | | | | | | |

<insert>

XXXX-XXX/xx/M

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Lab data is graded with CTCAE version 5.0.

Note: \* indicates baseline value.

## **Programming Note:**

\* Sorting order is by Subject ID, Test, Collection date.

Date: 26Feb2025

### Listing 16.2.8.3 Coagulation Tests Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | | | Result/ | | | Reference | |
|---|---|---|---|---|---|---|---|---|
| Subject | | | Collection Date Time | Change from | | Reference | Range | CTCAE |
| ID/Age/Sex | Test | Visit | (Study Day)/ | Baseline | Units | Range | Indicator | Grade |
| XXXX-XXX/xx/F | Partial thromboplastin time | Screening | DDMMMYYYY HH:MM (XX) | XX.X | XX | XXX,XXX | Low | 1 |
| | | C1D1 | DDMMMYYYY HH:MM (XX) | XX.X* | XX | XXX,XXX | Normal | 0 |
| | | C1D8 | DDMMMYYYY HH:MM (XX) | XX.X/XX.X | XX | XXX,XXX | High | 2 |
| | | <insert></insert> | | | | | | |
| | <insert></insert> | | | | | | | |

XXXX-XXX/xx/M

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: Lab data is graded with CTCAE version 5.0.

Note: \* indicates baseline value.

## **Programming Note:**

\* Sorting order is by Subject ID, Test, Collection date.
Date: 26Feb2025

Listing 16.4.8.4 Urinalysis Tests Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| Subject | | Collection Date Time | |
|---|---|---|---|
| ID/Age/Sex Test | Visit | (Study Day) | Result |
| XXXX-XXX/xx/F Turbidity | Screening | DDMMMYYYY HH:MM (XX) | Clear |
| | C1D1* | DDMMMYYYY HH:MM (XX) | Slightly Cloudy |
| | C1D8 | DDMMMYYYY HH:MM (XX) | Cloudy |
| | C1D15 | DDMMMYYYY HH:MM (XX) | Cloudy |
| | <insert></insert> | DDMMMYYYY HH:MM (XX) | Turbid |
| <insert></insert> | | | |

XXXX-XXX/xx/M

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: \* indicates baseline value.

## **Programming Note:**

\* Sorting order is by Subject ID, Test, Collection date.

Date: 26Feb2025

#### Listing 16.4.8.5 Thyroid Stimulating Hormone Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| Subject<br>ID/Age/Sex | Test | Visit | Collection Date Time<br>(Study Day)/ | Result/<br>Change from Baseline | Unit |
|---|---|---|---|---|---|
| XXXX-XXX/xx/F | Thyroid stimulating hormone | Screening | DDMMMYYYY HH:MM (XX) | XX.X | XX |
| AAAA AAA/AA/I | ingloid Scimulating normone | C1D1 | DDMMYYYY HH:MM (XX) | XX.X* | XX |
| | | C1D8 | DDMMMYYYY HH:MM (XX) | XX.X/XX.X | XX |
| | | <insert></insert> | | | |

<insert>

XXXX-XXX/xx/M

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: \* indicates baseline value.

- \* Sorting order is by Subject ID, Test, Collection date.
- \* including Thyroid stimulating hormone (TSH), Free triiodothyronine (T3), Free thyroxine (T4), Total triiodothyronine (T3), Total thyroxine (T4)

Date: 26Feb2025

# Listing 16.4.8.6 Pregnancy Test Safety Analysis Set

| Cohort | Dose level or<br>Arm/Disease | Subject<br>ID/Age/Sex | Visit | Collection Date Time<br>(Study Day) | Pregnancy<br>Test Type | Pregnancy<br>Test Result |
|---|---|---|---|---|---|---|
| Dose Escalation | WTX-330 0.016 mg/kg | XXXX-XXX/xx/F | Screening<br>C1D15<br><insert></insert> | DDMMMYYYY HH:MM (XX) DDMMMYYYY HH:MM (XX) DDMMMYYYY HH:MM (XX) | Serum<br>Urine<br>Urine | Negative<br>Negative<br>Negative |
| | | XXXX-XXX/xx/F | | | | |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

# **Programming Note:**

\* Sorting order is by Cohort, Dose level or Arm/Disease, Subject ID, Collection Date.

Date: 26Feb2025

Date: 26Feb2025

#### Listing 16.4.9.1 12-Lead ECG Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| | | | ECG | | | | | |
|---|---|---|---|---|---|---|---|---|
| Subject | Test | | Position | ECG Date Time | | | | Mean/Change |
| ID/Age/Sex | (unit) | Visit | of Subject | (Study Day) | Time Point | ECG # | Result | from Baseline |
| XXXX-XXX/xx/F | PR (msec) | Screening | | DDMMMYYYY HH:MM(XX) | Screening | | xxx.x | |
| | | C1D1 | Sitting | DDMMMYYYY HH:MM(XX) | Pre-dose | 1 | XXX.X | XX.X* |
| | | | | DDMMMYYYY HH:MM(XX) | Pre-dose | 2 | XXX.X | |
| | | | | DDMMMYYYY HH:MM(XX) | Pre-dose | 3 | XXX.X | |
| | | C1D1 | Sitting | DDMMMYYYY HH:MM(XX) | Immediately after WTX-330 infusion | 1 | XXX.X | XX.X/XX.X |
| | | | | DDMMMYYYY HH:MM(XX) | Immediately after WTX-330 infusion | 2 | XXX.X | |
| | | | | DDMMMYYYY HH:MM(XX) | Immediately after WTX-330 infusion | 3 | XXX.X | |
| | | C1D1 | Sitting | DDMMMYYYY HH:MM(XX) | 4 hours after WTX-330 infusion | 1 | xxx.x | XX.X/XX.X |
| | | | | DDMMMYYYY HH:MM(XX) | 4 hours after WTX-330 infusion | 2 | xxx.x | |
| | | | | DDMMMYYYY HH:MM(XX) | 4 hours after WTX-330 infusion | 3 | xxx.x | |
| | | <insert></insert> | | | | | | |

#### XXXX-XXX

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: \* indicates baseline value.

- \* Sorting order is by Subject ID, Test, ECG Date, Time Point, ECG#
- \* Mean/Change from Baseline is reported in the row of ECG# =1.

Date: 26Feb2025

Listing 16.4.9.2 Vital Signs Safety Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| Subject | | | Vital Signs Date Time | | |
|---|---|---|---|---|---|
| ID/Age/Sex Test (unit) | | Visit | Visit (Study Day) Result | | Baseline |
| XXXX-XXX/xx/F | Weight (kg) | Screening | DDMMMYYYY HH:MM(XX) | XXX.X | |
| | | C1D1 | DDMMMYYYY HH:MM(XX) | xxx.x* | |
| | | C1D2 | DDMMMYYYY HH:MM(XX) | XXX.X | XX.X |
| | | C1D3 | DDMMMYYYY HH:MM(XX) | XXX.X | XX.X |
| | | C1D8 | DDMMMYYYY HH:MM(XX) | XXX.X | XX.X |
| | | C1D15 | DDMMMYYYY HH:MM(XX) | XXX.X | XX.X |
| | | <insert></insert> | | | |

XXXX-XXX/xx/M

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: \* indicates baseline value.

# **Programming Note:**

\* Sorting order is by Subject ID, Test, Vital Signs Date

Date: 26Feb2025

#### Listing 16.4.9.3 ECOG Performance Status Safety Analysis Set

| Cohort | Dose level or Arm/Disease | Subject<br>ID/Age/Sex | Performed?/<br>Reason Not Done | Visit | Date of<br>Assessment<br>(Study Day) | Result |
|---|---|---|---|---|---|---|
| Dose Escalation | WTX-330 0.016 mg/kg | XXXX-XXX/xx/F | Yes | Screening | DDMMMYYYY (XX) | 0 |
| | | | | C1D1 | DDMMMYYYY (XX) | 1 |
| | | | No, Other: XXXXXXXX | C1D8 | | |
| | | | | <insert></insert> | | |
| | | XXXX-XXX/xx/M | Yes | Screening | DDMMMYYYY (XX) | 0 |
| | | | Yes | C1D1 | DDMMMYYYY (XX) | 0 |
| | | | Yes | C1D8 | DDMMMYYYY (XX) | 2 |
| | | | No, COVID-19 Related | C1D15 | | |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

Note: 0 - Fully active, able to carry on all pre-disease performance without restriction; 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work;

- 2 Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4 Completely disabled. Cannot carry
- on any selfcare. Totally confined to bed or chair

## **Programming Note:**

\* Sorting order is by Cohort, Dose level or Arm/Disease, Subject ID, Visit.

Date: 26Feb2025

Listing 16.4.9.4 Physical Examination Safety Analysis Set

| Cohort | Dose level or<br>Arm/Disease | Subject<br>ID/Age/Sex | Performed?/<br>Reason Not Done | Visit | Date of<br>Assessment<br>(Study Day) | Physical<br>Exam Result | Clinical<br>Significance |
|---|---|---|---|---|---|---|---|
| Dose Escalation | WTX-330 0.016 mg/kg | XXXX-XXX/xx/F | Yes | Screening | DDMMMYYYY (XX) | Normal | |
| | | | | C1D1 | DDMMMYYYY (XX) | Abnormal | No |
| | | | No, Other: XXXXXXXX | C1D8 | | Not Done | |
| | | | | <insert></insert> | | | |
| | | XXXX-XXX/xx/M | Yes | Screening | DDMMMYYYY (XX) | Normal | |
| | | | Yes | C1D1 | DDMMMYYYY (XX) | Abnormal | Yes: XXXXXX |
| | | | Yes | C1D8 | DDMMMYYYY (XX) | Normal | |
| | | | No, COVID-19 Related | C1D15 | | Not Done | |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

<sup>\*</sup> Sorting order is by Cohort, Dose level or Arm/Disease, Subject ID, Visit.

Date: 26Feb2025

# $\begin{tabular}{ll} Listing 16.4.10.1.1 \\ WTX-330 Plasma Concentrations ($\mu g/ml$) \\ Pharmacokinetic Analysis Set \\ \end{tabular}$

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| Subject | | Collection Date Time | | |
|---|---|---|---|---|
| ID/Age/Sex | Visit | (Study Day) | Time Point | Result |
| XXXX-XXX/xx/F | C1D1 | DDMMMYYYY HH:MM(XX) | Pre-dose | XXX.X |
| | C1D1 | DDMMMYYYY HH:MM(XX) | Immediately after (±2 minutes) WTX-330 infusion | XXX.X |
| | C1D1 | DDMMMYYYY HH:MM(XX) | 4 hours (±30 minutes) post start of WTX-330 infusion | XXX.X |
| | C1D1 | DDMMMYYYY HH:MM(XX) | 8 hours (±30 minutes) post start of WTX-330 infusion | XXX.X |
| | C1D2 | DDMMMYYYY HH:MM(XX) | 24 hours (±2 hours) post start of WTX-330 infusion | XXX.X |
| | C1D3 | DDMMMYYYY HH:MM(XX) | 48 hours (±2 hours) post start of WTX-330 infusion | xxx.x |
| | C1D8 | DDMMMYYYY HH:MM(XX) | 168 hours (±4 hours) post start of WTX-330 Infusion | XXX.X |
| | <insert></insert> | | | |

XXXX-XXX

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

# **Programming Note:**

\* Sorting order is by Subject ID, Visit, Time Point

Date: 26Feb2025

# Listing 16.4.10.1.2 Free IL-12 Plasma Concentrations (pg/ml) Pharmacokinetic Analysis Set

Dose Escalation: WTX-330 0.016 mg/kg (Phase Therapy: Dose level or Arm/Disease)

| Subject | | Collection Date Time | | |
|---|---|---|---|---|
| ID/Age/Sex | Visit | (Study Day) | Time Point | Result |
| XXXX-XXX/xx/F | C1D1 | DDMMMYYYY HH:MM(XX) | Pre-dose | XXX.X |
| | C1D1 | DDMMMYYYY HH:MM(XX) | Immediately after (±2 minutes) WTX-330 infusion | XXX.X |
| | C1D1 | DDMMMYYYY HH:MM(XX) | 4 hours (±30 minutes) post start of WTX-330 infusion | XXX.X |
| | C1D1 | DDMMMYYYY HH:MM(XX) | 8 hours (±30 minutes) post start of WTX-330 infusion | XXX.X |
| | C1D2 | DDMMMYYYY HH:MM(XX) | 24 hours (±2 hours) post start of WTX-330 infusion | XXX.X |
| | C1D3 | DDMMMYYYY HH:MM(XX) | 48 hours (±2 hours) post start of WTX-330 infusion | XXX.X |
| | C1D8 | DDMMMYYYY HH:MM(XX) | 168 hours (±4 hours) post start of WTX-330 Infusion | XXX.X |
| | <insert></insert> | | | |

XXXX-XXX

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

# **Programming Note:**

\* Sorting order is by Subject ID, Visit, Time Point

Date: 26Feb2025

#### Listing 16.4.10.2.1 WTX-330 Pharmacokinetic Parameters Pharmacokinetic Analysis Set

| | | Subject | | | | |
|---|---|---|---|---|---|---|
| Cohort | Dose level or Arm/Disease | ID/Age/Sex | Cycle | Parameter | Result | Unit |
| Dose Escalation | WTX-330 0.016 mg/kg | XXXX-XXX/xx/F | Cycle 1 | AUC <sub>0-14d</sub> | XX.X | XXXX |
| | | | | $C_{\text{max}}$ | XX.X | XXXX |
| | | | | $T_{	exttt{max}}$ | XX.X | XXXX |
| | | | | <insert></insert> | XX.X | XXXX |
| | | | Cycle 2 | AUC <sub>0-14d</sub> | XX.X | XXXX |
| | | | | $C_{\text{max}}$ | XX.X | XXXX |
| | | | | $T_{	exttt{max}}$ | XX.X | XXXX |
| | | | | <insert></insert> | XX.X | XXXX |
| | | <insert></insert> | | | | |

<sup>\*</sup> Sorting order is by Cohort, Dose level or Arm/Disease, Subject ID, Cycle.

Date: 26Feb2025

# Listing 16.4.10.2.1 Free IL-12 Pharmacokinetic Parameters Pharmacokinetic Analysis Set

| | Subject | | | | |
|---|---|---|---|---|---|
| Dose level or Arm/Disease | ID/Age/Sex | Cycle | Parameter | Result | Unit |
| WTX-330 0.016 mg/kg | XXXX-XXX/xx/F | Cycle 1 | AUC <sub>0-14d</sub> | XX.X | XXXX |
| | | | $C_{\text{max}}$ | XX.X | XXXX |
| | | | $T_{	exttt{max}}$ | XX.X | XXXX |
| | | | <insert></insert> | XX.X | XXXX |
| | | Cycle 2 | AUC <sub>0-14d</sub> | XX.X | XXXX |
| | | | $C_{\text{max}}$ | XX.X | XXXX |
| | | | $T_{	exttt{max}}$ | XX.X | XXXX |
| | | | <insert></insert> | XX.X | XXXX |
| | <insert></insert> | | | | |
| | <u>-</u> | Dose level or Arm/Disease ID/Age/Sex WTX-330 0.016 mg/kg XXXX-XXX/xx/F | Dose level or Arm/Disease ID/Age/Sex Cycle WTX-330 0.016 mg/kg XXXX-XXX/xx/F Cycle 1 Cycle 2 | Dose level or Arm/Disease ID/Age/Sex Cycle Parameter WTX-330 0.016 mg/kg XXXX-XXX/xx/F Cycle 1 $\begin{array}{c} AUC_{0-14d} \\ C_{max} \\ T_{max} \\ < insert > \\ C_{max} \\ T_{max} \\ < insert > \\ \end{array}$ | $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ |

<sup>\*</sup> Sorting order is by Cohort, Dose level or Arm/Disease, Subject ID, Cycle.

Date: 26Feb2025

# Listing 16.4.10.3 Anti-Drug Antibody Anti-Drug Antibody Analysis Set

| Cohort | Dose level or Arm/Disease | Subject<br>ID/Age/Sex | Visit | Collection Date Time<br>(Study Day)/ | Time Point | Numeric<br>Result | Categoric<br>Result |
|---|---|---|---|---|---|---|---|
| Dose Escalation | WTX-330 0.016 mg/kg | XXXX-XXX/xx/F | C1D1 | DDMMMYYYY HH:MM (XX) | Pre-dose | XX.X | Negative |
| | | | C1D15 | DDMMMYYYY HH:MM (XX) | Pre-dose | XX.X | Negative |
| | | | C2D1 | DDMMMYYYY HH:MM (XX) | Pre-dose | XX.X | Positive |
| | | | C2D15 | DDMMMYYYY HH:MM (XX) | Any time | XX.X | Positive |
| | | | C3D1 | DDMMMYYYY HH:MM (XX) | Pre-dose | XX.X | Positive |
| | | | <insert></insert> | | | | |
| | | <insert></insert> | | | | | |

Note: Study day = Assessment date - Date of Day 1 + 1 if assessment date is on/after the first WTX-330 dose; Study day = Assessment date - Date of Day 1 if assessment date is before the first WTX-330 dose.

# **Programming Note:**

\* Sorting order is by Cohort, Dose level or Arm/Disease, Subject ID, Visit.



#### **Certificate Of Completion**

Envelope Id: 2EC316E2-48C0-4ED4-8261-DCEF7D99307B Status: Completed Subject: Complete with Docusign: WTX-330x2101 (WWT21330) SAP text 2.pdf, WTX-330x2101 (WWT21330) TFL she...

Source Envelope:

Document Pages: 193 Certificate Pages: 5 AutoNav: Enabled

**Envelopeld Stamping: Disabled** Time Zone: (UTC) Monrovia, Reykjavik Signatures: 4 Initials: 0

Inc 2700 Wycliff Road, Suite 340

Raleigh, NC 27607 Shuangli.Guo@caidya.com IP Address: 71.206.118.21

Sent: 26-Feb-2025 | 19:27

Viewed: 26-Feb-2025 | 19:28

Signed: 26-Feb-2025 | 19:29

Envelope Originator:

Shuangli Guo

#### **Record Tracking**

Status: Original Holder: Shuangli Guo Location: DocuSign

| 26-Feb-2025 19:20 | Shuangli.Guo@caidya.com | |
|---|---|---|
| Signer Events | Signature | Timestamp |
| Oliver Schönborn-Kellenberger<br>oliver.schoenborn-kellenberger@cogitars.com<br>Security Level: Email, Account Authentication<br>(Required) | Oliver Schönborn-Kıllenberger | Sent: 26-Feb-2025 19:27<br>Viewed: 26-Feb-2025 19:55<br>Signed: 26-Feb-2025 20:00 |
| | Signature Adoption: Pre-selected Style | |
| | Signature ID: | |
| | 988B94B1-FDA2-4A35-AEB8-361DCA46EBF3 | |
| | Using IP Address: 176.199.208.46 | |
| | Signed using mobile | |
| | With Signing Authentication via Docusign password | |
| | With Signing Reasons (on each tab): | |
| | Ich genehmige dieses Dokument | |
| | Ich habe dieses Dokument geprüft | |
| Electronic Record and Signature Disclosure: | | |
| A | | |

Accepted: 26-Feb-2025 | 19:55

ID: f4e5de15-c617-41b7-9f36-373027ccec1e

Shuangli Guo

shuangli.guo@caidya.com Senior Manager, Biostatistics

Caidya

Security Level: Email, Account Authentication (Required)

Sungli Gua

Signature Adoption: Pre-selected Style

Signature ID:

3F1277AD-321D-4048-BF56-4AE5BED08E47

Using IP Address: 71.206.118.21

With Signing Authentication via Docusign password

With Signing Reasons (on each tab): I am the author of this document I am the author of this document

#### **Electronic Record and Signature Disclosure:**

Not Offered via Docusign

| In Person Signer Events | Signature | Timestamp |
|------------------------------|-----------|-----------|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |

| Certified Delivery Events | Status | Timestamp |
|---|---|---|
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Summary Events Envelope Sent | Status Hashed/Encrypted | <b>Timestamps</b><br>26-Feb-2025 19:27 |
| • | | • |
| Envelope Sent | Hashed/Encrypted | 26-Feb-2025 19:27 |
| Envelope Sent<br>Certified Delivered | Hashed/Encrypted Security Checked | 26-Feb-2025 19:27<br>26-Feb-2025 19:28 |
| Envelope Sent Certified Delivered Signing Complete | Hashed/Encrypted Security Checked Security Checked | 26-Feb-2025 19:27<br>26-Feb-2025 19:28<br>26-Feb-2025 19:29 |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Caidya (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

## Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

### **How to contact Caidya:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: rupali.kumbhar@caidya.com

### To advise Caidya of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at rupali.kumbhar@caidya.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

## To request paper copies from Caidya

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to rupali.kumbhar@caidya.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

### To withdraw your consent with Caidya

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to rupali.kumbhar@caidya.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Caidya as described above, you consent to receive exclusively
  through electronic means all notices, disclosures, authorizations, acknowledgements, and
  other documents that are required to be provided or made available to you by Caidya
  during the course of your relationship with Caidya.